CLINICAL TRIAL: NCT02528253
Title: A PHASE 3, RANDOMIZED, DOUBLE BLIND, PLACEBO AND ACTIVE-CONTROLLED, MULTICENTER, PARALLEL-GROUP STUDY OF THE ANALGESIC EFFICACY AND SAFETY OF TANEZUMAB IN ADULT SUBJECTS WITH CHRONIC LOW BACK PAIN
Brief Title: A Phase 3 Study of Tanezumab for Chronic Low Back Pain
Acronym: TANGO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A4091059; 2012-005495-34 (EudraCT Number); CLBP SC STUDY (Other: Alias Study Number); A4091059 (Other: Pfizer); TANGO (Other: Alias Study Number)
Record Dates: First submitted 2015-08-11; First posted 2015-08-19 (Estimated); Results first posted 2020-02-21 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Low Back Pain
Keywords: Chronic low back pain; Chronic pain
MeSH Terms: conditions — Low Back Pain; Chronic Pain | interventions — tanezumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Placebo to Week 16; tanezumab 5 mg SC (Placebo Comparator)
  Interventions: Biological: Placebo to Week 16; tanezumab 5mg SC
- Placebo to Week 16, tanezumab 10 mg SC (Placebo Comparator)
  Interventions: Biological: Placebo to Week 16, tanezumab 10 mg SC
- Tanezumab 5 mg SC (Experimental)
  Interventions: Biological: Tanezumab 5 mg SC
- Tanezumab 10 mg SC (Experimental)
  Interventions: Biological: Tanezumab 10 mg SC
- Tramadol PR oral (Active Comparator)
  Interventions: Biological: Tramadol PR oral

INTERVENTIONS:
Biological: Placebo to Week 16; tanezumab 5mg SC — Placebo SC injection every 8 weeks for 2 injections followed by tanezumab 5 mg injection every 8 weeks for 5 injections
  Arms: Placebo to Week 16; tanezumab 5 mg SC
Biological: Placebo to Week 16, tanezumab 10 mg SC — Placebo SC injection every 8 weeks for 2 injections, followed by tanezumab 10 mg SC injection for 5 injections
  Arms: Placebo to Week 16, tanezumab 10 mg SC
Biological: Tanezumab 5 mg SC — Tanezumab 5 mg SC
  Arms: Tanezumab 5 mg SC
Biological: Tanezumab 10 mg SC — Tanezumab 10 mg SC
  Arms: Tanezumab 10 mg SC
Biological: Tramadol PR oral — Tramadol PR oral
  Arms: Tramadol PR oral

SUMMARY:
This study will investigate the efficacy and safety of tanezumab 5 mg and 10 mg administered by subcutaneous injection seven times at 8 week intervals (56 weeks). The primary objective of this study is to evaluate the effectiveness of tanezumab 10 mg and 5 mg compared to placebo for the treatment of chronic low back pain. Secondary objectives are to evaluate the long-term safety and effectiveness of tanezumab 10 mg and 5 mg compared to placebo for the treatment of chronic low back pain. In addition, the study will evaluate the effectiveness and long term safety profile of tanezumab treatment for chronic low back pain compared to tramadol Prolonged Release (PR), a medication commonly utilized for the treatment of chronic low back pain.

DETAILED DESCRIPTION:
This is a randomized, double blind, placebo and active controlled, multicenter, parallel group Phase 3 study of the efficacy and safety of tanezumab when administered by SC injection for up to 56 weeks in subjects with chronic low back pain. Approximately 1800 subjects will be randomized to 1 of 4 treatment groups in a 2:2:2:3 ratio (ie, 400 subjects per treatment group for the placebo, tanezumab 5 mg and tanezumab 10 mg treatment groups and 600 subjects in the tramadol PR treatment group). Treatment groups will include: 1.) Placebo administered SC at an 8 week interval plus placebo matching tramadol PR up to Week 16. At the Week 16 visit, subjects in this group who meet the efficacy responder criteria will be switched in a blinded fashion in a 1:1 ratio to either tanezumab 5 mg or tanezumab 10 mg administered SC at an 8 week interval plus placebo matching tramadol PR to Week 56; 2.)Tanezumab 5 mg SC administered at an 8 week interval plus placebo matching tramadol PR to Week 56; 3.) Tanezumab 10 mg SC administered at an 8 week interval plus placebo matching tramadol PR to Week 56; 4.) Oral tramadol PR plus placebo administered SC at an 8 week interval to Week 56. The study is designed with a total duration (post randomization) of up to 80 weeks and will consist of three periods: Screening (up to a maximum of 37 days; includes a Washout Period and an Initial Pain Assessment Period), a Double blind Treatment Period (comprised of a 16 week Primary Efficacy Phase and a 40 week Long Term Safety and Efficacy Phase), and a Follow up Period (24 weeks). The Screening Period (beginning up to 37 days prior to Randomization) includes a Washout Period (lasting 2 32 days), if required, and an Initial Pain Assessment Period (the 5 days prior to Randomization/Baseline). Prior to entering the study, subjects must have a documented history of previous inadequate treatment response to medications in 3 different categories of agents commonly used to treat and generally considered effective for the treatment of chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

-Chronic low back pain ≥3 months in duration, Quebec Task Force in Spinal Disorders class 1 or 2, with documented history of previous inadequate treatment response to at least 3 different categories of agents commonly used and generally considered effective for the treatment of chronic low back pain.

Exclusion Criteria:

--Diagnosis of osteoarthritis of the knee or hip as defined by the American College of Rheumatology (ACR) criteria.

* Subjects who have Kellgren Lawrence Grade > or =2 radiographic evidence of hip or Grade > or=3 radiographic evidence of knee osteoarthritis will be excluded;
* History or radiographic evidence of other diseases that could confound efficacy or safety assessments (e.g., rheumatoid arthritis).
* History or radiographic evidence of orthopedic conditions that may increase the risk of, or confound assessment of joint safety conditions during the study.
* Signs and symptoms of clinically significant cardiac disease within 6 months of the study (e.g., unstable angina, myocardial infarction, resting bradycardia, poorly controlled or untreated hypertension) as defined in the protocol or subjects with any other cardiovascular illness that in the opinion of the Investigator would render a subject unsuitable to participate in the study
* History, diagnosis, or signs and symptoms of clinically significant neurological disease (e.g., transient ischemic attack, stroke, peripheral or autonomic neuropathy) as specified in the protocol
* Subjects with evidence or symptoms consistent with autonomic dysfunction (e.g., orthostatic hypotension and/or autonomic symptoms) as defined in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1832 (Actual)
Dates: Start 2015-08-18 (Actual); Primary Completion 2017-10-17 (Actual); Study Completion 2018-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (262):
- United States (179):
  - Central Alabama Research, Birmingham, Alabama
  - Cahaba Research, Birmingham, Alabama
  - Alabama Clinical Research, LLC, Mobile, Alabama
  - Alabama Orthopaedic Clinic, P.C., Mobile, Alabama
  - Coastal Clinical Research, Mobile, Alabama
  - Horizon Research Partners, LLC, Mobile, Alabama
  - The Center for Clinical Trials, Inc., Saraland, Alabama
  - Ferguson Family Medicine, Mesa, Arizona
  - The Pain Center of Arizona, Phoenix, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - Valley Pain Consultants, Scottsdale, Arizona
  - KLR Business Group dba Arkansas Clinical Research, Little Rock, Arkansas
  - Lynn Institute of the Ozarks, Little Rock, Arkansas
  - Primary Care of Arkansas, P.A., Little Rock, Arkansas
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Core Healthcare Group, Cerritos, California
  - eStudySite, Chula Vista, California
  - Triwest Research Associates, LLC, El Cajon, California
  - Research Center of Fresno, Inc., Fresno, California
  - Neuro-Pain Medical Center, Fresno, California
  - Valley Research-Trials, Fresno, California
  - Collaborative Neuroscience Network, LLC., Garden Grove, California
  - eStudySite, La Mesa, California
  - Collaborative Neuroscience Network, LLC., Long Beach, California
  - University of Southern California, Los Angeles, California
  - USC IDS Pharmacy, Los Angeles, California
  - Catalina Research Institute, LLC, Montclair, California
  - Providence Clinical Research, North Hollywood, California
  - Northern California Research, Sacramento, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Encompass Clinical Research, Spring Valley, California
  - Bayview Research Group, Valley Village, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Elite Clinical Trials, Inc., Wildomar, California
  - Alpine Clinical Research Center, Boulder, Colorado
  - Mountain View Clinical Research, Inc., Denver, Colorado
  - Mountain View Clinical Research, Inc, Denver, Colorado
  - New England Research Associates, LLC, Bridgeport, Connecticut
  - My Health 1st Urgent Care, Milford, Connecticut
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - JEM Research Institute, Atlantis, Florida
  - Orthopedic Research Institute, Boynton Beach, Florida
  - Clinical Research of South Florida, Coral Gables, Florida
  - Avail Clinical Research,LLC, DeLand, Florida
  - Midland Florida Clinical Research Center, LLC, DeLand, Florida
  - S&W Clinical Research, Fort Lauderdale, Florida
  - MD Clinical, Hallandale, Florida
  - Pines Clinical Research Inc., Hollywood, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Health Awareness, Inc., Jupiter, Florida
  - Columbus Clinical Services, LLC, Miami, Florida
  - Larkin Imaging Center, Miami, Florida
  - M & M Medical Center, Inc, Miami, Florida
  - Quality Research & Medical Center LLC, Miami, Florida
  - Crystal Biomedical Research, LLC, Miami Lakes, Florida
  - Sensible Healthcare, LLC., Ocoee, Florida
  - Compass Research, LLC, Orlando, Florida
  - National Pain Research Institute, Orlando, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Gulfcoast Research Institute, Sarasota, Florida
  - Meridien Research, St. Petersburg, Florida
  - Meridien Research, Tampa, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - River Birch Research Alliance, LLC, Blue Ridge, Georgia
  - Columbus Regional Research Institute, Columbus, Georgia
  - Center for Advanced Research & Education, Gainesville, Georgia
  - Drug Studies America, Marietta, Georgia
  - Georgia Institute for Clinical Research, LLC, Marietta, Georgia
  - Non-Surgical Orthopaedics, P.C., Marietta, Georgia
  - Better Health Clinical Research Inc, Newnan, Georgia
  - Better Health Clinical Research, Inc., Newnan, Georgia
  - Southeast Regional Research Group, Savannah, Georgia
  - North Georgia Clinical Research, Woodstock, Georgia
  - North Georgia Internal Medicine, Woodstock, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Medex Healthcare Research Inc, Chicago, Illinois
  - Chicago Clinical Research Institute, Inc., Chicago, Illinois
  - Northwestern Memorial Hospital - Arkes Pavilion, Diagnostic Testing Center, Chicago, Illinois
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Northwestern University, Feinberg School of Medicine, Lavin Pavilion, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Chicago Anesthesia Pain Specialists, Chicago, Illinois
  - Clinical Investigation Specialists, Inc., Skokie, Illinois
  - Investigators Research Group, LLC, Brownsburg, Indiana
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - Lafayette Clinical Research Group, Lafayette, Indiana
  - Lafayette Regional Vein and Laser Center, Lafayette, Indiana
  - Buynak Clinical Research, P.C., Valparaiso, Indiana
  - The Iowa Clinic - Internal Medicine, Des Moines, Iowa
  - The Iowa Clinic Medical Imaging, Des Moines, Iowa
  - The Iowa Clinic, Des Moines, Iowa
  - The Iowa Clinic Medical Imaging, West Des Moines, Iowa
  - The Iowa Clinic, West Des Moines, Iowa
  - Mid-America Physiatrists, P.A., Overland Park, Kansas
  - Professional Research Network of Kansas, LLC, Wichita, Kansas
  - Mayfield Imaging Center, Crestview Hills, Kentucky
  - Otri-Med Corporation, Edgewood, Kentucky
  - St Elizabeth Hospital Edgewood, Edgewood, Kentucky
  - Willis-Knighton Physician Network/ Spine and Pain Specialist, Bossier City, Louisiana
  - Willis-Knighton Physician Network/WKB Family Medicine Associates, Bossier City, Louisiana
  - Centex Studies, Inc, Lake Charles, Louisiana
  - Best Clinical Trials, LLC, New Orleans, Louisiana
  - George Stanley Walker, MD, New Orleans, Louisiana
  - Klein & Associates, M.D., P.A., Cumberland, Maryland
  - The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Chestnut Hill, Massachusetts
  - Beacon Clinical Research, LLC, Quincy, Massachusetts
  - MedVadis Research Corporation, Watertown, Massachusetts
  - Great Lakes Research Group, Inc., Bay City, Michigan
  - Michigan Orthopaedic Spine Surgeons, Rochester Hills, Michigan
  - Oakland Medical Research, Troy, Michigan
  - Michigan Pain Consultants, Wyoming, Michigan
  - CRC of Jackson, LLC, Jackson, Mississippi
  - Physician's Surgery Center, Jackson, Mississippi
  - Olive Branch Family Medical Center, Olive Branch, Mississippi
  - Medex Healthcare Research, Inc., St Louis, Missouri
  - Heartland Clinical Research, Inc., Omaha, Nebraska
  - Affiliated Clinical Research, Inc., Las Vegas, Nevada
  - Office of Stephen H. Miller, MD, Las Vegas, Nevada
  - Office of Robert Kaplan, DO, Las Vegas, Nevada
  - Advanced Biomedical Research of America, Las Vegas, Nevada
  - ActivMed Practices & Research, Inc., Portsmouth, New Hampshire
  - Comprehensive Clinical Research, Berlin, New Jersey
  - CRI Worldwide, LLC, Marlton, New Jersey
  - University Clinical Research Center, Somerset, New Jersey
  - Premier Research, Trenton, New Jersey
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - New Mexico Clinical Research & Osteoporosis Center, Inc., Albuquerque, New Mexico
  - Healthwise Medical Associates, Brooklyn, New York
  - Drug Trials America, Hartsdale, New York
  - The Medical Research Network, LLC, New York, New York
  - AAIR Research Center, Rochester, New York
  - University of Rochester, Rochester, New York
  - Northstate Clinical Research, Lenoir, North Carolina
  - On Site Clinical Solutions, LLC, Mooresville, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - PMG Research of Winston-Salem, LLC, Winston-Salem, North Carolina
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - Lillestol Research, LLC, Fargo, North Dakota
  - Plains Clinical Research Center, LLC, Fargo, North Dakota
  - Heartland Diagnostics, Frgi, North Dakota
  - Clinical Inquest Center Ltd, Beavercreek, Ohio
  - Valley Medical Research/Valley Medical Primary Care, Centerville, Ohio
  - Hightop Medical Research Center, Cincinnati, Ohio
  - New Horizons Clinical Research, Cincinnati, Ohio
  - Optimed Research LTD, Columbus, Ohio
  - Prestige Clinical Research, Franklin, Ohio
  - Great Lakes Medical Research, LLC, Mentor, Ohio
  - Oaktree Clinic, Mentor, Ohio
  - Bone Joint & Spine Surgeons, Inc., Toledo, Ohio
  - COR Clinical Research, L.L.C, Oklahoma City, Oklahoma
  - Health Research of Oklahoma, Oklahoma City, Oklahoma
  - NPC Research, Oklahoma City, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Brandywine Clinical Research, Downingtown, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - TLM Medical Services, Columbia, South Carolina
  - DeGarmo Institute of Medical Research, Greer, South Carolina
  - Lowcountry Orthopaedics & Sports Medicine, North Charleston, South Carolina
  - Health Concepts, Rapid City, South Dakota
  - PCET Research Center, LLC, Knoxville, Tennessee
  - Quality Medical Research, Nashville, Tennessee
  - KRK Medical Research, Arlington, Texas
  - Advances In Health, Houston, Texas
  - Centex Studies, Inc./Clear Lake Family Physicians, Houston, Texas
  - Clinical Trial Network, Houston, Texas
  - The Pain Relief Center, Plano, Texas
  - Quality Research, Inc., San Antonio, Texas
  - Lee Medical Associates, PA, San Antonio, Texas
  - Progressive Clinical Research, PA, San Antonio, Texas
  - Physicians Research Options, LLC, Draper, Utah
  - Charlottesville Medical Research Center, LLC, Charlottesville, Virginia
  - Virginia Research Center, Midlothian, Virginia
  - National Clinical Research - Richmond, Inc., Richmond, Virginia
  - Washington Center for Pain Management, Bellevue, Washington
  - Northwest Clinical Research Center, Bellevue, Washington
- Canada (5):
  - SKDS Research Inc., Newmarket, Ontario
  - London Road Diagnostic Clinic & Medical Centre, Sarnia, Ontario
  - G.R.M.O. (Groupe de recherche en maladies osseuses) Inc., Québec, Quebec
  - Centre de recherche Saint-Louis, Québec, Quebec
  - Diex Research Sherbrooke Inc., Sherbrooke, Quebec
- A2 reumatologi og idraesmedicin ApS, Hillerød, Denmark
- Hopital Cochin, Paris, France
- Hungary (8):
  - Bekes Megyei Koezponti Korhaz Dr Rethy Pal Tagkorhaz, Békéscsaba
  - Clinexpert Egeszsegugyi Szolgaltato es Kereskedelmi Kft., Budapest
  - Obudai Egeszsegugyi Centrum Ktf., Budapest
  - Jutrix Kft., Kecskemét
  - CRU Hungary Ltd., MISEK HOSPITAL, Miskolc
  - CRU Hungary Ltd., MISEK-Radiology Department, Miskolc
  - Clinfan Kft., Szekszárd
  - Tolna Megyei Balassa Janos Korhaz, Ortopediai osztaly, Szekszárd
- Japan (40):
  - Aichi Medical University Hospital, Nagakute, Aichi-ken
  - Nagoya University Hospital, Showa-ku, Nagoya, Aichi-ken
  - Chiba University Hospital, Chuo-ku, Chiba, Chiba
  - Funabashi Municipal Medical Center, Funabashi, Chiba
  - Chiba Rosai Hospital, Ichihara, Chiba
  - Chiba Central Medical Center, Wakaba-ku, Chiba, Chiba
  - Fukuoka Mirai Hospital, Higashi-ku,Fukuoka, Fukuoka
  - Kyushu Rosai Hospital, Kokuraminami-ku,Kitakyushu, Fukuoka
  - Takagi Hospital, Ōkawa, Fukuoka
  - Fukushima Medical University Aizu Medical Center, Aizu-Wakamatsu, Fukushima
  - Hakodate Central General Hospital, Hakodate, Hokkaido
  - Hakodate Ohmura Orthopedic Hospital, Hakodate, Hokkaido
  - Kobe Konan Yamate Clinic, Higashinada-ku, Kobe, Hyōgo
  - Omuro Orthopedic Clinic, Himeji, Hyōgo
  - Medical corporate corporation hoshikai Onishi medical clinic, Kako-gun, Hyōgo
  - Kobe Red Cross Hospital, Kobe, Hyōgo
  - National Hospital Organization Kanazawa Medical Center, Kanazawa, Ishikawa-ken
  - Morita Hospital, Komatsu, Ishikawa-ken
  - Marunouchi Hospital, Matsumoto, Nagano
  - National Hospital Organization Beppu Medical Center, Beppu, Oita Prefecture
  - Sobajima Clinic, Higashiosaka, Osaka
  - Rinku General Medical Center, Izumisano, Osaka
  - Minamiosaka Hospital, Suminoe-ku, Osaka, Osaka
  - Saitama Jikei Hospital, Kumagaya, Saitama
  - Hamamatsu University School of Medicine, University Hospital, Hamamatsu, Shizuoka
  - Tokyo Medical and Dental University Medical Hospital, Bunkyo-ku, Tokyo
  - Fussa Hospital, Fussa, Tokyo
  - Tokyo Saiseikai Central Hospital, Minato-ku, Tokyo
  - Kohno Clinical Medicine Research Institute Daisan Kitashinagawa Hospital, Shinagawa-ku, Tokyo
  - Ohimachi Orthopaedic Clinic, Shinagawa-ku, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - Yonezawa City Hospital, Yonezawa, Yamagata
  - Shimonoseki City Hospital, Shimonoseki-shi, Yamaguchi
  - Yamaguchi University Hospital, Ube, Yamaguchi
  - Chihaya Hospital, Fukuoka
  - Kuroda Orthopedic Hospital, Fukuoka
  - Fukushima Medical University Hospital, Fukushima
  - Hiroshima Red Cross Hospital & Atomic-bomb Survivors Hospital, Hiroshima
  - Saitama Municipal Hospital, Saitama
  - Toyama University Hospital, Toyama
- South Korea (6):
  - CTC Pharmacy, Seoul National University Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - CTC Pharmacy, Severance Hospital, Seoul
  - Severance Hospital, Seoul
  - Clinical Trial Pharmacy, Samsung Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (18):
  - Hospital Nuestra Senora de la Esperanza, Santiago de Compostela, A Coruna
  - Complejo Hospitalario Universitario A Coruna. Servicio de Farmacia, A Coruña
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Instituto de Ciencias Medicas, Alicante
  - Hospital de Mar Servicio de Radiologia, Barcelona
  - Hospital del Mar Servicio de Farmacia, Barcelona
  - Specialist, S.L., Barcelona
  - Specialist. Farmacia, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Universitario Quiron-Dexeus, Barcelona
  - Hospital Universitario Quiron-Dexeus. Servicio de Farmacia, Barcelona
  - Hospital Sanitas CIMA, Barcelona
  - Hospital Universitario La Paz., Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital La Moraleja. Pharmacy Service, Madrid
  - Hospital La Moraleja, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Regional Universitario del Malaga, Málaga
- Sweden (4):
  - CTC (Clinical Trial Center) Sahlgrenska University Hospital, Gothenburg
  - Pharmasite, Helsingborg
  - Pharmasite, Malmo
  - ProbarE i Stockholm AB, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Markman JD, Schnitzer TJ, Perrot S, Beydoun SR, Ohtori S, Viktrup L, Yang R, Bramson C, West CR, Verburg KM. Clinical Meaningfulness of Response to Tanezumab in Patients with Chronic Low Back Pain: Analysis From a 56-Week, Randomized, Placebo- and Tramadol-Controlled, Phase 3 Trial. Pain Ther. 2022 Dec;11(4):1267-1285. doi: 10.1007/s40122-022-00424-7. Epub 2022 Aug 13. PMID 35962939
- [Derived] Markman JD, Bolash RB, McAlindon TE, Kivitz AJ, Pombo-Suarez M, Ohtori S, Roemer FW, Li DJ, Viktrup L, Bramson C, West CR, Verburg KM. Tanezumab for chronic low back pain: a randomized, double-blind, placebo- and active-controlled, phase 3 study of efficacy and safety. Pain. 2020 Sep 1;161(9):2068-2078. doi: 10.1097/j.pain.0000000000001928. PMID 32453139
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4091059

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1832 participants were enrolled in the study, however, only those participants were included in participant flow section who received at least 1 dose of study drug.
Pre-assignment Details: Treatment period was up to Week 56. Safety follow up period started at Week 64, thus Weeks 64 and 80 time points were during safety follow up period. Percentage (%) reduction in low back pain intensity (LBPI) and participants global assessment (PGA) 2-point reduction are efficacy measures and not applicable during safety follow up.
Groups:
- Placebo Followed by Tanezumab 5 mg: Placebo matched to tanezumab (RN624 or PF-04383119) injection administered subcutaneously (SC) once every 8 weeks and placebo tablets matched to tramadol prolonged release (PR), orally, once daily from Day 1 (baseline) up to week 16. At week 16, participants who met efficacy responder criteria (greater than equal to [>=] 30 percent [%] reduction in average LBPI score and >=15% reduction in average LBPI score relative to baseline at any week from week 1 to week 15), then received tanezumab 5 milligram (mg), SC, once every 8 weeks plus placebo tablets matched to tramadol PR, orally, once daily from week 16 to week 56.
- Placebo Followed by Tanezumab 10 mg: Placebo matched to tanezumab (RN624 or PF-04383119) injection administered SC, once every 8 weeks and placebo tablets matched to tramadol PR, orally, once daily from Day 1 (baseline) up to week 16. At week 16, participants who met efficacy responder criteria, then received tanezumab 10 mg, SC, once every 8 weeks plus placebo tablets matched to tramadol PR, orally, once daily from week 16 to week 56.
- Pooled Tanezumab 5 mg: Tanezumab (RN624 or PF-04383119) 5 mg injection administered SC once every 8 weeks and placebo tablets matched to tramadol PR, orally, once daily from Day 1 up to week 56.
- Pooled Tanezumab 10 mg: Tanezumab (RN624 or PF-04383119) 10 mg injection administered SC once every 8 weeks and placebo tablets matched to tramadol PR, orally, once daily from Day 1 up to week 56.
- Tramadol: Tramadol PR tablet of 100 mg (during baseline to week 4, dose increments by 100 mg was allowed up to a maximum of 300 mg, depending on pain relief or tolerability), once daily and placebo injection matched to tramadol, administered SC once every 8 weeks, from Day 1 up to week 56.
Period: Overall Study
Arm/Group | Placebo Followed by Tanezumab 5 mg | Placebo Followed by Tanezumab 10 mg | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Started | 205 | 204 | 407 | 407 | 602
Intent to Treat Population | 202 | 204 | 407 | 407 | 605 (3 participants randomized to placebo arm received tramadol during the course of study)
Treated at Week 16 | 99 | 95 | 236 | 242 | 307
Completed | 130 | 134 | 267 | 271 | 379
Not Completed | 75 | 70 | 140 | 136 | 223
Not completed — Adverse Event | 3 | 4 | 4 | 8 | 18
Not completed — Death | 2 | 2 | 1 | 0 | 1
Not completed — Insufficient clinical response | 7 | 10 | 13 | 12 | 16
Not completed — Lost to Follow-up | 16 | 9 | 31 | 16 | 34
Not completed — Other | 21 | 22 | 58 | 52 | 76
Not completed — Withdrawal by Subject | 25 | 20 | 29 | 48 | 73
Not completed — Protocol Violation | 1 | 2 | 4 | 0 | 4
Not completed — Withdrawn Due to Pregnancy | 0 | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The safety population was defined as all participants treated with tanezumab or placebo SC.
Groups:
- Placebo Followed by Tanezumab 5 mg: Placebo matched to tanezumab (RN624 or PF-04383119) injection administered SC once every 8 weeks and placebo tablets matched to tramadol PR, orally, once daily from Day 1 (baseline) up to week 16. At week 16, participants who met efficacy responder criteria >=30 percent [%] reduction in average LBPI score and >=15% reduction in average LBPI score relative to baseline at any week from week 1 to week 15), then received tanezumab 5 milligram (mg), SC, once every 8 weeks plus placebo tablets matched to tramadol PR, orally, once daily from week 16 to week 56.
- Total: Total of all reporting groups
Arm/Group | Placebo Followed by Tanezumab 5 mg | Placebo Followed by Tanezumab 10 mg | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol | Total
Number analyzed (Participants) | 205 | 204 | 407 | 407 | 602 | 1825
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.01 (13.76) | 48.97 (12.00) | 48.66 (12.36) | 49.15 (12.36) | 48.42 (13.08) | 48.77 (12.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123 | 113 | 248 | 218 | 339 | 1041
  Male | 82 | 91 | 159 | 189 | 263 | 784
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 154 | 142 | 295 | 303 | 428 | 1322
  Black or African American | 35 | 35 | 65 | 66 | 102 | 303
  Asian | 13 | 25 | 39 | 28 | 65 | 170
  Other | 3 | 2 | 8 | 10 | 7 | 30
  Unknown | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average Low Back Pain Intensity (LBPI) Score for Tanezumab Versus (Vs) Placebo at Week 16
Description: Average low back pain was assessed on an 11-point numeric rating scale (NRS) captured through an interactive response technology (IRT). Participants described their average low back pain during the past 24 hours on a scale ranging from 0 (no pain) to 10 (worst possible pain), where higher scores indicated higher pain.
Time Frame: Baseline, Week 16
Population: ITT population:randomized participants who received at least 1 dose of SC study medication(either tanezumab or matching placebo).Pre-specified intent of study for efficacy data up to W16 was to analyze participants who received placebo from Day1 and then received tanezumab 5/10 mg at W16,together,in placebo arm.Data has been reported per four arms.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Placebo: Placebo matched to tanezumab (RN624 or PF-04383119) injection administered SC, once every 8 weeks from Day 1 (baseline), and placebo tablets matched to tramadol PR, orally, once daily from Day 1 up to Week 16. At Week 16, participants who met efficacy responder criteria (30 percent % reduction in average (LBPI) score and >=15% reduction in average LBPI score relative to baseline at any week from week 1 to week 15), then received tanezumab 5 mg or 10 mg, SC, once every 8 weeks plus placebo tablets matched to tramadol PR, orally, once daily from week 16 to week 56.
- Pooled Tanezumab 5 mg: Tanezumab (RN624 or PF-04383119) 5 mg injection administered SC once every 8 weeks from Day 1 and placebo tablets matched to tramadol PR, orally, once daily from Day 1 up to week 56.
- Pooled Tanezumab 10 mg: Tanezumab (RN624 or PF-04383119) 10 mg injection administered SC once every 8 weeks from Day 1, and placebo tablets matched to tramadol PR, orally, once daily from Day 1 up to week 56.
Arm/Group | Placebo | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 406 | 407 | 407 | 605
units on a scale | -2.68 (0.15) | -2.98 (0.14) | -3.08 (0.14) | -2.81 (0.12)
Statistical Analysis 1: Comparison: Placebo vs Pooled Tanezumab 5 mg; Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. Analysis of covariance (ANCOVA) model for imputed datasets included treatment as a fixed effect, and baseline LBPI as a covariates, and study site as a random effect; Test type: Superiority; p = 0.1117, ANCOVA; Least Square (LS) Mean Difference = -0.30, 95% CI 2-sided [-0.66 to 0.07], Standard Error of Mean 0.19
Statistical Analysis 2: Comparison: Placebo vs Pooled Tanezumab 10 mg; Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as a fixed effect, and baseline LBPI as a covariates, and study site as a random effect; Test type: Superiority; p = 0.0281, ANCOVA; LS Mean Difference = -0.40, 95% CI 2-sided [-0.76 to -0.04], Standard Error of Mean 0.18

2. Secondary Outcome: Change From Baseline in Roland Morris Disability Questionnaire (RMDQ) at Week 16 for Tanezumab Versus (Vs) Placebo
Description: The RMDQ is a self-administered, widely used health status measure index of how well participants with low back pain (LBP) are able to function with regard to daily activities. It measures pain and function, using 24 items describing limitations to everyday life that can be caused by LBP. The total score of the RMDQ from the total number of items checked ranged from 0 (no disability) to 24 (maximum disability), where higher scores indicated greater disability.
Time Frame: Baseline, Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 406 | 407 | 407 | 605
units on a scale | -4.95 (0.36) | -6.27 (0.35) | -6.69 (0.35) | -5.21 (0.30)
Statistical Analysis 1: Comparison: Placebo vs Pooled Tanezumab 5 mg; Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline RMDQ, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.0035, ANCOVA; LS Mean Difference = -1.32, 95% CI 2-sided [-2.21 to -0.43], Standard Error of Mean 0.45
Statistical Analysis 2: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0002, ANCOVA; LS Mean Difference = -1.74, 95% CI 2-sided [-2.64 to -0.83], Standard Error of Mean 0.46

3. Secondary Outcome: Change From Baseline in Average Low Back Pain Intensity (LBPI) Score for Tanezumab Versus (Vs) Tramadol at Week 16
Description: Average LBP was assessed on an 11-point NRS captured through an IRT. Participants described their average LBP during the past 24 hours on a scale ranging from 0 (no pain) to 10 (worst possible pain), where higher scores indicated higher pain.
Time Frame: Baseline, Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 406 | 407 | 407 | 605
units on a scale | -2.68 (0.15) | -2.98 (0.14) | -3.08 (0.14) | -2.81 (0.12)
Statistical Analysis 1: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as a fixed effect, and baseline average LBPI as a covariates, and study site as a random effect; Test type: Superiority; p = 0.3118, ANCOVA; LS Mean Difference = -0.17, 95% CI 2-sided [-0.50 to 0.16], Standard Error of Mean 0.17
Statistical Analysis 2: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0958, ANCOVA; LS Mean Difference = -0.28, 95% CI 2-sided [-0.60 to 0.05], Standard Error of Mean 0.17

4. Secondary Outcome: Change From Baseline in Average Low Back Pain Intensity (LBPI) Score at Weeks 2, 4, 8, 12, 24, 32, 40, 48 and 56
Description: Average LBP was assessed on an 11-point NRS captured through an IRT. The LBPI score was captured once daily from baseline up to week 16, and once weekly from week 16 to week 64. Participants described their average LBP during the past 24 hours on a scale ranging from 0 (no pain) to 10 (worst possible pain), where higher scores indicated higher pain. Pre-specified intent of study for efficacy data up to W16 was to analyze participants who received placebo from Day1 and then received tanezumab 5/10 mg at W16,together,in placebo arm.Data has been reported per four arms.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 24, 32, 40, 48 and 56
Population: ITT population.Data were not collected after W16 in placebo arm for this outcome measure, as those who met criteria to continue, switched to active treatment with tanezumab after W16.Pre-specified intent of study was to compare tanezumab Vs placebo for data up to & including W16 & comparisons of tanezumab Vs tramadol for data up to & including W56.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 406 | 407 | 407 | 605
units on a scale
  Change at Week 2 | -1.17 (0.09) | -1.54 (0.09) | -1.59 (0.09) | -1.36 (0.08)
  Change at Week 4 | -1.75 (0.12) | -2.24 (0.12) | -2.43 (0.12) | -1.99 (0.10)
  Change at Week 8 | -2.10 (0.13) | -2.64 (0.13) | -2.79 (0.13) | -2.43 (0.11)
  Change at Week 12 | -2.54 (0.13) | -2.92 (0.13) | -3.12 (0.13) | -2.74 (0.11)
  Change at Week 24: number analyzed (Participants) | 0 | 407 | 407 | 605
  Change at Week 24 |  | -2.76 (0.16) | -2.92 (0.16) | -2.64 (0.14)
  Change at Week 32: number analyzed (Participants) | 0 | 407 | 407 | 605
  Change at Week 32 |  | -2.74 (0.17) | -2.75 (0.16) | -2.52 (0.14)
  Change at Week 40: number analyzed (Participants) | 0 | 407 | 407 | 605
  Change at Week 40 |  | -2.64 (0.17) | -2.67 (0.17) | -2.49 (0.14)
  Change at Week 48: number analyzed (Participants) | 0 | 407 | 407 | 605
  Change at Week 48 |  | -2.58 (0.17) | -2.62 (0.17) | -2.43 (0.15)
  Change at Week 56: number analyzed (Participants) | 0 | 407 | 407 | 605
  Change at Week 56 |  | -2.52 (0.17) | -2.62 (0.17) | -2.40 (0.15)
Statistical Analysis 1: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 2: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as a fixed effect, and baseline average LBPI as a covariates, and study site as a random effect; Test type: Superiority; p = 0.0015, ANCOVA; LS Mean Difference = -0.37, 95% CI 2-sided [-0.60 to -0.14], Standard Error of Mean 0.12
Statistical Analysis 2: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0004, ANCOVA; LS Mean Difference = -0.42, 95% CI 2-sided [-0.65 to -0.19], Standard Error of Mean 0.12
Statistical Analysis 3: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0959, ANCOVA; LS Mean Difference = -0.18, 95% CI 2-sided [-0.39 to 0.03], Standard Error of Mean 0.11
Statistical Analysis 4: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0370, ANCOVA; LS Mean Difference = -0.23, 95% CI 2-sided [-0.44 to -0.01], Standard Error of Mean 0.11
Statistical Analysis 5: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 4: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as a fixed effect, and baseline average LBPI as a covariates, and study site as a random effect; Test type: Superiority; p = 0.0008, ANCOVA; LS Mean Difference = -0.48, 95% CI 2-sided [-0.76 to -0.20], Standard Error of Mean 0.14
Statistical Analysis 6: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 4, analysis 5]; Test type: Superiority; p < .0001, ANCOVA; LS Mean Difference = -0.68, 95% CI 2-sided [-0.96 to -0.39], Standard Error of Mean 0.14
Statistical Analysis 7: Comparison: Placebo vs Tramadol; [analysis description as in outcome 4, analysis 5]; Test type: Superiority; p = 0.0711, ANCOVA; LS Mean Difference = -0.24, 95% CI 2-sided [-0.50 to 0.02], Standard Error of Mean 0.13
Statistical Analysis 8: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 4, analysis 5]; Test type: Superiority; p = 0.0661, ANCOVA; LS Mean Difference = -0.24, 95% CI 2-sided [-0.50 to 0.02], Standard Error of Mean 0.13
Statistical Analysis 9: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 4, analysis 5]; Test type: Superiority; p = 0.0009, ANCOVA; LS Mean Difference = -0.44, 95% CI 2-sided [-0.70 to -0.18], Standard Error of Mean 0.13
Statistical Analysis 10: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 8: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as a fixed effect, and baseline average LBPI as a covariates, and study site as a random effect; Test type: Superiority; p = 0.0008, ANCOVA; LS Mean Difference = -0.53, 95% CI 2-sided [-0.84 to -0.22], Standard Error of Mean 0.16
Statistical Analysis 11: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 4, analysis 10]; Test type: Superiority; p < .0001, ANCOVA; LS Mean Difference = -0.69, 95% CI 2-sided [-1.00 to -0.38], Standard Error of Mean 0.16
Statistical Analysis 12: Comparison: Placebo vs Tramadol; [analysis description as in outcome 4, analysis 10]; Test type: Superiority; p = 0.0274, ANCOVA; LS Mean Difference = -0.32, 95% CI 2-sided [-0.61 to -0.04], Standard Error of Mean 0.15
Statistical Analysis 13: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 4, analysis 10]; Test type: Superiority; p = 0.1495, ANCOVA; LS Mean Difference = -0.21, 95% CI 2-sided [-0.50 to 0.08], Standard Error of Mean 0.15
Statistical Analysis 14: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 4, analysis 10]; Test type: Superiority; p = 0.0123, ANCOVA; LS Mean Difference = -0.37, 95% CI 2-sided [-0.65 to -0.08], Standard Error of Mean 0.15
Statistical Analysis 15: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 12: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as a fixed effect, and baseline average LBPI as a covariates, and study site as a random effect; Test type: Superiority; p = 0.0307, ANCOVA; LS Mean Difference = -0.37, 95% CI 2-sided [-0.71 to -0.03], Standard Error of Mean 0.17
Statistical Analysis 16: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 4, analysis 15]; Test type: Superiority; p = 0.0009, ANCOVA; LS Mean Difference = -0.58, 95% CI 2-sided [-0.91 to -0.24], Standard Error of Mean 0.17
Statistical Analysis 17: Comparison: Placebo vs Tramadol; [analysis description as in outcome 4, analysis 15]; Test type: Superiority; p = 0.2103, ANCOVA; LS Mean Difference = -0.20, 95% CI 2-sided [-0.51 to 0.11], Standard Error of Mean 0.16
Statistical Analysis 18: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 4, analysis 15]; Test type: Superiority; p = 0.2656, ANCOVA; LS Mean Difference = -0.18, 95% CI 2-sided [-0.48 to 0.13], Standard Error of Mean 0.16
Statistical Analysis 19: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 4, analysis 15]; Test type: Superiority; p = 0.0152, ANCOVA; LS Mean Difference = -0.38, 95% CI 2-sided [-0.68 to -0.07], Standard Error of Mean 0.16
Statistical Analysis 20: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 24: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as a fixed effect, and baseline average LBPI as a covariates, and study site as a random effect; Test type: Superiority; p = 0.5164, ANCOVA; LS Mean Difference = -0.12, 95% CI 2-sided [-0.50 to 0.25], Standard Error of Mean 0.19
Statistical Analysis 21: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 4, analysis 20]; Test type: Superiority; p = 0.1488, ANCOVA; LS Mean Difference = -0.28, 95% CI 2-sided [-0.66 to 0.10], Standard Error of Mean 0.19
Statistical Analysis 22: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 32: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as a fixed effect, and baseline average LBPI as a covariates, and study site as a random effect; Test type: Superiority; p = 0.2431, ANCOVA; LS Mean Difference = -0.22, 95% CI 2-sided [-0.60 to 0.15], Standard Error of Mean 0.19
Statistical Analysis 23: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 4, analysis 22]; Test type: Superiority; p = 0.2428, ANCOVA; LS Mean Difference = -0.23, 95% CI 2-sided [-0.62 to 0.16], Standard Error of Mean 0.20
Statistical Analysis 24: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 40: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as a fixed effect, and baseline average LBPI as a covariates, and study site as a random effect; Test type: Superiority; p = 0.4561, ANCOVA; LS Mean Difference = -0.15, 95% CI 2-sided [-0.54 to 0.24], Standard Error of Mean 0.20
Statistical Analysis 25: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 4, analysis 24]; Test type: Superiority; p = 0.3523, ANCOVA; LS Mean Difference = -0.18, 95% CI 2-sided [-0.56 to 0.20], Standard Error of Mean 0.20
Statistical Analysis 26: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 48: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as a fixed effect, and baseline average LBPI as a covariates, and study site as a random effect; Test type: Superiority; p = 0.4403, ANCOVA; LS Mean Difference = -0.15, 95% CI 2-sided [-0.53 to 0.23], Standard Error of Mean 0.20
Statistical Analysis 27: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 4, analysis 26]; Test type: Superiority; p = 0.3205, ANCOVA; LS Mean Difference = -0.20, 95% CI 2-sided [-0.58 to 0.19], Standard Error of Mean 0.20
Statistical Analysis 28: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 56: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as a fixed effect, and baseline average LBPI as a covariates, and study site as a random effect; Test type: Superiority; p = 0.5763, ANCOVA; LS Mean Difference = -0.11, 95% CI 2-sided [-0.51 to 0.28], Standard Error of Mean 0.20
Statistical Analysis 29: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 4, analysis 28]; Test type: Superiority; p = 0.2887, ANCOVA; LS Mean Difference = -0.21, 95% CI 2-sided [-0.61 to 0.18], Standard Error of Mean 0.20

5. Secondary Outcome: Change From Baseline in Daily Average Low Back Pain Intensity (LBPI) Score at Week 64
Description: Average LBP was assessed on an 11-point NRS captured through an IRT. The LBPI score was captured once a week for week 64. Participants described their average LBP during the past 24 hours on a scale ranging from 0 (no pain) to 10 (worst possible pain), where higher scores indicated higher pain.
Time Frame: Baseline, Week 64
Population: ITT population included all randomized participants who received at least one dose of SC study medication (either tanezumab or matching placebo). 'Number analyzed' (n)= participants evaluable for this outcome measure (OM) at specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Followed by Tanezumab 5 mg | Placebo Followed by Tanezumab 10 mg | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 202 | 204 | 407 | 407 | 605
units on a scale
  Baseline: number analyzed (Participants) | 200 | 204 | 406 | 406 | 605
  Baseline | 7.16 (1.15) | 7.23 (1.09) | 7.25 (1.08) | 7.18 (1.13) | 7.17 (1.16)
  Change at Week 64: number analyzed (Participants) | 58 | 53 | 126 | 145 | 176
  Change at Week 64 | -4.36 (2.28) | -4.32 (2.01) | -4.04 (2.15) | -3.71 (2.39) | -4.08 (2.12)

6. Secondary Outcome: Change From Baseline in Roland Morris Disability Questionnaire (RMDQ) Total Score at Weeks 2, 4, 8, 16 (for Tanezumab vs Tramadol) 24, 32, 40, 48 and 56
Description: The RMDQ is a self-administered, widely used health status measure index of how well participants with LBP are able to function with regard to daily activities. It measures pain and function, using 24 items describing limitations to everyday life that can be caused by LBP. The total score of the RMDQ is the total number of items checked ranging from 0 (no disability) to 24 (maximum disability), where higher scores indicated greater disability. Pre-specified intent of study for efficacy data up to W16 was to analyze participants who received placebo from Day1 and then received tanezumab 5/10 mg at W16,together,in placebo arm.Data has been reported per four arms.
Time Frame: Baseline, Weeks 2, 4, 8, 16, 24, 32, 40, 48 and 56
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Placebo: Placebo matched to tanezumab (RN624 or PF-04383119) injection administered SC once every 8 weeks from Day 1 (baseline), and placebo tablets matched to tramadol PR, orally, once daily from Day 1 up to week 16. At week 16, participants who met efficacy responder criteria (>=30 percentage % reduction in average LBPI score and >=15% reduction in average LBPI score relative to baseline at any week from week 1 to week 15), then received tanezumab 5 mg or 10 mg, SC, once every 8 weeks plus placebo tablets matched to tramadol PR, orally, once daily from week 16 to week 56.
Arm/Group | Placebo | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 406 | 407 | 407 | 605
units on a scale
  Change at Week 2 | -2.46 (0.26) | -3.30 (0.25) | -3.84 (0.26) | -2.74 (0.21)
  Change at Week 4 | -3.37 (0.29) | -4.58 (0.29) | -5.32 (0.29) | -3.67 (0.25)
  Change at Week 8 | -3.90 (0.31) | -5.27 (0.31) | -5.85 (0.31) | -4.51 (0.27)
  Change at Week 16 | -4.95 (0.36) | -6.27 (0.35) | -6.69 (0.35) | -5.21 (0.30)
  Change at Week 24: number analyzed (Participants) | 0 | 407 | 407 | 605
  Change at Week 24 |  | -5.57 (0.41) | -5.92 (0.41) | -4.59 (0.35)
  Change at Week 32: number analyzed (Participants) | 0 | 407 | 407 | 605
  Change at Week 32 |  | -5.46 (0.42) | -5.71 (0.42) | -4.74 (0.35)
  Change at Week 40: number analyzed (Participants) | 0 | 407 | 407 | 605
  Change at Week 40 |  | -5.12 (0.43) | -5.24 (0.44) | -4.53 (0.36)
  Change at Week 48: number analyzed (Participants) | 0 | 407 | 407 | 605
  Change at Week 48 |  | -4.92 (0.43) | -5.14 (0.43) | -4.44 (0.37)
  Change at Week 56: number analyzed (Participants) | 0 | 407 | 407 | 605
  Change at Week 56 |  | -4.85 (0.45) | -5.23 (0.44) | -4.41 (0.36)
Statistical Analysis 1: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 2: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline RMDQ, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.0121, ANCOVA; LS Mean Difference = -0.84, 95% CI 2-sided [-1.50 to -0.18], Standard Error of Mean 0.34
Statistical Analysis 2: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p < .0001, ANCOVA; LS Mean Difference = -1.38, 95% CI 2-sided [-2.05 to -0.71], Standard Error of Mean 0.34
Statistical Analysis 3: Comparison: Placebo vs Tramadol; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.3697, ANCOVA; LS Mean Difference = -0.28, 95% CI 2-sided [-0.89 to 0.33], Standard Error of Mean 0.31
Statistical Analysis 4: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.0658, ANCOVA; LS Mean Difference = -0.56, 95% CI 2-sided [-1.16 to 0.04], Standard Error of Mean 0.30
Statistical Analysis 5: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.0004, ANCOVA; LS Mean Difference = -1.10, 95% CI 2-sided [-1.70 to -0.50], Standard Error of Mean 0.31
Statistical Analysis 6: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 4: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline RMDQ, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.0013, ANCOVA; LS Mean Difference = -1.22, 95% CI 2-sided [-1.96 to -0.48], Standard Error of Mean 0.38
Statistical Analysis 7: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 6, analysis 6]; Test type: Superiority; p < .0001, ANCOVA; LS Mean Difference = -1.96, 95% CI 2-sided [-2.70 to -1.21], Standard Error of Mean 0.38
Statistical Analysis 8: Comparison: Placebo vs Tramadol; [analysis description as in outcome 6, analysis 6]; Test type: Superiority; p = 0.3906, ANCOVA; LS Mean Difference = -0.30, 95% CI 2-sided [-0.99 to 0.39], Standard Error of Mean 0.35
Statistical Analysis 9: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 6, analysis 6]; Test type: Superiority; p = 0.0082, ANCOVA; LS Mean Difference = -0.92, 95% CI 2-sided [-1.60 to -0.24], Standard Error of Mean 0.35
Statistical Analysis 10: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 6, analysis 6]; Test type: Superiority; p < .0001, ANCOVA; LS Mean Difference = -1.65, 95% CI 2-sided [-2.34 to -0.97], Standard Error of Mean 0.35
Statistical Analysis 11: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 8: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline RMDQ, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.0006, ANCOVA; LS Mean Difference = -1.37, 95% CI 2-sided [-2.15 to -0.58], Standard Error of Mean 0.40
Statistical Analysis 12: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 6, analysis 11]; Test type: Superiority; p < .0001, ANCOVA; LS Mean Difference = -1.95, 95% CI 2-sided [-2.73 to -1.16], Standard Error of Mean 0.40
Statistical Analysis 13: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 6, analysis 11]; Test type: Superiority; p = 0.0385, ANCOVA; LS Mean Difference = -0.76, 95% CI 2-sided [-1.47 to -0.04], Standard Error of Mean 0.37
Statistical Analysis 14: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 6, analysis 11]; Test type: Superiority; p = 0.0003, ANCOVA; LS Mean Difference = -1.34, 95% CI 2-sided [-2.06 to -0.61], Standard Error of Mean 0.37
Statistical Analysis 15: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 16: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline RMDQ, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.0035, ANCOVA; LS Mean Difference = -1.32, 95% CI 2-sided [-2.21 to -0.43], Standard Error of Mean 0.45
Statistical Analysis 16: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 6, analysis 15]; Test type: Superiority; p = 0.0002, ANCOVA; LS Mean Difference = -1.74, 95% CI 2-sided [-2.64 to -0.83], Standard Error of Mean 0.46
Statistical Analysis 17: Comparison: Placebo vs Tramadol; [analysis description as in outcome 6, analysis 15]; Test type: Superiority; p = 0.5412, ANCOVA; LS Mean Difference = -0.26, 95% CI 2-sided [-1.09 to 0.57], Standard Error of Mean 0.42
Statistical Analysis 18: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 6, analysis 15]; Test type: Superiority; p = 0.0107, ANCOVA; LS Mean Difference = -1.06, 95% CI 2-sided [-1.87 to -0.25], Standard Error of Mean 0.42
Statistical Analysis 19: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 6, analysis 15]; Test type: Superiority; p = 0.0004, ANCOVA; LS Mean Difference = -1.48, 95% CI 2-sided [-2.29 to -0.66], Standard Error of Mean 0.42
Statistical Analysis 20: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 24: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline RMDQ, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.0464, ANCOVA; LS Mean Difference = -0.98, 95% CI 2-sided [-1.94 to -0.02], Standard Error of Mean 0.49
Statistical Analysis 21: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 6, analysis 20]; Test type: Superiority; p = 0.0068, ANCOVA; LS Mean Difference = -1.33, 95% CI 2-sided [-2.30 to -0.37], Standard Error of Mean 0.49
Statistical Analysis 22: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 32: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline RMDQ, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.1485, ANCOVA; LS Mean Difference = -0.72, 95% CI 2-sided [-1.70 to 0.26], Standard Error of Mean 0.50
Statistical Analysis 23: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 6, analysis 22]; Test type: Superiority; p = 0.0507, ANCOVA; LS Mean Difference = -0.97, 95% CI 2-sided [-1.94 to 0.00], Standard Error of Mean 0.50
Statistical Analysis 24: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 40: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline RMDQ, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.2480, ANCOVA; LS Mean Difference = -0.59, 95% CI 2-sided [-1.60 to 0.41], Standard Error of Mean 0.51
Statistical Analysis 25: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 6, analysis 24]; Test type: Superiority; p = 0.1605, ANCOVA; LS Mean Difference = -0.71, 95% CI 2-sided [-1.71 to 0.28], Standard Error of Mean 0.51
Statistical Analysis 26: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 48: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline RMDQ, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.3654, ANCOVA; LS Mean Difference = -0.47, 95% CI 2-sided [-1.50 to 0.55], Standard Error of Mean 0.52
Statistical Analysis 27: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 6, analysis 26]; Test type: Superiority; p = 0.1782, ANCOVA; LS Mean Difference = -0.70, 95% CI 2-sided [-1.71 to 0.32], Standard Error of Mean 0.52
Statistical Analysis 28: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 56: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline RMDQ, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.3981, ANCOVA; LS Mean Difference = -0.44, 95% CI 2-sided [-1.47 to 0.58], Standard Error of Mean 0.52
Statistical Analysis 29: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 6, analysis 28]; Test type: Superiority; p = 0.1089, ANCOVA; LS Mean Difference = -0.83, 95% CI 2-sided [-1.84 to 0.18], Standard Error of Mean 0.52

7. Secondary Outcome: Change From Baseline in Roland Morris Disability Questionnaire (RMDQ) Score at Weeks 64 and 80: Observed Data
Description: The RMDQ is a self-administered, widely used health status measure index of how well participants with LBP are able to function with regard to daily activities. It measures pain and function, using 24 items describing limitations to everyday life that can be caused by LBP. The total score of the RMDQ is the total number of items checked ranging from 0 (no disability) to 24 (maximum disability), where higher scores indicated greater disability.
Time Frame: Baseline, Weeks 64 and 80
Population: ITT population included all randomized participants who received at least one dose of SC study medication (either tanezumab or matching placebo). Here, 'number analyzed' = participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Followed by Tanezumab 5 mg | Placebo Followed by Tanezumab 10 mg | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 202 | 204 | 407 | 407 | 605
units on a scale
  Baseline: number analyzed (Participants) | 202 | 204 | 405 | 407 | 605
  Baseline | 14.64 (5.26) | 14.98 (5.03) | 15.02 (5.21) | 15.06 (4.92) | 15.10 (5.11)
  Change at Week 64: number analyzed (Participants) | 63 | 59 | 141 | 149 | 204
  Change at Week 64 | -8.35 (6.72) | -8.71 (5.78) | -8.72 (6.32) | -7.64 (5.96) | -8.87 (5.88)
  Change at Week 80: number analyzed (Participants) | 62 | 59 | 135 | 146 | 193
  Change at Week 80 | -8.03 (7.00) | -7.27 (6.79) | -8.80 (6.68) | -7.13 (5.99) | -8.35 (6.01)

8. Secondary Outcome: Change From Baseline in Patient's Global Assessment (PGA) of Low Back Pain at Weeks 2, 4, 8, 16, 24, 32, 40, 48 and 56
Description: PGA of LBP was assessed by asking a question to participants: "Considering all the ways your low back pain affects you, how are you doing today?" Participants responded on a 5 point Likert scale ranging from 1-5, using IRT, where 1=very good (asymptomatic and no limitation of normal activities); 2=good (mild symptoms and no limitation of normal activities); 3=fair (moderate symptoms and limitation of some normal activities); 4=poor (severe symptoms and inability to carry out most normal activities); and 5=very poor (very severe symptoms which are intolerable and inability to carry out all normal activities). Higher scores indicated worsening of condition. Pre-specified intent of study for efficacy data up to W16 was to analyze participants who received placebo from Day1 and then received tanezumab 5/10 mg at W16,together,in placebo arm.Data has been reported per four arms.
Time Frame: Baseline, Weeks 2, 4, 8, 16, 24, 32, 40, 48 and 56
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 406 | 407 | 407 | 605
units on a scale
  Change at Week 2 | -0.54 (0.04) | -0.62 (0.04) | -0.67 (0.04) | -0.54 (0.03)
  Change at Week 4 | -0.64 (0.04) | -0.82 (0.04) | -0.86 (0.04) | -0.66 (0.04)
  Change at Week 8 | -0.69 (0.05) | -0.82 (0.05) | -0.89 (0.05) | -0.76 (0.04)
  Change at Week 16 | -0.86 (0.05) | -0.98 (0.05) | -1.02 (0.05) | -0.85 (0.04)
  Change at Week 24: number analyzed (Participants) | 0 | 407 | 407 | 605
  Change at Week 24 |  | -0.83 (0.06) | -0.82 (0.06) | -0.74 (0.05)
  Change at Week 32: number analyzed (Participants) | 0 | 407 | 407 | 605
  Change at Week 32 |  | -0.80 (0.06) | -0.79 (0.06) | -0.74 (0.05)
  Change at Week 40: number analyzed (Participants) | 0 | 407 | 407 | 605
  Change at Week 40 |  | -0.80 (0.06) | -0.75 (0.06) | -0.70 (0.05)
  Change at Week 48: number analyzed (Participants) | 0 | 407 | 407 | 605
  Change at Week 48 |  | -0.74 (0.07) | -0.72 (0.07) | -0.66 (0.06)
  Change at Week 56: number analyzed (Participants) | 0 | 407 | 407 | 605
  Change at Week 56 |  | -0.76 (0.06) | -0.74 (0.07) | -0.66 (0.06)
Statistical Analysis 1: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 2: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline PGA, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.1472, ANCOVA; LS Mean Difference = -0.08, 95% CI 2-sided [-0.18 to 0.03], Standard Error of Mean 0.05
Statistical Analysis 2: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.0135, ANCOVA; LS Mean Difference = -0.13, 95% CI 2-sided [-0.24 to -0.03], Standard Error of Mean 0.05
Statistical Analysis 3: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.0893, ANCOVA; LS Mean Difference = -0.08, 95% CI 2-sided [-0.18 to 0.01], Standard Error of Mean 0.05
Statistical Analysis 4: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.0044, ANCOVA; LS Mean Difference = -0.14, 95% CI 2-sided [-0.23 to -0.04], Standard Error of Mean 0.05
Statistical Analysis 5: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 4: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline PGA, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.0025, ANCOVA; LS Mean Difference = -0.17, 95% CI 2-sided [-0.28 to -0.06], Standard Error of Mean 0.06
Statistical Analysis 6: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 8, analysis 5]; Test type: Superiority; p = 0.0002, ANCOVA; LS Mean Difference = -0.21, 95% CI 2-sided [-0.32 to -0.10], Standard Error of Mean 0.06
Statistical Analysis 7: Comparison: Placebo vs Tramadol; [analysis description as in outcome 8, analysis 5]; Test type: Superiority; p = 0.8348, ANCOVA; LS Mean Difference = -0.01, 95% CI 2-sided [-0.11 to 0.09], Standard Error of Mean 0.05
Statistical Analysis 8: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 8, analysis 5]; Test type: Superiority; p = 0.0020, ANCOVA; LS Mean Difference = -0.16, 95% CI 2-sided [-0.26 to -0.06], Standard Error of Mean 0.05
Statistical Analysis 9: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 8, analysis 5]; Test type: Superiority; p = 0.0001, ANCOVA; LS Mean Difference = -0.20, 95% CI 2-sided [-0.30 to -0.10], Standard Error of Mean 0.05
Statistical Analysis 10: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 8: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline PGA, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.0272, ANCOVA; LS Mean Difference = -0.13, 95% CI 2-sided [-0.25 to -0.01], Standard Error of Mean 0.06
Statistical Analysis 11: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 8, analysis 10]; Test type: Superiority; p = 0.0009, ANCOVA; LS Mean Difference = -0.20, 95% CI 2-sided [-0.31 to -0.08], Standard Error of Mean 0.06
Statistical Analysis 12: Comparison: Placebo vs Tramadol; [analysis description as in outcome 8, analysis 10]; Test type: Superiority; p = 0.1680, ANCOVA; LS Mean Difference = -0.07, 95% CI 2-sided [-0.18 to 0.03], Standard Error of Mean 0.05
Statistical Analysis 13: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 8, analysis 10]; Test type: Superiority; p = 0.2968, ANCOVA; LS Mean Difference = -0.06, 95% CI 2-sided [-0.16 to 0.05], Standard Error of Mean 0.05
Statistical Analysis 14: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 8, analysis 10]; Test type: Superiority; p = 0.0219, ANCOVA; LS Mean Difference = -0.12, 95% CI 2-sided [-0.23 to -0.02], Standard Error of Mean 0.05
Statistical Analysis 15: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 16: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline PGA, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.0717, ANCOVA; LS Mean Difference = -0.12, 95% CI 2-sided [-0.25 to 0.01], Standard Error of Mean 0.07
Statistical Analysis 16: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 8, analysis 15]; Test type: Superiority; p = 0.0207, ANCOVA; LS Mean Difference = -0.16, 95% CI 2-sided [-0.29 to -0.02], Standard Error of Mean 0.07
Statistical Analysis 17: Comparison: Placebo vs Tramadol; [analysis description as in outcome 8, analysis 15]; Test type: Superiority; p = 0.8399, ANCOVA; LS Mean Difference = 0.01, 95% CI 2-sided [-0.11 to 0.13], Standard Error of Mean 0.06
Statistical Analysis 18: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 8, analysis 15]; Test type: Superiority; p = 0.0299, ANCOVA; LS Mean Difference = -0.13, 95% CI 2-sided [-0.25 to -0.01], Standard Error of Mean 0.06
Statistical Analysis 19: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 8, analysis 15]; Test type: Superiority; p = 0.0060, ANCOVA; LS Mean Difference = -0.17, 95% CI 2-sided [-0.29 to -0.05], Standard Error of Mean 0.06
Statistical Analysis 20: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 24: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline PGA, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.1974, ANCOVA; LS Mean Difference = -0.09, 95% CI 2-sided [-0.24 to 0.05], Standard Error of Mean 0.07
Statistical Analysis 21: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 6, analysis 20]; Test type: Superiority; p = 0.2780, ANCOVA; LS Mean Difference = -0.08, 95% CI 2-sided [-0.22 to 0.06], Standard Error of Mean 0.07
Statistical Analysis 22: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 32: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline PGA, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.4330, ANCOVA; LS Mean Difference = -0.06, 95% CI 2-sided [-0.21 to 0.09], Standard Error of Mean 0.07
Statistical Analysis 23: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 8, analysis 22]; Test type: Superiority; p = 0.4946, ANCOVA; LS Mean Difference = -0.05, 95% CI 2-sided [-0.20 to 0.09], Standard Error of Mean 0.07
Statistical Analysis 24: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 40: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline PGA, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.1884, ANCOVA; LS Mean Difference = -0.10, 95% CI 2-sided [-0.25 to 0.05], Standard Error of Mean 0.08
Statistical Analysis 25: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 8, analysis 24]; Test type: Superiority; p = 0.5210, ANCOVA; LS Mean Difference = -0.05, 95% CI 2-sided [-0.20 to 0.10], Standard Error of Mean 0.08
Statistical Analysis 26: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 48: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline PGA, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.3329, ANCOVA; LS Mean Difference = -0.08, 95% CI 2-sided [-0.23 to 0.08], Standard Error of Mean 0.08
Statistical Analysis 27: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 8, analysis 26]; Test type: Superiority; p = 0.5173, ANCOVA; LS Mean Difference = -0.05, 95% CI 2-sided [-0.21 to 0.10], Standard Error of Mean 0.08
Statistical Analysis 28: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 56: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline PGA, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.2346, ANCOVA; LS Mean Difference = -0.10, 95% CI 2-sided [-0.25 to 0.06], Standard Error of Mean 0.08
Statistical Analysis 29: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 8, analysis 28]; Test type: Superiority; p = 0.3634, ANCOVA; LS Mean Difference = -0.07, 95% CI 2-sided [-0.23 to 0.09], Standard Error of Mean 0.08

9. Secondary Outcome: Change From Baseline in Patient's Global Assessment (PGA) of Low Back Pain at Week 64: Observed Data
Description: PGA of LBP was assessed by asking a question to participants: "Considering all the ways your low back pain affects you, how are you doing today?" Participants responded on a 5 point Likert scale ranging from 1-5, using IRT, where 1=very good (asymptomatic and no limitation of normal activities); 2=good (mild symptoms and no limitation of normal activities); 3=fair (moderate symptoms and limitation of some normal activities); 4=poor (severe symptoms and inability to carry out most normal activities); and 5=very poor (very severe symptoms which are intolerable and inability to carry out all normal activities). Higher scores indicated worsening of condition.
Time Frame: Baseline, Week 64
Population: ITT population included all randomized participants who received at least one dose of SC study medication (either tanezumab or matching placebo). Here, 'Number analyzed' = participants evaluable for this outcome measure at specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Followed by Tanezumab 5 mg | Placebo Followed by Tanezumab 10 mg | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 202 | 204 | 407 | 407 | 605
units on a scale
  Baseline: number analyzed (Participants) | 202 | 204 | 405 | 407 | 605
  Baseline | 3.47 (0.65) | 3.49 (0.60) | 3.47 (0.61) | 3.53 (0.63) | 3.50 (0.63)
  Change at Week 64: number analyzed (Participants) | 63 | 57 | 140 | 147 | 200
  Change at Week 64 | -1.21 (1.02) | -1.16 (0.86) | -1.03 (0.98) | -1.01 (0.92) | -1.14 (0.88)

10. Secondary Outcome: Percentage of Participants With Cumulative Percent Change From Baseline in Daily Average Low Back Pain Intensity (LBPI) Score at Weeks 16, 24 and 56: Mixed Baseline Observation Carried Forward (BOCF)/Last Observation Carried Forward (LOCF)
Description: Average LBP was assessed on an 11-point NRS captured through an IRT. LBPI score was captured once a week for week 64. Participants described their average LBP during the past 24 hours on a scale ranging from 0 (no pain) to 10 (worst possible pain), where higher scores indicated higher pain.Percentage of participants with cumulative reduction (as percent) (greater than [>] 0%; >= 10, 20, 30, 40, 50, 60, 70, 80, 90 and equals to [=] 100 %) in LBPI from baseline to weeks 16, 24 and 56 were reported, participants (%) are reported more than once in categories specified.Missing data was imputed using mixed BOCF/LOCF.Pre-specified intent of study for efficacy data up to W16 was to analyze participants who received placebo from Day1 and then received tanezumab 5/10 mg at W16,together,in placebo arm.Data has been reported per four arms.Also, intent of study was to compare tanezumab Vs placebo for data up to & including W16 & comparisons of tanezumab Vs tramadol for data up to & including W56.
Time Frame: Baseline, Weeks 16, 24 and 56
Population: ITT population.Data were not collected after W16 in placebo arm for this outcome measure, as those who met criteria to continue, switched to active treatment with tanezumab after W16. Overall Number of Participants analyzed(N)=participants evaluable for this outcome measure (OM).
Measure: Number; unit: percentage of participants
Groups:
- Pooled Tanezumab 5 mg: Tanezumab (RN624 or PF-04383119) 5 mg injection administered SC once every 8 weeks from Day 1, and placebo tablets matched to tramadol PR, orally, once daily from Day 1 up to week 56.
Arm/Group | Placebo | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 404 | 406 | 406 | 605
percentage of participants
  Week 16: >0% | 80.8 | 85.3 | 87.2 | 80.8
  Week 16: >=10% | 73.6 | 79.1 | 82.1 | 74.5
  Week 16: >=20% | 64.8 | 72.5 | 73.2 | 64.8
  Week 16: >=30% | 55.7 | 64.6 | 65.4 | 57.9
  Week 16: >=40% | 46.8 | 52.1 | 56.3 | 49.9
  Week 16: >=50% | 37.2 | 43.2 | 46.2 | 42.8
  Week 16: >=60% | 29.3 | 33.4 | 36.9 | 32.2
  Week 16: >=70% | 18.5 | 21.6 | 25.1 | 20.2
  Week 16: >=80% | 10.3 | 13.3 | 15.7 | 13.4
  Week 16: >=90% | 5.4 | 7.4 | 6.6 | 6.3
  Week 16: =100% | 2.7 | 3.9 | 2.7 | 4.1
  Week 24: >0%: number analyzed (Participants) | 0 | 406 | 406 | 605
  Week 24: >0% |  | 71.9 | 72.4 | 66.4
  Week 24: >=10%: number analyzed (Participants) | 0 | 406 | 406 | 605
  Week 24: >=10% |  | 68.5 | 69.2 | 63.1
  Week 24: >=20%: number analyzed (Participants) | 0 | 406 | 406 | 605
  Week 24: >=20% |  | 61.8 | 64.8 | 58.0
  Week 24: >=30%: number analyzed (Participants) | 0 | 406 | 406 | 605
  Week 24: >=30% |  | 57.6 | 62.1 | 53.6
  Week 24: >=40%: number analyzed (Participants) | 0 | 406 | 406 | 605
  Week 24: >=40% |  | 51.5 | 55.9 | 47.8
  Week 24: >=50%: number analyzed (Participants) | 0 | 406 | 406 | 605
  Week 24: >=50% |  | 44.1 | 48.8 | 41.2
  Week 24: >=60%: number analyzed (Participants) | 0 | 406 | 406 | 605
  Week 24: >=60% |  | 33.7 | 37.4 | 32.2
  Week 24: >=70%: number analyzed (Participants) | 0 | 406 | 406 | 605
  Week 24: >=70% |  | 24.4 | 27.6 | 23.8
  Week 24: >=80%: number analyzed (Participants) | 0 | 406 | 406 | 605
  Week 24: >=80% |  | 16.5 | 15.3 | 14.2
  Week 24: >=90%: number analyzed (Participants) | 0 | 406 | 406 | 605
  Week 24: >=90% |  | 6.2 | 7.1 | 6.6
  Week 24: =100%: number analyzed (Participants) | 0 | 406 | 406 | 605
  Week 24: =100% |  | 3.4 | 5.2 | 3.8
  Week 56: >=0%: number analyzed (Participants) | 0 | 406 | 406 | 605
  Week 56: >=0% |  | 59.9 | 61.1 | 58.2
  Week 56: >=10%: number analyzed (Participants) | 0 | 406 | 406 | 605
  Week 56: >=10% |  | 57.6 | 58.9 | 55.7
  Week 56: >=20%: number analyzed (Participants) | 0 | 406 | 406 | 605
  Week 56: >=20% |  | 53.2 | 55.7 | 51.2
  Week 56: >=30%: number analyzed (Participants) | 0 | 406 | 406 | 605
  Week 56: >=30% |  | 50.7 | 53.9 | 46.8
  Week 56: >=40%: number analyzed (Participants) | 0 | 406 | 406 | 605
  Week 56: >=40% |  | 46.1 | 50.7 | 42.1
  Week 56: >=50%: number analyzed (Participants) | 0 | 406 | 406 | 605
  Week 56: >=50% |  | 41.6 | 45.3 | 38.7
  Week 56: >=60%: number analyzed (Participants) | 0 | 406 | 406 | 605
  Week 56: >=60% |  | 34.5 | 36.0 | 31.1
  Week 56: >=70%: number analyzed (Participants) | 0 | 406 | 406 | 605
  Week 56: >=70% |  | 27.1 | 27.6 | 23.3
  Week 56: >=80%: number analyzed (Participants) | 0 | 406 | 406 | 605
  Week 56: >=80% |  | 17.2 | 19.0 | 15.5
  Week 56: >=90%: number analyzed (Participants) | 0 | 406 | 406 | 605
  Week 56: >=90% |  | 8.9 | 10.3 | 9.3
  Week 56: =100%: number analyzed (Participants) | 0 | 406 | 406 | 605
  Week 56: =100% |  | 6.7 | 7.9 | 6.1

11. Secondary Outcome: Percentage of Participants Achieving Average LBPI Reduction of >=30 Percent(%), >=50%, >=70% and >=90% From Baseline at Weeks 2, 4, 8, 12, 16, 24, 32, 40, 48 and 56: Mixed Baseline Observation Carried Forward (BOCF)/Last Observation Carried Forward (LOCF)
Description: Average LBP was assessed on an 11-point NRS captured through an IRT. The LBPI score was captured once a week for week 64. Participants described their average LBP during the past 24 hours on a scale ranging from 0 (no pain) to 10 (worst possible pain), where higher scores indicated higher pain. Percentage of participants with reduction in LBPI of at least (>=) 30%, 50%, 70% and 90% at weeks 2, 4, 8, 12, 16, 24, 32, 40, 48 and 56 compared to baseline were classified as responders to LBPI and are reported here, participants (%) are reported more than once in categories specified.Pre-specified intent of study for efficacy data up to W16 was to analyze participants who received placebo from Day1 and then received tanezumab 5/10 mg at W16,together,in placebo arm.Data has been reported per four arms.Also, intent of study was to compare tanezumab Vs placebo for data up to & including W16 & comparisons of tanezumab Vs tramadol for data up to & including W56.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 24, 32, 40, 48 and 56
Population: ITT population.Data were not collected after W16 in placebo arm for this outcome measure, as those who met criteria to continue, switched to active treatment with tanezumab after W16. N=participants evaluable for this OM.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 404 | 406 | 406 | 605
percentage of participants
  Week 2: At least 30% reduction | 20.8 | 31.3 | 31.8 | 28.6
  Week 2: At least 50% reduction | 8.9 | 13.1 | 14.8 | 11.2
  Week 2: At least 70% reduction | 2.7 | 5.2 | 5.7 | 3.3
  Week 2: At least 90% reduction | 1.0 | 1.0 | 1.7 | 0.8
  Week 4: At least 30% reduction | 35.6 | 47.5 | 53.2 | 42.1
  Week 4: At least 50% reduction | 19.1 | 26.1 | 30.8 | 23.0
  Week 4: At least 70% reduction | 7.4 | 12.8 | 17.7 | 9.1
  Week 4: At least 90% reduction | 2.7 | 2.7 | 3.7 | 2.5
  Week 8: At least 30% reduction | 42.6 | 56.2 | 59.4 | 51.2
  Week 8: At least 50% reduction | 24.0 | 35.7 | 40.1 | 31.9
  Week 8: At least 70% reduction | 10.9 | 15.3 | 21.7 | 14.2
  Week 8: At least 90% reduction | 4.0 | 4.4 | 4.4 | 3.8
  Week 12: At least 30% reduction | 53.5 | 61.3 | 66.5 | 56.7
  Week 12: At least 50% reduction | 34.7 | 41.9 | 47.3 | 38.2
  Week 12: At least 70% reduction | 14.9 | 19.7 | 26.4 | 19.3
  Week 12: At least 90% reduction | 5.0 | 7.6 | 7.9 | 6.1
  Week 16: At least 30% reduction | 55.9 | 64.8 | 65.5 | 57.9
  Week 16: At least 50% reduction | 37.4 | 43.3 | 46.3 | 42.8
  Week 16: At least 70% reduction | 18.6 | 21.7 | 25.1 | 20.2
  Week 16: At least 90% reduction | 5.4 | 7.4 | 6.7 | 6.3
  Week 24: At least 30% reduction: number analyzed (Participants) | 0 | 406 | 406 | 605
  Week 24: At least 30% reduction |  | 57.6 | 62.1 | 53.6
  Week 24: At least 50% reduction: number analyzed (Participants) | 0 | 406 | 406 | 605
  Week 24: At least 50% reduction |  | 44.1 | 48.8 | 41.2
  Week 24: At least 70% reduction: number analyzed (Participants) | 0 | 406 | 406 | 605
  Week 24: At least 70% reduction |  | 24.4 | 27.6 | 23.8
  Week 24: At least 90% reduction: number analyzed (Participants) | 0 | 406 | 406 | 605
  Week 24: At least 90% reduction |  | 6.2 | 7.1 | 6.6
  Week 32: At least 30% reduction: number analyzed (Participants) | 0 | 406 | 406 | 605
  Week 32: At least 30% reduction |  | 56.7 | 57.6 | 50.6
  Week 32: At least 50% reduction: number analyzed (Participants) | 0 | 406 | 406 | 605
  Week 32: At least 50% reduction |  | 44.6 | 46.3 | 39.7
  Week 32: At least 70% reduction: number analyzed (Participants) | 0 | 406 | 406 | 605
  Week 32: At least 70% reduction |  | 27.1 | 25.6 | 22.5
  Week 32: At least 90% reduction: number analyzed (Participants) | 0 | 406 | 406 | 605
  Week 32: At least 90% reduction |  | 7.6 | 9.6 | 7.3
  Week 40: At least 30% reduction: number analyzed (Participants) | 0 | 406 | 406 | 605
  Week 40: At least 30% reduction |  | 53.0 | 53.9 | 49.4
  Week 40: At least 50% reduction: number analyzed (Participants) | 0 | 406 | 406 | 605
  Week 40: At least 50% reduction |  | 43.1 | 44.8 | 39.7
  Week 40: At least 70% reduction: number analyzed (Participants) | 0 | 406 | 406 | 605
  Week 40: At least 70% reduction |  | 26.4 | 28.1 | 24.1
  Week 40: At least 90% reduction: number analyzed (Participants) | 0 | 406 | 406 | 605
  Week 40: At least 90% reduction |  | 9.6 | 11.3 | 7.6
  Week 48: At least 30% reduction: number analyzed (Participants) | 0 | 406 | 406 | 605
  Week 48: At least 30% reduction |  | 52.2 | 53.0 | 48.6
  Week 48: At least 50% reduction: number analyzed (Participants) | 0 | 406 | 406 | 605
  Week 48: At least 50% reduction |  | 43.1 | 44.6 | 38.7
  Week 48: At least 70% reduction: number analyzed (Participants) | 0 | 406 | 406 | 605
  Week 48: At least 70% reduction |  | 27.1 | 26.6 | 23.5
  Week 48: At least 90% reduction: number analyzed (Participants) | 0 | 406 | 406 | 605
  Week 48: At least 90% reduction |  | 9.4 | 11.1 | 8.3
  Week 56: At least 30% reduction: number analyzed (Participants) | 0 | 406 | 406 | 605
  Week 56: At least 30% reduction |  | 50.7 | 53.9 | 46.8
  Week 56: At least 50% reduction: number analyzed (Participants) | 0 | 406 | 406 | 605
  Week 56: At least 50% reduction |  | 41.6 | 45.3 | 38.7
  Week 56: At least 70% reduction: number analyzed (Participants) | 0 | 406 | 406 | 605
  Week 56: At least 70% reduction |  | 27.1 | 27.6 | 23.3
  Week 56: At least 90% reduction: number analyzed (Participants) | 0 | 406 | 406 | 605
  Week 56: At least 90% reduction |  | 8.9 | 10.3 | 9.3
Statistical Analysis 1: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 2, >=30%: Odds ratio (OR) and 95% Confidence interval (CI) estimated from logistic regression model. Logistic regression model included baseline average LBPI and treatment; Test type: Superiority; p = 0.0007, Regression, Logistic; Odds Ratio (OR) = 1.74, 95% CI 2-sided [1.26 to 2.39]
Statistical Analysis 2: Comparison: Placebo vs Pooled Tanezumab 10 mg; Week 2, >=30%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline average LBPI and treatment; Test type: Superiority; p = 0.0004, Regression, Logistic; Odds Ratio (OR) = 1.77, 95% CI 2-sided [1.29 to 2.44]
Statistical Analysis 3: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 11, analysis 2]; Test type: Superiority; p = 0.3456, Regression, Logistic; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.87 to 1.50]
Statistical Analysis 4: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 11, analysis 2]; Test type: Superiority; p = 0.2771, Regression, Logistic; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.89 to 1.53]
Statistical Analysis 5: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 2, >=50%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline average LBPI and treatment; Test type: Superiority; p = 0.0594, Regression, Logistic; Odds Ratio (OR) = 1.54, 95% CI 2-sided [0.98 to 2.41]
Statistical Analysis 6: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 11, analysis 5]; Test type: Superiority; p = 0.0105, Regression, Logistic; Odds Ratio (OR) = 1.77, 95% CI 2-sided [1.14 to 2.75]
Statistical Analysis 7: Comparison: Placebo vs Tramadol; [analysis description as in outcome 11, analysis 5]; Test type: Superiority; p = 0.2360, Regression, Logistic; Odds Ratio (OR) = 1.29, 95% CI 2-sided [0.85 to 1.98]
Statistical Analysis 8: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 11, analysis 5]; Test type: Superiority; p = 0.3746, Regression, Logistic; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.81 to 1.75]
Statistical Analysis 9: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 11, analysis 5]; Test type: Superiority; p = 0.0974, Regression, Logistic; Odds Ratio (OR) = 1.37, 95% CI 2-sided [0.94 to 1.99]
Statistical Analysis 10: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 2, >=70%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline average LBPI and treatment; Test type: Superiority; p = 0.0806, Regression, Logistic; Odds Ratio (OR) = 1.94, 95% CI 2-sided [0.92 to 4.08]
Statistical Analysis 11: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 11, analysis 10]; Test type: Superiority; p = 0.0407, Regression, Logistic; Odds Ratio (OR) = 2.15, 95% CI 2-sided [1.03 to 4.47]
Statistical Analysis 12: Comparison: Placebo vs Tramadol; [analysis description as in outcome 11, analysis 10]; Test type: Superiority; p = 0.5966, Regression, Logistic; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.58 to 2.58]
Statistical Analysis 13: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 11, analysis 10]; Test type: Superiority; p = 0.1492, Regression, Logistic; Odds Ratio (OR) = 1.59, 95% CI 2-sided [0.85 to 2.96]
Statistical Analysis 14: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 11, analysis 10]; Test type: Superiority; p = 0.0720, Regression, Logistic; Odds Ratio (OR) = 1.76, 95% CI 2-sided [0.95 to 3.24]
Statistical Analysis 15: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 2, >=90%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline average LBPI and treatment; Test type: Superiority; p = 0.9926, Regression, Logistic; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.25 to 4.00]
Statistical Analysis 16: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 11, analysis 15]; Test type: Superiority; p = 0.3726, Regression, Logistic; Odds Ratio (OR) = 1.75, 95% CI 2-sided [0.51 to 6.04]
Statistical Analysis 17: Comparison: Placebo vs Tramadol; [analysis description as in outcome 11, analysis 15]; Test type: Superiority; p = 0.7874, Regression, Logistic; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.22 to 3.12]
Statistical Analysis 18: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 11, analysis 15]; Test type: Superiority; p = 0.7950, Regression, Logistic; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.32 to 4.46]
Statistical Analysis 19: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 11, analysis 15]; Test type: Superiority; p = 0.2065, Regression, Logistic; Odds Ratio (OR) = 2.10, 95% CI 2-sided [0.66 to 6.68]
Statistical Analysis 20: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 4, >=30%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline average LBPI and treatment; Test type: Superiority; p = 0.0006, Regression, Logistic; Odds Ratio (OR) = 1.64, 95% CI 2-sided [1.23 to 2.17]
Statistical Analysis 21: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 11, analysis 20]; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 2.05, 95% CI 2-sided [1.55 to 2.72]
Statistical Analysis 22: Comparison: Placebo vs Tramadol; [analysis description as in outcome 11, analysis 20]; Test type: Superiority; p = 0.0387, Regression, Logistic; Odds Ratio (OR) = 1.32, 95% CI 2-sided [1.01 to 1.71]
Statistical Analysis 23: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 11, analysis 20]; Test type: Superiority; p = 0.0903, Regression, Logistic; Odds Ratio (OR) = 1.24, 95% CI 2-sided [0.97 to 1.60]
Statistical Analysis 24: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 11, analysis 20]; Test type: Superiority; p = 0.0006, Regression, Logistic; Odds Ratio (OR) = 1.56, 95% CI 2-sided [1.21 to 2.01]
Statistical Analysis 25: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 4, >=50%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline average LBPI and treatment; Test type: Superiority; p = 0.0166, Regression, Logistic; Odds Ratio (OR) = 1.50, 95% CI 2-sided [1.08 to 2.09]
Statistical Analysis 26: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 11, analysis 25]; Test type: Superiority; p = 0.0001, Regression, Logistic; Odds Ratio (OR) = 1.89, 95% CI 2-sided [1.36 to 2.62]
Statistical Analysis 27: Comparison: Placebo vs Tramadol; [analysis description as in outcome 11, analysis 25]; Test type: Superiority; p = 0.1389, Regression, Logistic; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.93 to 1.73]
Statistical Analysis 28: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 11, analysis 25]; Test type: Superiority; p = 0.2504, Regression, Logistic; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.89 to 1.59]
Statistical Analysis 29: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 11, analysis 25]; Test type: Superiority; p = 0.0057, Regression, Logistic; Odds Ratio (OR) = 1.49, 95% CI 2-sided [1.12 to 1.98]
Statistical Analysis 30: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 4, >=70%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline average LBPI and treatment; Test type: Superiority; p = 0.0126, Regression, Logistic; Odds Ratio (OR) = 1.83, 95% CI 2-sided [1.14 to 2.93]
Statistical Analysis 31: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 11, analysis 30]; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 2.69, 95% CI 2-sided [1.71 to 4.22]
Statistical Analysis 32: Comparison: Placebo vs Tramadol; [analysis description as in outcome 11, analysis 30]; Test type: Superiority; p = 0.3485, Regression, Logistic; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.79 to 1.99]
Statistical Analysis 33: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 11, analysis 30]; Test type: Superiority; p = 0.0642, Regression, Logistic; Odds Ratio (OR) = 1.46, 95% CI 2-sided [0.98 to 2.19]
Statistical Analysis 34: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 11, analysis 30]; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 2.16, 95% CI 2-sided [1.48 to 3.14]
Statistical Analysis 35: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 4, >=90%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline average LBPI and treatment; Test type: Superiority; p = 0.9819, Regression, Logistic; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.42 to 2.31]
Statistical Analysis 36: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 11, analysis 35]; Test type: Superiority; p = 0.4333, Regression, Logistic; Odds Ratio (OR) = 1.37, 95% CI 2-sided [0.62 to 3.02]
Statistical Analysis 37: Comparison: Placebo vs Tramadol; [analysis description as in outcome 11, analysis 35]; Test type: Superiority; p = 0.8140, Regression, Logistic; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.41 to 2.00]
Statistical Analysis 38: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 11, analysis 35]; Test type: Superiority; p = 0.8331, Regression, Logistic; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.49 to 2.40]
Statistical Analysis 39: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 11, analysis 35]; Test type: Superiority; p = 0.2682, Regression, Logistic; Odds Ratio (OR) = 1.51, 95% CI 2-sided [0.73 to 3.12]
Statistical Analysis 40: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 8, >=30%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline average LBPI and treatment; Test type: Superiority; p = 0.0001, Regression, Logistic; Odds Ratio (OR) = 1.73, 95% CI 2-sided [1.31 to 2.29]
Statistical Analysis 41: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 11, analysis 40]; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 1.97, 95% CI 2-sided [1.49 to 2.61]
Statistical Analysis 42: Comparison: Placebo vs Tramadol; [analysis description as in outcome 11, analysis 40]; Test type: Superiority; p = 0.0071, Regression, Logistic; Odds Ratio (OR) = 1.42, 95% CI 2-sided [1.10 to 1.83]
Statistical Analysis 43: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 11, analysis 40]; Test type: Superiority; p = 0.1187, Regression, Logistic; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.95 to 1.57]
Statistical Analysis 44: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 11, analysis 40]; Test type: Superiority; p = 0.0110, Regression, Logistic; Odds Ratio (OR) = 1.39, 95% CI 2-sided [1.08 to 1.79]
Statistical Analysis 45: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 8, >=50%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline average LBPI and treatment; Test type: Superiority; p = 0.0003, Regression, Logistic; Odds Ratio (OR) = 1.76, 95% CI 2-sided [1.30 to 2.39]
Statistical Analysis 46: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 11, analysis 45]; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 2.12, 95% CI 2-sided [1.57 to 2.87]
Statistical Analysis 47: Comparison: Placebo vs Tramadol; [analysis description as in outcome 11, analysis 45]; Test type: Superiority; p = 0.0069, Regression, Logistic; Odds Ratio (OR) = 1.48, 95% CI 2-sided [1.11 to 1.97]
Statistical Analysis 48: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 11, analysis 45]; Test type: Superiority; p = 0.2076, Regression, Logistic; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.91 to 1.55]
Statistical Analysis 49: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 11, analysis 45]; Test type: Superiority; p = 0.0072, Regression, Logistic; Odds Ratio (OR) = 1.43, 95% CI 2-sided [1.10 to 1.86]
Statistical Analysis 50: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 8, >=70%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline average LBPI and treatment; Test type: Superiority; p = 0.0694, Regression, Logistic; Odds Ratio (OR) = 1.47, 95% CI 2-sided [0.97 to 2.22]
Statistical Analysis 51: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 11, analysis 50]; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 2.27, 95% CI 2-sided [1.53 to 3.36]
Statistical Analysis 52: Comparison: Placebo vs Tramadol; [analysis description as in outcome 11, analysis 50]; Test type: Superiority; p = 0.1210, Regression, Logistic; Odds Ratio (OR) = 1.36, 95% CI 2-sided [0.92 to 2.00]
Statistical Analysis 53: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 11, analysis 50]; Test type: Superiority; p = 0.6706, Regression, Logistic; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.76 to 1.54]
Statistical Analysis 54: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 11, analysis 50]; Test type: Superiority; p = 0.0022, Regression, Logistic; Odds Ratio (OR) = 1.67, 95% CI 2-sided [1.20 to 2.32]
Statistical Analysis 55: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 8, >=90%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline average LBPI and treatment; Test type: Superiority; p = 0.7546, Regression, Logistic; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.56 to 2.22]
Statistical Analysis 56: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 11, analysis 55]; Test type: Superiority; p = 0.7347, Regression, Logistic; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.57 to 2.24]
Statistical Analysis 57: Comparison: Placebo vs Tramadol; [analysis description as in outcome 11, analysis 55]; Test type: Superiority; p = 0.9029, Regression, Logistic; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.50 to 1.84]
Statistical Analysis 58: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 11, analysis 55]; Test type: Superiority; p = 0.6402, Regression, Logistic; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.62 to 2.18]
Statistical Analysis 59: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 11, analysis 55]; Test type: Superiority; p = 0.6199, Regression, Logistic; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.62 to 2.20]
Statistical Analysis 60: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 12, >=30%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline average LBPI and treatment; Test type: Superiority; p = 0.0229, Regression, Logistic; Odds Ratio (OR) = 1.38, 95% CI 2-sided [1.05 to 1.83]
Statistical Analysis 61: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 11, analysis 60]; Test type: Superiority; p = 0.0002, Regression, Logistic; Odds Ratio (OR) = 1.73, 95% CI 2-sided [1.30 to 2.30]
Statistical Analysis 62: Comparison: Placebo vs Tramadol; [analysis description as in outcome 11, analysis 60]; Test type: Superiority; p = 0.3150, Regression, Logistic; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.88 to 1.47]
Statistical Analysis 63: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 11, analysis 60]; Test type: Superiority; p = 0.1370, Regression, Logistic; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.94 to 1.57]
Statistical Analysis 64: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 11, analysis 60]; Test type: Superiority; p = 0.0018, Regression, Logistic; Odds Ratio (OR) = 1.52, 95% CI 2-sided [1.17 to 1.97]
Statistical Analysis 65: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 12, >=50%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline average LBPI and treatment; Test type: Superiority; p = 0.0342, Regression, Logistic; Odds Ratio (OR) = 1.36, 95% CI 2-sided [1.02 to 1.81]
Statistical Analysis 66: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 11, analysis 65]; Test type: Superiority; p = 0.0003, Regression, Logistic; Odds Ratio (OR) = 1.69, 95% CI 2-sided [1.27 to 2.24]
Statistical Analysis 67: Comparison: Placebo vs Tramadol; [analysis description as in outcome 11, analysis 65]; Test type: Superiority; p = 0.2561, Regression, Logistic; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.90 to 1.51]
Statistical Analysis 68: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 11, analysis 65]; Test type: Superiority; p = 0.2358, Regression, Logistic; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.90 to 1.51]
Statistical Analysis 69: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 11, analysis 65]; Test type: Superiority; p = 0.0040, Regression, Logistic; Odds Ratio (OR) = 1.45, 95% CI 2-sided [1.13 to 1.87]
Statistical Analysis 70: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 12, >=70%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline average LBPI and treatment; Test type: Superiority; p = 0.0723, Regression, Logistic; Odds Ratio (OR) = 1.40, 95% CI 2-sided [0.97 to 2.02]
Statistical Analysis 71: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 11, analysis 70]; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 2.06, 95% CI 2-sided [1.45 to 2.92]
Statistical Analysis 72: Comparison: Placebo vs Tramadol; [analysis description as in outcome 11, analysis 70]; Test type: Superiority; p = 0.0653, Regression, Logistic; Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.98 to 1.94]
Statistical Analysis 73: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 11, analysis 70]; Test type: Superiority; p = 0.9177, Regression, Logistic; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.74 to 1.40]
Statistical Analysis 74: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 11, analysis 70]; Test type: Superiority; p = 0.0088, Regression, Logistic; Odds Ratio (OR) = 1.49, 95% CI 2-sided [1.11 to 2.01]
Statistical Analysis 75: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 12, >=90%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline average LBPI and treatment; Test type: Superiority; p = 0.1197, Regression, Logistic; Odds Ratio (OR) = 1.58, 95% CI 2-sided [0.89 to 2.83]
Statistical Analysis 76: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 11, analysis 75]; Test type: Superiority; p = 0.0913, Regression, Logistic; Odds Ratio (OR) = 1.64, 95% CI 2-sided [0.92 to 2.92]
Statistical Analysis 77: Comparison: Placebo vs Tramadol; [analysis description as in outcome 11, analysis 75]; Test type: Superiority; p = 0.4317, Regression, Logistic; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.72 to 2.19]
Statistical Analysis 78: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 11, analysis 75]; Test type: Superiority; p = 0.3498, Regression, Logistic; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.77 to 2.08]
Statistical Analysis 79: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 11, analysis 75]; Test type: Superiority; p = 0.2768, Regression, Logistic; Odds Ratio (OR) = 1.31, 95% CI 2-sided [0.80 to 2.15]
Statistical Analysis 80: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 16, >=30%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline average LBPI and treatment; Test type: Superiority; p = 0.0101, Regression, Logistic; Odds Ratio (OR) = 1.45, 95% CI 2-sided [1.09 to 1.92]
Statistical Analysis 81: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 11, analysis 80]; Test type: Superiority; p = 0.0054, Regression, Logistic; Odds Ratio (OR) = 1.50, 95% CI 2-sided [1.13 to 1.99]
Statistical Analysis 82: Comparison: Placebo vs Tramadol; [analysis description as in outcome 11, analysis 80]; Test type: Superiority; p = 0.5493, Regression, Logistic; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.84 to 1.39]
Statistical Analysis 83: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 11, analysis 80]; Test type: Superiority; p = 0.0269, Regression, Logistic; Odds Ratio (OR) = 1.34, 95% CI 2-sided [1.03 to 1.74]
Statistical Analysis 84: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 11, analysis 80]; Test type: Superiority; p = 0.0144, Regression, Logistic; Odds Ratio (OR) = 1.38, 95% CI 2-sided [1.07 to 1.80]
Statistical Analysis 85: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 16, >=50%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline average LBPI and treatment; Test type: Superiority; p = 0.0846, Regression, Logistic; Odds Ratio (OR) = 1.28, 95% CI 2-sided [0.97 to 1.70]
Statistical Analysis 86: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 11, analysis 85]; Test type: Superiority; p = 0.0101, Regression, Logistic; Odds Ratio (OR) = 1.45, 95% CI 2-sided [1.09 to 1.91]
Statistical Analysis 87: Comparison: Placebo vs Tramadol; [analysis description as in outcome 11, analysis 85]; Test type: Superiority; p = 0.0848, Regression, Logistic; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.97 to 1.62]
Statistical Analysis 88: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 11, analysis 85]; Test type: Superiority; p = 0.8732, Regression, Logistic; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.79 to 1.32]
Statistical Analysis 89: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 11, analysis 85]; Test type: Superiority; p = 0.2734, Regression, Logistic; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.89 to 1.48]
Statistical Analysis 90: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 16, >=70%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline average LBPI and treatment; Test type: Superiority; p = 0.2839, Regression, Logistic; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.86 to 1.70]
Statistical Analysis 91: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 11, analysis 90]; Test type: Superiority; p = 0.0238, Regression, Logistic; Odds Ratio (OR) = 1.47, 95% CI 2-sided [1.05 to 2.07]
Statistical Analysis 92: Comparison: Placebo vs Tramadol; [analysis description as in outcome 11, analysis 90]; Test type: Superiority; p = 0.5212, Regression, Logistic; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.81 to 1.53]
Statistical Analysis 93: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 11, analysis 90]; Test type: Superiority; p = 0.5954, Regression, Logistic; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.80 to 1.48]
Statistical Analysis 94: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 11, analysis 90]; Test type: Superiority; p = 0.0638, Regression, Logistic; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.98 to 1.79]
Statistical Analysis 95: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 16, >=90%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline average LBPI and treatment; Test type: Superiority; p = 0.2661, Regression, Logistic; Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.78 to 2.44]
Statistical Analysis 96: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 11, analysis 95]; Test type: Superiority; p = 0.4717, Regression, Logistic; Odds Ratio (OR) = 1.24, 95% CI 2-sided [0.69 to 2.21]
Statistical Analysis 97: Comparison: Placebo vs Tramadol; [analysis description as in outcome 11, analysis 95]; Test type: Superiority; p = 0.5798, Regression, Logistic; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.68 to 2.00]
Statistical Analysis 98: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 11, analysis 95]; Test type: Superiority; p = 0.5027, Regression, Logistic; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.72 to 1.95]
Statistical Analysis 99: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 11, analysis 95]; Test type: Superiority; p = 0.8165, Regression, Logistic; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.64 to 1.77]
Statistical Analysis 100: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 24, >=30%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline average LBPI and treatment; Test type: Superiority; p = 0.1996, Regression, Logistic; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.92 to 1.52]
Statistical Analysis 101: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 11, analysis 100]; Test type: Superiority; p = 0.0074, Regression, Logistic; Odds Ratio (OR) = 1.42, 95% CI 2-sided [1.10 to 1.83]
Statistical Analysis 102: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 24, >=50%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline average LBPI and treatment; Test type: Superiority; p = 0.3557, Regression, Logistic; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.87 to 1.45]
Statistical Analysis 103: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 11, analysis 102]; Test type: Superiority; p = 0.0170, Regression, Logistic; Odds Ratio (OR) = 1.36, 95% CI 2-sided [1.06 to 1.75]
Statistical Analysis 104: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 24, >=70%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline average LBPI and treatment; Test type: Superiority; p = 0.8641, Regression, Logistic; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.76 to 1.38]
Statistical Analysis 105: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 11, analysis 104]; Test type: Superiority; p = 0.1768, Regression, Logistic; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.91 to 1.62]
Statistical Analysis 106: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 24, >=90%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline average LBPI and treatment; Test type: Superiority; p = 0.7696, Regression, Logistic; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.55 to 1.55]
Statistical Analysis 107: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 11, analysis 106]; Test type: Superiority; p = 0.7433, Regression, Logistic; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.66 to 1.78]
Statistical Analysis 108: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 32, >=30%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline average LBPI and treatment; Test type: Superiority; p = 0.0562, Regression, Logistic; Odds Ratio (OR) = 1.28, 95% CI 2-sided [0.99 to 1.65]
Statistical Analysis 109: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 11, analysis 108]; Test type: Superiority; p = 0.0274, Regression, Logistic; Odds Ratio (OR) = 1.33, 95% CI 2-sided [1.03 to 1.71]
Statistical Analysis 110: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 32, >=50%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline average LBPI and treatment; Test type: Superiority; p = 0.1206, Regression, Logistic; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.95 to 1.58]
Statistical Analysis 111: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 11, analysis 110]; Test type: Superiority; p = 0.0365, Regression, Logistic; Odds Ratio (OR) = 1.31, 95% CI 2-sided [1.02 to 1.69]
Statistical Analysis 112: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 32, >=70%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline average LBPI and treatment; Test type: Superiority; p = 0.0964, Regression, Logistic; Odds Ratio (OR) = 1.28, 95% CI 2-sided [0.96 to 1.71]
Statistical Analysis 113: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 11, analysis 112]; Test type: Superiority; p = 0.2515, Regression, Logistic; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.89 to 1.59]
Statistical Analysis 114: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 32, >=90%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline average LBPI and treatment; Test type: Superiority; p = 0.8122, Regression, Logistic; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.66 to 1.71]
Statistical Analysis 115: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 11, analysis 114]; Test type: Superiority; p = 0.1848, Regression, Logistic; Odds Ratio (OR) = 1.36, 95% CI 2-sided [0.86 to 2.13]
Statistical Analysis 116: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 40, >=30%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline average LBPI and treatment; Test type: Superiority; p = 0.2622, Regression, Logistic; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.90 to 1.49]
Statistical Analysis 117: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 11, analysis 116]; Test type: Superiority; p = 0.1579, Regression, Logistic; Odds Ratio (OR) = 1.20, 95% CI 2-sided [0.93 to 1.54]
Statistical Analysis 118: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 40, >=50%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline average LBPI and treatment; Test type: Superiority; p = 0.2773, Regression, Logistic; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.89 to 1.49]
Statistical Analysis 119: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 11, analysis 118]; Test type: Superiority; p = 0.1032, Regression, Logistic; Odds Ratio (OR) = 1.24, 95% CI 2-sided [0.96 to 1.59]
Statistical Analysis 120: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 40, >=70%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline average LBPI and treatment; Test type: Superiority; p = 0.4418, Regression, Logistic; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.84 to 1.50]
Statistical Analysis 121: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 11, analysis 120]; Test type: Superiority; p = 0.1608, Regression, Logistic; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.92 to 1.63]
Statistical Analysis 122: Comparison: Pooled Tanezumab 10 mg vs Tramadol; Week 40, >=90%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline average LBPI and treatment; Test type: Superiority; p = 0.2628, Regression, Logistic; Odds Ratio (OR) = 1.29, 95% CI 2-sided [0.83 to 2.02]
Statistical Analysis 123: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 11, analysis 122]; Test type: Superiority; p = 0.0447, Regression, Logistic; Odds Ratio (OR) = 1.55, 95% CI 2-sided [1.01 to 2.39]
Statistical Analysis 124: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 48, >=30%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline average LBPI and treatment; Test type: Superiority; p = 0.2560, Regression, Logistic; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.90 to 1.49]
Statistical Analysis 125: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 11, analysis 124]; Test type: Superiority; p = 0.1741, Regression, Logistic; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.93 to 1.53]
Statistical Analysis 126: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 48, >=50%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline average LBPI and treatment; Test type: Superiority; p = 0.1647, Regression, Logistic; Odds Ratio (OR) = 1.20, 95% CI 2-sided [0.93 to 1.55]
Statistical Analysis 127: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 11, analysis 126]; Test type: Superiority; p = 0.0619, Regression, Logistic; Odds Ratio (OR) = 1.28, 95% CI 2-sided [0.99 to 1.65]
Statistical Analysis 128: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 48, >=70%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline average LBPI and treatment; Test type: Superiority; p = 0.2025, Regression, Logistic; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.90 to 1.61]
Statistical Analysis 129: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 11, analysis 128]; Test type: Superiority; p = 0.2601, Regression, Logistic; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.88 to 1.58]
Statistical Analysis 130: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 48, >=90%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline average LBPI and treatment; Test type: Superiority; p = 0.5635, Regression, Logistic; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.73 to 1.77]
Statistical Analysis 131: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 11, analysis 130]; Test type: Superiority; p = 0.1338, Regression, Logistic; Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.91 to 2.11]
Statistical Analysis 132: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 56, >=30%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline average LBPI and treatment; Test type: Superiority; p = 0.2137, Regression, Logistic; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.91 to 1.51]
Statistical Analysis 133: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 11, analysis 132]; Test type: Superiority; p = 0.0256, Regression, Logistic; Odds Ratio (OR) = 1.33, 95% CI 2-sided [1.04 to 1.72]
Statistical Analysis 134: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 56, >=50%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline average LBPI and treatment; Test type: Superiority; p = 0.3531, Regression, Logistic; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.87 to 1.46]
Statistical Analysis 135: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 11, analysis 134]; Test type: Superiority; p = 0.0358, Regression, Logistic; Odds Ratio (OR) = 1.31, 95% CI 2-sided [1.02 to 1.70]
Statistical Analysis 136: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 56, >=70%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline average LBPI and treatment; Test type: Superiority; p = 0.1840, Regression, Logistic; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.91 to 1.62]
Statistical Analysis 137: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 11, analysis 136]; Test type: Superiority; p = 0.1250, Regression, Logistic; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.94 to 1.67]
Statistical Analysis 138: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 56, >=90%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline average LBPI and treatment; Test type: Superiority; p = 0.8266, Regression, Logistic; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.61 to 1.48]
Statistical Analysis 139: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 11, analysis 138]; Test type: Superiority; p = 0.5673, Regression, Logistic; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.74 to 1.72]

12. Secondary Outcome: Percentage of Participants Achieving RMDQ Reduction of >=30%, >=50%, >=70% and >=90% From Baseline at Weeks 2, 4, 8, 16, 24, 32, 40, 48 and 56: Mixed Baseline Observation Carried Forward (BOCF)/Last Observation Carried Forward (LOCF)
Description: RMDQ: health status measure index of how well participants with LBP are able to function with regard to daily activities. Measures pain and function using 24 items describing limitations to everyday life. Total score of RMDQ is total number of items checked ranging from 0=no disability to 24=maximum disability, higher scores=greater disability. Percentage of participants with reduction in LBPI of at least (>=) 30, 50, 70 and 90% at specified weeks compared to baseline were classified as responders to LBPI and are reported here. Pre-specified intent of study for efficacy data up to W16 was to analyze participants who received placebo from Day1 and then received tanezumab 5/10 mg at W16,together,in placebo arm.Data has been reported per four arms. Also, intent of study was to compare tanezumab Vs placebo for data up to & including W16 & comparisons of tanezumab Vs tramadol for data up to & including W56.
Time Frame: Baseline, Weeks 2, 4, 8, 16, 24, 32, 40, 48 and 56
Population: ITT population.Data were not collected after W16 in placebo arm for this outcome measure, as those who met criteria to continue, switched to active treatment with tanezumab after W16. N =participants evaluable for this OM.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 406 | 405 | 407 | 605
percentage of participants
  Week 2: At least 30% reduction | 24.1 | 32.3 | 38.3 | 29.3
  Week 2: At least 50% reduction | 13.5 | 20.0 | 21.4 | 16.9
  Week 2: At least 70% reduction | 5.7 | 10.6 | 10.3 | 6.6
  Week 2: At least 90% reduction | 1.7 | 4.2 | 5.4 | 2.3
  Week 4: At least 30% reduction | 34.5 | 46.2 | 50.4 | 39.7
  Week 4: At least 50% reduction | 19.2 | 30.9 | 34.2 | 25.3
  Week 4: At least 70% reduction | 10.1 | 17.5 | 21.1 | 10.9
  Week 4: At least 90% reduction | 4.2 | 7.9 | 9.6 | 3.1
  Week 8: At least 30% reduction | 41.1 | 52.8 | 56.8 | 48.6
  Week 8: At least 50% reduction | 26.4 | 36.8 | 40.8 | 33.4
  Week 8: At least 70% reduction | 12.8 | 23.2 | 24.8 | 16.4
  Week 8: At least 90% reduction | 4.9 | 12.1 | 13.8 | 6.4
  Week 16: At least 30% reduction | 48.5 | 58.3 | 62.2 | 52.2
  Week 16: At least 50% reduction | 34.7 | 46.7 | 48.2 | 38.7
  Week 16: At least 70% reduction | 20.7 | 32.1 | 34.6 | 22.3
  Week 16: At least 90% reduction | 9.1 | 17.0 | 15.5 | 8.6
  Week 24: At least 30% reduction: number analyzed (Participants) | 0 | 405 | 407 | 605
  Week 24: At least 30% reduction |  | 50.1 | 53.3 | 44.8
  Week 24: At least 50% reduction: number analyzed (Participants) | 0 | 405 | 407 | 605
  Week 24: At least 50% reduction |  | 42.5 | 45.0 | 34.0
  Week 24: At least 70% reduction: number analyzed (Participants) | 0 | 405 | 407 | 605
  Week 24: At least 70% reduction |  | 29.4 | 31.7 | 20.7
  Week 24: At least 90% reduction: number analyzed (Participants) | 0 | 405 | 407 | 605
  Week 24: At least 90% reduction |  | 16.5 | 18.4 | 8.3
  Week 32: At least 30% reduction: number analyzed (Participants) | 0 | 405 | 407 | 605
  Week 32: At least 30% reduction |  | 48.6 | 49.4 | 43.0
  Week 32: At least 50% reduction: number analyzed (Participants) | 0 | 405 | 407 | 605
  Week 32: At least 50% reduction |  | 42.0 | 44.7 | 35.9
  Week 32: At least 70% reduction: number analyzed (Participants) | 0 | 405 | 407 | 605
  Week 32: At least 70% reduction |  | 29.1 | 31.9 | 22.5
  Week 32: At least 90% reduction: number analyzed (Participants) | 0 | 405 | 407 | 605
  Week 32: At least 90% reduction |  | 17.8 | 17.9 | 11.6
  Week 40: At least 30% reduction: number analyzed (Participants) | 0 | 405 | 407 | 605
  Week 40: At least 30% reduction |  | 44.9 | 48.2 | 41.5
  Week 40: At least 50% reduction: number analyzed (Participants) | 0 | 405 | 407 | 605
  Week 40: At least 50% reduction |  | 38.5 | 40.8 | 34.4
  Week 40: At least 70% reduction: number analyzed (Participants) | 0 | 405 | 407 | 605
  Week 40: At least 70% reduction |  | 29.9 | 29.5 | 23.3
  Week 40: At least 90% reduction: number analyzed (Participants) | 0 | 405 | 407 | 605
  Week 40: At least 90% reduction |  | 17.3 | 17.2 | 11.4
  Week 48: At least 30% reduction: number analyzed (Participants) | 0 | 405 | 407 | 605
  Week 48: At least 30% reduction |  | 43.0 | 45.2 | 40.8
  Week 48: At least 50% reduction: number analyzed (Participants) | 0 | 405 | 407 | 605
  Week 48: At least 50% reduction |  | 38.0 | 37.8 | 33.2
  Week 48: At least 70% reduction: number analyzed (Participants) | 0 | 405 | 407 | 605
  Week 48: At least 70% reduction |  | 28.4 | 29.5 | 22.0
  Week 48: At least 90% reduction: number analyzed (Participants) | 0 | 405 | 407 | 605
  Week 48: At least 90% reduction |  | 16.3 | 17.7 | 11.4
  Week 56: At least 30% reduction: number analyzed (Participants) | 0 | 405 | 407 | 605
  Week 56: At least 30% reduction |  | 41.2 | 46.4 | 41.5
  Week 56: At least 50% reduction: number analyzed (Participants) | 0 | 405 | 407 | 605
  Week 56: At least 50% reduction |  | 36.5 | 38.8 | 32.2
  Week 56: At least 70% reduction: number analyzed (Participants) | 0 | 405 | 407 | 605
  Week 56: At least 70% reduction |  | 27.9 | 28.5 | 22.3
  Week 56: At least 90% reduction: number analyzed (Participants) | 0 | 405 | 407 | 605
  Week 56: At least 90% reduction |  | 17.8 | 18.7 | 11.7
Statistical Analysis 1: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 2, >=30%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline RMDQ, baseline average LBPI and treatment; Test type: Superiority; p = 0.0076, Regression, Logistic; Odds Ratio (OR) = 1.53, 95% CI 2-sided [1.12 to 2.08]
Statistical Analysis 2: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 1.98, 95% CI 2-sided [1.46 to 2.69]
Statistical Analysis 3: Comparison: Placebo vs Tramadol; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p = 0.0700, Regression, Logistic; Odds Ratio (OR) = 1.31, 95% CI 2-sided [0.98 to 1.74]
Statistical Analysis 4: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p = 0.2655, Regression, Logistic; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.89 to 1.54]
Statistical Analysis 5: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p = 0.0022, Regression, Logistic; Odds Ratio (OR) = 1.52, 95% CI 2-sided [1.16 to 1.98]
Statistical Analysis 6: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 2, >=50%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline RMDQ, baseline average LBPI and treatment; Test type: Superiority; p = 0.0125, Regression, Logistic; Odds Ratio (OR) = 1.61, 95% CI 2-sided [1.11 to 2.35]
Statistical Analysis 7: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 12, analysis 6]; Test type: Superiority; p = 0.0032, Regression, Logistic; Odds Ratio (OR) = 1.75, 95% CI 2-sided [1.21 to 2.54]
Statistical Analysis 8: Comparison: Placebo vs Tramadol; [analysis description as in outcome 12, analysis 6]; Test type: Superiority; p = 0.1528, Regression, Logistic; Odds Ratio (OR) = 1.30, 95% CI 2-sided [0.91 to 1.85]
Statistical Analysis 9: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 12, analysis 6]; Test type: Superiority; p = 0.1863, Regression, Logistic; Odds Ratio (OR) = 1.24, 95% CI 2-sided [0.90 to 1.72]
Statistical Analysis 10: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 12, analysis 6]; Test type: Superiority; p = 0.0667, Regression, Logistic; Odds Ratio (OR) = 1.35, 95% CI 2-sided [0.98 to 1.86]
Statistical Analysis 11: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 2, >=70%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline RMDQ, baseline average LBPI and treatment; Test type: Superiority; p = 0.0101, Regression, Logistic; Odds Ratio (OR) = 2.00, 95% CI 2-sided [1.18 to 3.39]
Statistical Analysis 12: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 12, analysis 11]; Test type: Superiority; p = 0.0162, Regression, Logistic; Odds Ratio (OR) = 1.91, 95% CI 2-sided [1.13 to 3.25]
Statistical Analysis 13: Comparison: Placebo vs Tramadol; [analysis description as in outcome 12, analysis 11]; Test type: Superiority; p = 0.5599, Regression, Logistic; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.69 to 1.99]
Statistical Analysis 14: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 12, analysis 11]; Test type: Superiority; p = 0.0202, Regression, Logistic; Odds Ratio (OR) = 1.71, 95% CI 2-sided [1.09 to 2.68]
Statistical Analysis 15: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 12, analysis 11]; Test type: Superiority; p = 0.0335, Regression, Logistic; Odds Ratio (OR) = 1.64, 95% CI 2-sided [1.04 to 2.57]
Statistical Analysis 16: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 2, >=90%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline RMDQ, baseline average LBPI and treatment; Test type: Superiority; p = 0.0416, Regression, Logistic; Odds Ratio (OR) = 2.53, 95% CI 2-sided [1.04 to 6.17]
Statistical Analysis 17: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 12, analysis 16]; Test type: Superiority; p = 0.0075, Regression, Logistic; Odds Ratio (OR) = 3.24, 95% CI 2-sided [1.37 to 7.69]
Statistical Analysis 18: Comparison: Placebo vs Tramadol; [analysis description as in outcome 12, analysis 16]; Test type: Superiority; p = 0.5374, Regression, Logistic; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.53 to 3.34]
Statistical Analysis 19: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 12, analysis 16]; Test type: Superiority; p = 0.0820, Regression, Logistic; Odds Ratio (OR) = 1.89, 95% CI 2-sided [0.92 to 3.89]
Statistical Analysis 20: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 12, analysis 16]; Test type: Superiority; p = 0.0108, Regression, Logistic; Odds Ratio (OR) = 2.43, 95% CI 2-sided [1.23 to 4.81]
Statistical Analysis 21: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 4, >=30%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline RMDQ, baseline average LBPI and treatment; Test type: Superiority; p = 0.0006, Regression, Logistic; Odds Ratio (OR) = 1.65, 95% CI 2-sided [1.24 to 2.20]
Statistical Analysis 22: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 12, analysis 21]; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 1.95, 95% CI 2-sided [1.47 to 2.59]
Statistical Analysis 23: Comparison: Placebo vs Tramadol; [analysis description as in outcome 12, analysis 21]; Test type: Superiority; p = 0.0963, Regression, Logistic; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.96 to 1.63]
Statistical Analysis 24: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 12, analysis 21]; Test type: Superiority; p = 0.0332, Regression, Logistic; Odds Ratio (OR) = 1.32, 95% CI 2-sided [1.02 to 1.71]
Statistical Analysis 25: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 12, analysis 21]; Test type: Superiority; p = 0.0007, Regression, Logistic; Odds Ratio (OR) = 1.56, 95% CI 2-sided [1.21 to 2.01]
Statistical Analysis 26: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 4, >=50%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline RMDQ, baseline average LBPI and treatment; Test type: Superiority; p = 0.0001, Regression, Logistic; Odds Ratio (OR) = 1.90, 95% CI 2-sided [1.37 to 2.64]
Statistical Analysis 27: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 12, analysis 26]; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 2.21, 95% CI 2-sided [1.60 to 3.05]
Statistical Analysis 28: Comparison: Placebo vs Tramadol; [analysis description as in outcome 12, analysis 26]; Test type: Superiority; p = 0.0235, Regression, Logistic; Odds Ratio (OR) = 1.43, 95% CI 2-sided [1.05 to 1.95]
Statistical Analysis 29: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 12, analysis 26]; Test type: Superiority; p = 0.0459, Regression, Logistic; Odds Ratio (OR) = 1.33, 95% CI 2-sided [1.01 to 1.76]
Statistical Analysis 30: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 12, analysis 26]; Test type: Superiority; p = 0.0020, Regression, Logistic; Odds Ratio (OR) = 1.54, 95% CI 2-sided [1.17 to 2.04]
Statistical Analysis 31: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 4, >=70%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline RMDQ, baseline average LBPI and treatment; Test type: Superiority; p = 0.0019, Regression, Logistic; Odds Ratio (OR) = 1.93, 95% CI 2-sided [1.27 to 2.91]
Statistical Analysis 32: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 12, analysis 31]; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 2.42, 95% CI 2-sided [1.62 to 3.62]
Statistical Analysis 33: Comparison: Placebo vs Tramadol; [analysis description as in outcome 12, analysis 31]; Test type: Superiority; p = 0.6765, Regression, Logistic; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.72 to 1.65]
Statistical Analysis 34: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 12, analysis 31]; Test type: Superiority; p = 0.0022, Regression, Logistic; Odds Ratio (OR) = 1.76, 95% CI 2-sided [1.23 to 2.54]
Statistical Analysis 35: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 12, analysis 31]; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 2.21, 95% CI 2-sided [1.56 to 3.15]
Statistical Analysis 36: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 4, >=90%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline RMDQ, baseline average LBPI and treatment; Test type: Superiority; p = 0.0270, Regression, Logistic; Odds Ratio (OR) = 1.98, 95% CI 2-sided [1.08 to 3.63]
Statistical Analysis 37: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 12, analysis 36]; Test type: Superiority; p = 0.0030, Regression, Logistic; Odds Ratio (OR) = 2.43, 95% CI 2-sided [1.35 to 4.38]
Statistical Analysis 38: Comparison: Placebo vs Tramadol; [analysis description as in outcome 12, analysis 36]; Test type: Superiority; p = 0.3770, Regression, Logistic; Odds Ratio (OR) = 0.74, 95% CI 2-sided [0.38 to 1.44]
Statistical Analysis 39: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 12, analysis 36]; Test type: Superiority; p = 0.0009, Regression, Logistic; Odds Ratio (OR) = 2.68, 95% CI 2-sided [1.49 to 4.79]
Statistical Analysis 40: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 12, analysis 36]; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 3.29, 95% CI 2-sided [1.87 to 5.78]
Statistical Analysis 41: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 8, >=30%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline RMDQ, baseline average LBPI and treatment; Test type: Superiority; p = 0.0011, Regression, Logistic; Odds Ratio (OR) = 1.59, 95% CI 2-sided [1.20 to 2.10]
Statistical Analysis 42: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 12, analysis 41]; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 1.87, 95% CI 2-sided [1.41 to 2.47]
Statistical Analysis 43: Comparison: Placebo vs Tramadol; [analysis description as in outcome 12, analysis 41]; Test type: Superiority; p = 0.0273, Regression, Logistic; Odds Ratio (OR) = 1.33, 95% CI 2-sided [1.03 to 1.72]
Statistical Analysis 44: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 12, analysis 41]; Test type: Superiority; p = 0.1736, Regression, Logistic; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.93 to 1.54]
Statistical Analysis 45: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 12, analysis 41]; Test type: Superiority; p = 0.0092, Regression, Logistic; Odds Ratio (OR) = 1.40, 95% CI 2-sided [1.09 to 1.81]
Statistical Analysis 46: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 8, >=50%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline RMDQ, baseline average LBPI and treatment; Test type: Superiority; p = 0.0015, Regression, Logistic; Odds Ratio (OR) = 1.63, 95% CI 2-sided [1.20 to 2.20]
Statistical Analysis 47: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 12, analysis 46]; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 1.95, 95% CI 2-sided [1.45 to 2.63]
Statistical Analysis 48: Comparison: Placebo vs Tramadol; [analysis description as in outcome 12, analysis 46]; Test type: Superiority; p = 0.0164, Regression, Logistic; Odds Ratio (OR) = 1.41, 95% CI 2-sided [1.06 to 1.86]
Statistical Analysis 49: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 12, analysis 46]; Test type: Superiority; p = 0.2857, Regression, Logistic; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.89 to 1.51]
Statistical Analysis 50: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 12, analysis 46]; Test type: Superiority; p = 0.0149, Regression, Logistic; Odds Ratio (OR) = 1.38, 95% CI 2-sided [1.07 to 1.80]
Statistical Analysis 51: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 8, >=70%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline RMDQ, baseline average LBPI and treatment; Test type: Superiority; p = 0.0001, Regression, Logistic; Odds Ratio (OR) = 2.08, 95% CI 2-sided [1.43 to 3.02]
Statistical Analysis 52: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 12, analysis 51]; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 2.27, 95% CI 2-sided [1.57 to 3.28]
Statistical Analysis 53: Comparison: Placebo vs Tramadol; [analysis description as in outcome 12, analysis 51]; Test type: Superiority; p = 0.1180, Regression, Logistic; Odds Ratio (OR) = 1.34, 95% CI 2-sided [0.93 to 1.92]
Statistical Analysis 54: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 12, analysis 51]; Test type: Superiority; p = 0.0062, Regression, Logistic; Odds Ratio (OR) = 1.56, 95% CI 2-sided [1.13 to 2.14]
Statistical Analysis 55: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 12, analysis 51]; Test type: Superiority; p = 0.0009, Regression, Logistic; Odds Ratio (OR) = 1.70, 95% CI 2-sided [1.24 to 2.32]
Statistical Analysis 56: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 8, >=90%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline RMDQ, baseline average LBPI and treatment; Test type: Superiority; p = 0.0003, Regression, Logistic; Odds Ratio (OR) = 2.69, 95% CI 2-sided [1.56 to 4.61]
Statistical Analysis 57: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 12, analysis 56]; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 3.10, 95% CI 2-sided [1.82 to 5.28]
Statistical Analysis 58: Comparison: Placebo vs Tramadol; [analysis description as in outcome 12, analysis 56]; Test type: Superiority; p = 0.3120, Regression, Logistic; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.76 to 2.32]
Statistical Analysis 59: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 12, analysis 56]; Test type: Superiority; p = 0.0019, Regression, Logistic; Odds Ratio (OR) = 2.02, 95% CI 2-sided [1.30 to 3.14]
Statistical Analysis 60: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 12, analysis 56]; Test type: Superiority; p = 0.0001, Regression, Logistic; Odds Ratio (OR) = 2.33, 95% CI 2-sided [1.52 to 3.59]
Statistical Analysis 61: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 16, >=30%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline RMDQ, baseline average LBPI and treatment; Test type: Superiority; p = 0.0064, Regression, Logistic; Odds Ratio (OR) = 1.47, 95% CI 2-sided [1.12 to 1.95]
Statistical Analysis 62: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 12, analysis 61]; Test type: Superiority; p = 0.0001, Regression, Logistic; Odds Ratio (OR) = 1.74, 95% CI 2-sided [1.32 to 2.31]
Statistical Analysis 63: Comparison: Placebo vs Tramadol; [analysis description as in outcome 12, analysis 61]; Test type: Superiority; p = 0.2757, Regression, Logistic; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.89 to 1.48]
Statistical Analysis 64: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 12, analysis 61]; Test type: Superiority; p = 0.0575, Regression, Logistic; Odds Ratio (OR) = 1.28, 95% CI 2-sided [0.99 to 1.65]
Statistical Analysis 65: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 12, analysis 61]; Test type: Superiority; p = 0.0015, Regression, Logistic; Odds Ratio (OR) = 1.52, 95% CI 2-sided [1.17 to 1.96]
Statistical Analysis 66: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 16, >=50%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline RMDQ, baseline average LBPI and treatment; Test type: Superiority; p = 0.0007, Regression, Logistic; Odds Ratio (OR) = 1.63, 95% CI 2-sided [1.23 to 2.16]
Statistical Analysis 67: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 12, analysis 66]; Test type: Superiority; p = 0.0001, Regression, Logistic; Odds Ratio (OR) = 1.74, 95% CI 2-sided [1.31 to 2.31]
Statistical Analysis 68: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 12, analysis 66]; Test type: Superiority; p = 0.0124, Regression, Logistic; Odds Ratio (OR) = 1.38, 95% CI 2-sided [1.07 to 1.79]
Statistical Analysis 69: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 12, analysis 66]; Test type: Superiority; p = 0.0025, Regression, Logistic; Odds Ratio (OR) = 1.48, 95% CI 2-sided [1.15 to 1.91]
Statistical Analysis 70: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 16, >=70%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline RMDQ, baseline average LBPI and treatment; Test type: Superiority; p = 0.0002, Regression, Logistic; Odds Ratio (OR) = 1.82, 95% CI 2-sided [1.33 to 2.51]
Statistical Analysis 71: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 12, analysis 70]; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 2.03, 95% CI 2-sided [1.48 to 2.79]
Statistical Analysis 72: Comparison: Placebo vs Tramadol; [analysis description as in outcome 12, analysis 70]; Test type: Superiority; p = 0.5701, Regression, Logistic; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.80 to 1.49]
Statistical Analysis 73: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 12, analysis 70]; Test type: Superiority; p = 0.0004, Regression, Logistic; Odds Ratio (OR) = 1.67, 95% CI 2-sided [1.26 to 2.22]
Statistical Analysis 74: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 12, analysis 70]; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 1.86, 95% CI 2-sided [1.40 to 2.46]
Statistical Analysis 75: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 16, >=90%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline RMDQ, baseline average LBPI and treatment; Test type: Superiority; p = 0.0008, Regression, Logistic; Odds Ratio (OR) = 2.07, 95% CI 2-sided [1.35 to 3.17]
Statistical Analysis 76: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 12, analysis 75]; Test type: Superiority; p = 0.0059, Regression, Logistic; Odds Ratio (OR) = 1.84, 95% CI 2-sided [1.19 to 2.83]
Statistical Analysis 77: Comparison: Placebo vs Tramadol; [analysis description as in outcome 12, analysis 75]; Test type: Superiority; p = 0.7741, Regression, Logistic; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.60 to 1.46]
Statistical Analysis 78: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 12, analysis 75]; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 2.21, 95% CI 2-sided [1.50 to 3.25]
Statistical Analysis 79: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 12, analysis 75]; Test type: Superiority; p = 0.0008, Regression, Logistic; Odds Ratio (OR) = 1.96, 95% CI 2-sided [1.32 to 2.90]
Statistical Analysis 80: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 24, >=30%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline RMDQ, baseline average LBPI and treatment; Test type: Superiority; p = 0.0890, Regression, Logistic; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.97 to 1.60]
Statistical Analysis 81: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 12, analysis 80]; Test type: Superiority; p = 0.0067, Regression, Logistic; Odds Ratio (OR) = 1.42, 95% CI 2-sided [1.10 to 1.83]
Statistical Analysis 82: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 24, >=50%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline RMDQ, baseline average LBPI and treatment; Test type: Superiority; p = 0.0072, Regression, Logistic; Odds Ratio (OR) = 1.43, 95% CI 2-sided [1.10 to 1.85]
Statistical Analysis 83: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 12, analysis 82]; Test type: Superiority; p = 0.0004, Regression, Logistic; Odds Ratio (OR) = 1.59, 95% CI 2-sided [1.23 to 2.06]
Statistical Analysis 84: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 24, >=70%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline RMDQ, baseline average LBPI and treatment; Test type: Superiority; p = 0.0013, Regression, Logistic; Odds Ratio (OR) = 1.61, 95% CI 2-sided [1.20 to 2.15]
Statistical Analysis 85: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 12, analysis 84]; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 1.79, 95% CI 2-sided [1.34 to 2.39]
Statistical Analysis 86: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 24, >=90%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline RMDQ, baseline average LBPI and treatment; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 2.23, 95% CI 2-sided [1.51 to 3.30]
Statistical Analysis 87: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 12, analysis 86]; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 2.53, 95% CI 2-sided [1.72 to 3.71]
Statistical Analysis 88: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 32, >=30%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline RMDQ, baseline average LBPI and treatment; Test type: Superiority; p = 0.0732, Regression, Logistic; Odds Ratio (OR) = 1.26, 95% CI 2-sided [0.98 to 1.62]
Statistical Analysis 89: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 12, analysis 88]; Test type: Superiority; p = 0.0399, Regression, Logistic; Odds Ratio (OR) = 1.30, 95% CI 2-sided [1.01 to 1.68]
Statistical Analysis 90: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 32, >=50%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline RMDQ, baseline average LBPI and treatment; Test type: Superiority; p = 0.0536, Regression, Logistic; Odds Ratio (OR) = 1.29, 95% CI 2-sided [1.00 to 1.67]
Statistical Analysis 91: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 12, analysis 90]; Test type: Superiority; p = 0.0043, Regression, Logistic; Odds Ratio (OR) = 1.45, 95% CI 2-sided [1.12 to 1.88]
Statistical Analysis 92: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 32, >=70%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline RMDQ, baseline average LBPI and treatment; Test type: Superiority; p = 0.0143, Regression, Logistic; Odds Ratio (OR) = 1.43, 95% CI 2-sided [1.07 to 1.91]
Statistical Analysis 93: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 12, analysis 92]; Test type: Superiority; p = 0.0007, Regression, Logistic; Odds Ratio (OR) = 1.63, 95% CI 2-sided [1.23 to 2.16]
Statistical Analysis 94: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 32, >=90%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline RMDQ, baseline average LBPI and treatment; Test type: Superiority; p = 0.0050, Regression, Logistic; Odds Ratio (OR) = 1.67, 95% CI 2-sided [1.17 to 2.38]
Statistical Analysis 95: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 12, analysis 94]; Test type: Superiority; p = 0.0043, Regression, Logistic; Odds Ratio (OR) = 1.68, 95% CI 2-sided [1.18 to 2.40]
Statistical Analysis 96: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 40, >=30%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline RMDQ, baseline average LBPI and treatment; Test type: Superiority; p = 0.2777, Regression, Logistic; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.89 to 1.48]
Statistical Analysis 97: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 12, analysis 96]; Test type: Superiority; p = 0.0326, Regression, Logistic; Odds Ratio (OR) = 1.32, 95% CI 2-sided [1.02 to 1.70]
Statistical Analysis 98: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 40, >=50%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline RMDQ, baseline average LBPI and treatment; Test type: Superiority; p = 0.1823, Regression, Logistic; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.92 to 1.55]
Statistical Analysis 99: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 12, analysis 98]; Test type: Superiority; p = 0.0350, Regression, Logistic; Odds Ratio (OR) = 1.32, 95% CI 2-sided [1.02 to 1.71]
Statistical Analysis 100: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 40, >=70%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline RMDQ, baseline average LBPI and treatment; Test type: Superiority; p = 0.0164, Regression, Logistic; Odds Ratio (OR) = 1.42, 95% CI 2-sided [1.07 to 1.88]
Statistical Analysis 101: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 12, analysis 100]; Test type: Superiority; p = 0.0257, Regression, Logistic; Odds Ratio (OR) = 1.38, 95% CI 2-sided [1.04 to 1.84]
Statistical Analysis 102: Comparison: Pooled Tanezumab 10 mg vs Tramadol; Week 40, >=90%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline RMDQ, baseline average LBPI and treatment; Test type: Superiority; p = 0.0070, Regression, Logistic; Odds Ratio (OR) = 1.64, 95% CI 2-sided [1.14 to 2.35]
Statistical Analysis 103: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 12, analysis 102]; Test type: Superiority; p = 0.0085, Regression, Logistic; Odds Ratio (OR) = 1.62, 95% CI 2-sided [1.13 to 2.32]
Statistical Analysis 104: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 48, >=30%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline RMDQ, baseline average LBPI and treatment; Test type: Superiority; p = 0.4925, Regression, Logistic; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.85 to 1.41]
Statistical Analysis 105: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 12, analysis 104]; Test type: Superiority; p = 0.1534, Regression, Logistic; Odds Ratio (OR) = 1.20, 95% CI 2-sided [0.93 to 1.55]
Statistical Analysis 106: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 48, >=50%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline RMDQ, baseline average LBPI and treatment; Test type: Superiority; p = 0.1202, Regression, Logistic; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.95 to 1.60]
Statistical Analysis 107: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 12, analysis 106]; Test type: Superiority; p = 0.1222, Regression, Logistic; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.95 to 1.60]
Statistical Analysis 108: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 48, >=70%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline RMDQ, baseline average LBPI and treatment; Test type: Superiority; p = 0.0179, Regression, Logistic; Odds Ratio (OR) = 1.42, 95% CI 2-sided [1.06 to 1.90]
Statistical Analysis 109: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 12, analysis 108]; Test type: Superiority; p = 0.0065, Regression, Logistic; Odds Ratio (OR) = 1.49, 95% CI 2-sided [1.12 to 1.99]
Statistical Analysis 110: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 48, >=90%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline RMDQ, baseline average LBPI and treatment; Test type: Superiority; p = 0.0223, Regression, Logistic; Odds Ratio (OR) = 1.53, 95% CI 2-sided [1.06 to 2.20]
Statistical Analysis 111: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 12, analysis 110]; Test type: Superiority; p = 0.0045, Regression, Logistic; Odds Ratio (OR) = 1.68, 95% CI 2-sided [1.17 to 2.40]
Statistical Analysis 112: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 56, >=30%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline RMDQ, baseline average LBPI and treatment; Test type: Superiority; p = 0.9385, Regression, Logistic; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.77 to 1.28]
Statistical Analysis 113: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 12, analysis 112]; Test type: Superiority; p = 0.1093, Regression, Logistic; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.95 to 1.59]
Statistical Analysis 114: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 56, >=50%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline RMDQ, baseline average LBPI and treatment; Test type: Superiority; p = 0.1631, Regression, Logistic; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.93 to 1.57]
Statistical Analysis 115: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 12, analysis 114]; Test type: Superiority; p = 0.0285, Regression, Logistic; Odds Ratio (OR) = 1.34, 95% CI 2-sided [1.03 to 1.74]
Statistical Analysis 116: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 56, >=70%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline RMDQ, baseline average LBPI and treatment; Test type: Superiority; p = 0.0389, Regression, Logistic; Odds Ratio (OR) = 1.36, 95% CI 2-sided [1.02 to 1.81]
Statistical Analysis 117: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 12, analysis 116]; Test type: Superiority; p = 0.0240, Regression, Logistic; Odds Ratio (OR) = 1.39, 95% CI 2-sided [1.04 to 1.86]
Statistical Analysis 118: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 56, >=90%: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline RMDQ, baseline average LBPI and treatment; Test type: Superiority; p = 0.0063, Regression, Logistic; Odds Ratio (OR) = 1.64, 95% CI 2-sided [1.15 to 2.34]
Statistical Analysis 119: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 12, analysis 118]; Test type: Superiority; p = 0.0021, Regression, Logistic; Odds Ratio (OR) = 1.74, 95% CI 2-sided [1.22 to 2.47]

13. Secondary Outcome: Percentage of Participants With Cumulative Percent Change From Baseline in Roland Morris Disability Questionnaire (RMDQ) Score at Weeks 16, 24 and 56
Description: The RMDQ is a self-administered, widely used health status measure index of how well participants with LBP are able to function with regard to daily activities. It measures pain and function, using 24 items describing limitations to everyday life that can be caused by LBP. The total score of the RMDQ is the total number of items checked ranging from 0 (no disability) to 24 (maximum disability), where higher scores indicated greater disability. Percentage of participants with cumulative reduction (as percent) (>0 %; >= 10 %, 20 %, 30 %, 40 %, 50 %, 60 %, 70 %, 80 %, 90% and =100 %) in RMDQ from Baseline to weeks 16, 24 and 56 were reported, participants (%) are reported more than once in categories specified.Pre-specified intent of study for efficacy data up to W16 was to analyze participants who received placebo from Day1 and then received tanezumab 5/10 mg at W16,together,in placebo arm.Data has been reported per four arms.
Time Frame: Baseline, Weeks 16, 24 and 56
Population: ITT population.Data were not collected after W16 in placebo arm for this OM,as those who met criteria to continue,switched to active treatment with tanezumab(tan) after W16.N=participants evaluable for this OM.Intent of study was to compare tan V placebo for data up to & including W16 & comparisons of tan Vs tramadol for data up to & including W56.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 406 | 405 | 407 | 605
percentage of participants
  Week 16: >=0% | 71.2 | 76.8 | 83.5 | 71.2
  Week 16: >=10% | 68.2 | 72.6 | 78.4 | 66.3
  Week 16: >=20% | 60.6 | 65.4 | 70.3 | 59.3
  Week 16: >=30% | 48.5 | 58.3 | 62.2 | 52.2
  Week 16: >=40% | 42.1 | 53.1 | 53.3 | 44.3
  Week 16: >=50% | 34.7 | 46.7 | 48.2 | 38.7
  Week 16: >=60% | 26.1 | 38.0 | 41.0 | 30.9
  Week 16: >=70% | 20.7 | 32.1 | 34.6 | 22.3
  Week 16: >=80% | 14.8 | 23.2 | 26.5 | 15.5
  Week 16: >=90% | 9.1 | 17.0 | 15.5 | 8.6
  Week 16: =100% | 6.4 | 13.3 | 9.3 | 4.8
  Week 24: >=0%: number analyzed (Participants) | 0 | 405 | 407 | 605
  Week 24: >=0% |  | 60.5 | 64.6 | 57.7
  Week 24: >=10%: number analyzed (Participants) | 0 | 405 | 407 | 605
  Week 24: >=10% |  | 58.3 | 61.9 | 55.7
  Week 24: >=20%: number analyzed (Participants) | 0 | 405 | 407 | 605
  Week 24: >=20% |  | 54.6 | 56.5 | 51.1
  Week 24: >=30%: number analyzed (Participants) | 0 | 405 | 407 | 605
  Week 24: >=30% |  | 50.1 | 53.3 | 44.8
  Week 24: >=40%: number analyzed (Participants) | 0 | 405 | 407 | 605
  Week 24: >=40% |  | 46.7 | 48.2 | 39.5
  Week 24: >=50%: number analyzed (Participants) | 0 | 405 | 407 | 605
  Week 24: >=50% |  | 42.5 | 45.0 | 34.0
  Week 24: >=60%: number analyzed (Participants) | 0 | 405 | 407 | 605
  Week 24: >=60% |  | 35.8 | 38.6 | 26.1
  Week 24: >=70%: number analyzed (Participants) | 0 | 405 | 407 | 605
  Week 24: >=70% |  | 29.4 | 31.7 | 20.7
  Week 24: >=80%: number analyzed (Participants) | 0 | 405 | 407 | 605
  Week 24: >=80% |  | 22.2 | 25.3 | 14.2
  Week 24: >=90%: number analyzed (Participants) | 0 | 405 | 407 | 605
  Week 24: >=90% |  | 16.5 | 18.4 | 8.3
  Week 24: =100%: number analyzed (Participants) | 0 | 405 | 407 | 605
  Week 24: =100% |  | 11.6 | 11.5 | 5.6
  Week 56: >0%: number analyzed (Participants) | 0 | 405 | 407 | 605
  Week 56: >0% |  | 51.6 | 56.5 | 52.6
  Week 56: >=10%: number analyzed (Participants) | 0 | 405 | 407 | 605
  Week 56: >=10% |  | 50.1 | 54.8 | 49.9
  Week 56: >=20%: number analyzed (Participants) | 0 | 405 | 407 | 605
  Week 56: >=20% |  | 46.2 | 50.9 | 46.0
  Week 56: >=30%: number analyzed (Participants) | 0 | 405 | 407 | 605
  Week 56: >=30% |  | 41.2 | 46.4 | 41.5
  Week 56: >=40%: number analyzed (Participants) | 0 | 405 | 407 | 605
  Week 56: >=40% |  | 38.0 | 42.5 | 36.2
  Week 56: >=50%: number analyzed (Participants) | 0 | 405 | 407 | 605
  Week 56: >=50% |  | 36.5 | 38.8 | 32.2
  Week 56: >=60%: number analyzed (Participants) | 0 | 405 | 407 | 605
  Week 56: >=60% |  | 31.9 | 33.2 | 27.1
  Week 56: >=70%: number analyzed (Participants) | 0 | 405 | 407 | 605
  Week 56: >=70% |  | 27.9 | 28.5 | 22.3
  Week 56: >=80%: number analyzed (Participants) | 0 | 405 | 407 | 605
  Week 56: >=80% |  | 22.7 | 24.3 | 17.2
  Week 56: >=90%: number analyzed (Participants) | 0 | 405 | 407 | 605
  Week 56: >=90% |  | 17.8 | 18.7 | 11.7
  Week 56: =100%: number analyzed (Participants) | 0 | 405 | 407 | 605
  Week 56: =100% |  | 13.8 | 14.0 | 7.4

14. Secondary Outcome: Change From Baseline in Brief Pain Inventory-short Form (BPI-sf) Score Worst Pain at Weeks 2, 4, 8, 16, 24, 32, 40, 48 and 56
Description: BPI-sf is a self-administered questionnaire developed to assess the severity of pain and pain interference on daily functions during 24 hours prior to evaluation. Severity of pain was measured based on questions 1 to 4 of pain at its 'worst', 'least', 'average' and 'right now'. For the Worst Pain item of the BPI-sf scale (11 point NRS scale; range: 0 [no pain] to 10 [pain as bad as you can imagine]), participants were asked to rate their pain by marking an "X" in one of the boxes that best described their pain at its worst, during 24 hours prior to evaluation, higher scores indicated greater pain severity. Question 5 (7-items) assessed level of pain interference on daily activities.Pre-specified intent of study for efficacy data up to W16 was to analyze participants who received placebo from Day1 and then received tanezumab 5/10 mg at W16,together,in placebo arm.Data has been reported per four arms.
Time Frame: Baseline, Weeks 2, 4, 8, 16, 24, 32, 40, 48 and 56
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 406 | 407 | 407 | 605
units on a scale
  Change at Week 2 | -1.17 (0.10) | -1.66 (0.10) | -1.76 (0.10) | -1.40 (0.09)
  Change at Week 4 | -1.73 (0.12) | -2.30 (0.12) | -2.50 (0.12) | -1.98 (0.11)
  Change at Week 8 | -2.11 (0.13) | -2.57 (0.13) | -2.86 (0.13) | -2.37 (0.11)
  Change at Week 16 | -2.67 (0.15) | -3.18 (0.14) | -3.21 (0.14) | -2.90 (0.12)
  Change at Week 24: number analyzed (Participants) | 0 | 407 | 407 | 605
  Change at Week 24 |  | -2.81 (0.17) | -3.01 (0.17) | -2.66 (0.14)
  Change at Week 32: number analyzed (Participants) | 0 | 407 | 407 | 605
  Change at Week 32 |  | -2.88 (0.17) | -2.95 (0.17) | -2.63 (0.15)
  Change at Week 40: number analyzed (Participants) | 0 | 407 | 407 | 605
  Change at Week 40 |  | -2.70 (0.18) | -2.78 (0.18) | -2.51 (0.15)
  Change at Week 48: number analyzed (Participants) | 0 | 407 | 407 | 605
  Change at Week 48 |  | -2.66 (0.19) | -2.73 (0.18) | -2.44 (0.15)
  Change at Week 56: number analyzed (Participants) | 0 | 407 | 407 | 605
  Change at Week 56 |  | -2.66 (0.19) | -2.74 (0.18) | -2.45 (0.15)
Statistical Analysis 1: Comparison: Placebo vs Pooled Tanezumab 5 mg; Change at Week 2: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf worst pain, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.0003, ANCOVA; LS Mean Difference = -0.49, 95% CI 2-sided [-0.75 to -0.22], Standard Error of Mean 0.13
Statistical Analysis 2: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 14, analysis 1]; Test type: Superiority; p < .0001, ANCOVA; LS Mean Difference = -0.59, 95% CI 2-sided [-0.85 to -0.33], Standard Error of Mean 0.13
Statistical Analysis 3: Comparison: Placebo vs Tramadol; [analysis description as in outcome 14, analysis 1]; Test type: Superiority; p = 0.0615, ANCOVA; LS Mean Difference = -0.23, 95% CI 2-sided [-0.47 to 0.01], Standard Error of Mean 0.12
Statistical Analysis 4: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 14, analysis 1]; Test type: Superiority; p = 0.0356, ANCOVA; LS Mean Difference = -0.26, 95% CI 2-sided [-0.50 to -0.02], Standard Error of Mean 0.12
Statistical Analysis 5: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 14, analysis 1]; Test type: Superiority; p = 0.0032, ANCOVA; LS Mean Difference = -0.36, 95% CI 2-sided [-0.60 to -0.12], Standard Error of Mean 0.12
Statistical Analysis 6: Comparison: Placebo vs Pooled Tanezumab 5 mg; Change at Week 4: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf worst pain, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.0003, ANCOVA; LS Mean Difference = -0.57, 95% CI 2-sided [-0.88 to -0.27], Standard Error of Mean 0.16
Statistical Analysis 7: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 14, analysis 6]; Test type: Superiority; p < .0001, ANCOVA; LS Mean Difference = -0.77, 95% CI 2-sided [-1.08 to -0.46], Standard Error of Mean 0.16
Statistical Analysis 8: Comparison: Placebo vs Tramadol; [analysis description as in outcome 14, analysis 6]; Test type: Superiority; p = 0.0844, ANCOVA; LS Mean Difference = -0.25, 95% CI 2-sided [-0.54 to 0.03], Standard Error of Mean 0.15
Statistical Analysis 9: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 14, analysis 6]; Test type: Superiority; p = 0.0258, ANCOVA; LS Mean Difference = -0.32, 95% CI 2-sided [-0.60 to -0.04], Standard Error of Mean 0.14
Statistical Analysis 10: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 14, analysis 6]; Test type: Superiority; p = 0.0004, ANCOVA; LS Mean Difference = -0.52, 95% CI 2-sided [-0.80 to -0.23], Standard Error of Mean 0.15
Statistical Analysis 11: Comparison: Placebo vs Pooled Tanezumab 5 mg; Change at Week 8: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf worst pain, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.0079, ANCOVA; LS Mean Difference = -0.45, 95% CI 2-sided [-0.78 to -0.12], Standard Error of Mean 0.17
Statistical Analysis 12: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 14, analysis 11]; Test type: Superiority; p < .0001, ANCOVA; LS Mean Difference = -0.75, 95% CI 2-sided [-1.08 to -0.41], Standard Error of Mean 0.17
Statistical Analysis 13: Comparison: Placebo vs Tramadol; [analysis description as in outcome 14, analysis 11]; Test type: Superiority; p = 0.0977, ANCOVA; LS Mean Difference = -0.26, 95% CI 2-sided [-0.57 to 0.05], Standard Error of Mean 0.16
Statistical Analysis 14: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 14, analysis 11]; Test type: Superiority; p = 0.2150, ANCOVA; LS Mean Difference = -0.19, 95% CI 2-sided [-0.50 to 0.11], Standard Error of Mean 0.15
Statistical Analysis 15: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 14, analysis 11]; Test type: Superiority; p = 0.0016, ANCOVA; LS Mean Difference = -0.49, 95% CI 2-sided [-0.79 to -0.18], Standard Error of Mean 0.15
Statistical Analysis 16: Comparison: Placebo vs Pooled Tanezumab 5 mg; Change at Week 16: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf worst pain, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.0058, ANCOVA; LS Mean Difference = -0.52, 95% CI 2-sided [-0.88 to -0.15], Standard Error of Mean 0.19
Statistical Analysis 17: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 14, analysis 16]; Test type: Superiority; p = 0.0038, ANCOVA; LS Mean Difference = -0.54, 95% CI 2-sided [-0.91 to -0.18], Standard Error of Mean 0.19
Statistical Analysis 18: Comparison: Placebo vs Tramadol; [analysis description as in outcome 14, analysis 16]; Test type: Superiority; p = 0.1707, ANCOVA; LS Mean Difference = -0.24, 95% CI 2-sided [-0.58 to 0.10], Standard Error of Mean 0.17
Statistical Analysis 19: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 14, analysis 16]; Test type: Superiority; p = 0.1083, ANCOVA; LS Mean Difference = -0.28, 95% CI 2-sided [-0.62 to 0.06], Standard Error of Mean 0.17
Statistical Analysis 20: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 14, analysis 16]; Test type: Superiority; p = 0.0734, ANCOVA; LS Mean Difference = -0.31, 95% CI 2-sided [-0.64 to 0.03], Standard Error of Mean 0.17
Statistical Analysis 21: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Change at Week 24: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf worst pain, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.4603, ANCOVA; LS Mean Difference = -0.15, 95% CI 2-sided [-0.56 to 0.25], Standard Error of Mean 0.21
Statistical Analysis 22: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 14, analysis 21]; Test type: Superiority; p = 0.0799, ANCOVA; LS Mean Difference = -0.35, 95% CI 2-sided [-0.74 to 0.04], Standard Error of Mean 0.20
Statistical Analysis 23: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Change at Week 32: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf worst pain, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.2339, ANCOVA; LS Mean Difference = -0.25, 95% CI 2-sided [-0.66 to 0.16], Standard Error of Mean 0.21
Statistical Analysis 24: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 14, analysis 23]; Test type: Superiority; p = 0.1199, ANCOVA; LS Mean Difference = -0.32, 95% CI 2-sided [-0.73 to 0.08], Standard Error of Mean 0.21
Statistical Analysis 25: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Change at Week 40: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf worst pain, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.3840, ANCOVA; LS Mean Difference = -0.18, 95% CI 2-sided [-0.60 to 0.23], Standard Error of Mean 0.21
Statistical Analysis 26: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 14, analysis 25]; Test type: Superiority; p = 0.2000, ANCOVA; LS Mean Difference = -0.27, 95% CI 2-sided [-0.68 to 0.14], Standard Error of Mean 0.21
Statistical Analysis 27: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Change at Week 48: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf worst pain, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.2997, ANCOVA; LS Mean Difference = -0.22, 95% CI 2-sided [-0.65 to 0.20], Standard Error of Mean 0.22
Statistical Analysis 28: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 14, analysis 27]; Test type: Superiority; p = 0.1778, ANCOVA; LS Mean Difference = -0.29, 95% CI 2-sided [-0.71 to 0.13], Standard Error of Mean 0.21
Statistical Analysis 29: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Change at Week 56: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf worst pain, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.3438, ANCOVA; LS Mean Difference = -0.21, 95% CI 2-sided [-0.65 to 0.23], Standard Error of Mean 0.22
Statistical Analysis 30: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 14, analysis 29]; Test type: Superiority; p = 0.1876, ANCOVA; LS Mean Difference = -0.29, 95% CI 2-sided [-0.71 to 0.14], Standard Error of Mean 0.22

15. Secondary Outcome: Change From Baseline in Brief Pain Inventory-Short Form (BPI-sf) Score Worst Pain at Week 64: Observed Data
Description: BPI-sf is a self-administered questionnaire developed to assess the severity of pain and pain interference on daily functions during 24 hours prior to evaluation. Severity of pain was measured based on questions 1 to 4 of pain at its 'worst', 'least', 'average' and 'right now'. For the Worst Pain item of the BPI-sf scale (11 point NRS scale; range: 0 [no pain] to 10 [pain as bad as you can imagine]), participants were asked to rate their pain by marking an "X" in one of the boxes that best described their pain at its worst, during 24 hours prior to evaluation, higher scores indicated greater pain severity. Question 5 (7-items) assessed level of pain interference on daily activities.
Time Frame: Baseline, Week 64
Population: ITT population included all randomized participants who received at least one dose of SC study medication (either tanezumab or matching placebo). Here, 'n' = participants evaluable for this OM at specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Followed by Tanezumab 5 mg | Placebo Followed by Tanezumab 10 mg | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 202 | 204 | 407 | 407 | 605
units on a scale
  Baseline: number analyzed (Participants) | 202 | 204 | 405 | 407 | 605
  Baseline | 7.93 (1.18) | 7.91 (1.09) | 7.95 (1.11) | 7.92 (1.19) | 7.92 (1.18)
  Change at Week 64: number analyzed (Participants) | 63 | 57 | 140 | 147 | 200
  Change at Week 64 | -3.90 (2.69) | -4.28 (2.37) | -4.01 (2.68) | -3.61 (2.52) | -4.23 (2.39)

16. Secondary Outcome: Change From Baseline in Brief Pain Inventory-Short Form (BPI-sf) Scores Average Pain at Weeks 2, 4, 8, 16, 24, 32, 40, 48 and 56: Observed Data
Description: BPI-sf is a self-administered questionnaire developed to assess the severity of pain and pain interference on daily functions during 24 hours prior to evaluation. Severity of pain was measured based on questions 1 to 4 of pain at its 'worst', 'least', 'average' and 'right now'. For the Average Pain item of the BPI-sf scale (11 point NRS scale; range: 0 [no pain] to 10 [pain as bad as you can imagine]), participants were asked to rate their pain by marking an "X" in one of the boxes that best described their pain during 24 hours prior to evaluation, higher scores indicated greater pain severity. Question 5 (7-items) assessed level of pain interference on daily activities.Pre-specified intent of study for efficacy data up to W16 was to analyze participants who received placebo from Day1 and then received tanezumab 5/10 mg at W16,together,in placebo arm.Data has been reported per four arms.
Time Frame: Baseline, Weeks 2, 4, 8, 16, 24, 32, 40, 48 and 56
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 406 | 407 | 407 | 605
units on a scale
  Change at Week 2 | -0.93 (0.10) | -1.40 (0.10) | -1.47 (0.10) | -1.20 (0.08)
  Change at Week 4 | -1.52 (0.12) | -2.04 (0.12) | -2.22 (0.12) | -1.76 (0.10)
  Change at Week 8 | -1.90 (0.12) | -2.36 (0.12) | -2.60 (0.12) | -2.20 (0.10)
  Change at Week 16 | -2.47 (0.14) | -2.84 (0.14) | -2.93 (0.14) | -2.64 (0.12)
  Change at Week 24: number analyzed (Participants) | 0 | 407 | 407 | 605
  Change at Week 24 |  | -2.58 (0.16) | -2.72 (0.16) | -2.45 (0.14)
  Change at Week 32: number analyzed (Participants) | 0 | 407 | 407 | 605
  Change at Week 32 |  | -2.61 (0.16) | -2.67 (0.16) | -2.43 (0.14)
  Change at Week 40: number analyzed (Participants) | 0 | 407 | 407 | 605
  Change at Week 40 |  | -2.46 (0.17) | -2.53 (0.17) | -2.32 (0.14)
  Change at Week 48: number analyzed (Participants) | 0 | 407 | 407 | 605
  Change at Week 48 |  | -2.40 (0.17) | -2.44 (0.17) | -2.29 (0.14)
  Change at Week 56: number analyzed (Participants) | 0 | 407 | 407 | 605
  Change at Week 56 |  | -2.32 (0.17) | -2.51 (0.17) | -2.29 (0.14)
Statistical Analysis 1: Comparison: Placebo vs Pooled Tanezumab 5 mg; Change at Week 2: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf average pain, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.0002, ANCOVA; LS Mean Difference = -0.47, 95% CI 2-sided [-0.72 to -0.22], Standard Error of Mean 0.13
Statistical Analysis 2: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 16, analysis 1]; Test type: Superiority; p < .0001, ANCOVA; LS Mean Difference = -0.54, 95% CI 2-sided [-0.79 to -0.29], Standard Error of Mean 0.13
Statistical Analysis 3: Comparison: Placebo vs Tramadol; [analysis description as in outcome 16, analysis 1]; Test type: Superiority; p = 0.0193, ANCOVA; LS Mean Difference = -0.27, 95% CI 2-sided [-0.50 to -0.04], Standard Error of Mean 0.12
Statistical Analysis 4: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 16, analysis 1]; Test type: Superiority; p = 0.0845, ANCOVA; LS Mean Difference = -0.20, 95% CI 2-sided [-0.42 to 0.03], Standard Error of Mean 0.12
Statistical Analysis 5: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 16, analysis 1]; Test type: Superiority; p = 0.0212, ANCOVA; LS Mean Difference = -0.27, 95% CI 2-sided [-0.49 to -0.04], Standard Error of Mean 0.12
Statistical Analysis 6: Comparison: Placebo vs Pooled Tanezumab 5 mg; Change at Week 4: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf average pain, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.0003, ANCOVA; LS Mean Difference = -0.53, 95% CI 2-sided [-0.81 to -0.24], Standard Error of Mean 0.15
Statistical Analysis 7: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 16, analysis 6]; Test type: Superiority; p < .0001, ANCOVA; LS Mean Difference = -0.70, 95% CI 2-sided [-0.99 to -0.41], Standard Error of Mean 0.15
Statistical Analysis 8: Comparison: Placebo vs Tramadol; [analysis description as in outcome 14, analysis 6]; Test type: Superiority; p = 0.0790, ANCOVA; LS Mean Difference = -0.24, 95% CI 2-sided [-0.50 to 0.03], Standard Error of Mean 0.14
Statistical Analysis 9: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 16, analysis 6]; Test type: Superiority; p = 0.0336, ANCOVA; LS Mean Difference = -0.29, 95% CI 2-sided [-0.55 to -0.02], Standard Error of Mean 0.14
Statistical Analysis 10: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 16, analysis 6]; Test type: Superiority; p = 0.0008, ANCOVA; LS Mean Difference = -0.46, 95% CI 2-sided [-0.73 to -0.19], Standard Error of Mean 0.14
Statistical Analysis 11: Comparison: Placebo vs Pooled Tanezumab 5 mg; Change at Week 8: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf average pain, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.0034, ANCOVA; LS Mean Difference = -0.46, 95% CI 2-sided [-0.77 to -0.15], Standard Error of Mean 0.16
Statistical Analysis 12: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 16, analysis 11]; Test type: Superiority; p < .0001, ANCOVA; LS Mean Difference = -0.70, 95% CI 2-sided [-1.01 to -0.39], Standard Error of Mean 0.16
Statistical Analysis 13: Comparison: Placebo vs Tramadol; [analysis description as in outcome 16, analysis 11]; Test type: Superiority; p = 0.0361, ANCOVA; LS Mean Difference = -0.31, 95% CI 2-sided [-0.59 to -0.02], Standard Error of Mean 0.15
Statistical Analysis 14: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 16, analysis 11]; Test type: Superiority; p = 0.2786, ANCOVA; LS Mean Difference = -0.16, 95% CI 2-sided [-0.44 to 0.13], Standard Error of Mean 0.15
Statistical Analysis 15: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 16, analysis 11]; Test type: Superiority; p = 0.0058, ANCOVA; LS Mean Difference = -0.40, 95% CI 2-sided [-0.68 to -0.11], Standard Error of Mean 0.14
Statistical Analysis 16: Comparison: Placebo vs Pooled Tanezumab 5 mg; Change at Week 16: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf average pain, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.0365, ANCOVA; LS Mean Difference = -0.37, 95% CI 2-sided [-0.71 to -0.02], Standard Error of Mean 0.18
Statistical Analysis 17: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 16, analysis 16]; Test type: Superiority; p = 0.0092, ANCOVA; LS Mean Difference = -0.46, 95% CI 2-sided [-0.80 to -0.11], Standard Error of Mean 0.18
Statistical Analysis 18: Comparison: Placebo vs Tramadol; [analysis description as in outcome 16, analysis 16]; Test type: Superiority; p = 0.2923, ANCOVA; LS Mean Difference = -0.17, 95% CI 2-sided [-0.49 to 0.15], Standard Error of Mean 0.16
Statistical Analysis 19: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 16, analysis 16]; Test type: Superiority; p = 0.2231, ANCOVA; LS Mean Difference = -0.20, 95% CI 2-sided [-0.51 to 0.12], Standard Error of Mean 0.16
Statistical Analysis 20: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 16, analysis 16]; Test type: Superiority; p = 0.0724, ANCOVA; LS Mean Difference = -0.29, 95% CI 2-sided [-0.60 to 0.03], Standard Error of Mean 0.16
Statistical Analysis 21: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Change at Week 24: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf average pain, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.4776, ANCOVA; LS Mean Difference = -0.13, 95% CI 2-sided [-0.50 to 0.23], Standard Error of Mean 0.19
Statistical Analysis 22: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 16, analysis 21]; Test type: Superiority; p = 0.1482, ANCOVA; LS Mean Difference = -0.27, 95% CI 2-sided [-0.64 to 0.10], Standard Error of Mean 0.19
Statistical Analysis 23: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Change at Week 32: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf average pain, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.3249, ANCOVA; LS Mean Difference = -0.19, 95% CI 2-sided [-0.56 to 0.18], Standard Error of Mean 0.19
Statistical Analysis 24: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 16, analysis 23]; Test type: Superiority; p = 0.1997, ANCOVA; LS Mean Difference = -0.24, 95% CI 2-sided [-0.62 to 0.13], Standard Error of Mean 0.19
Statistical Analysis 25: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Change at Week 40: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf average pain, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.4823, ANCOVA; LS Mean Difference = -0.14, 95% CI 2-sided [-0.53 to 0.25], Standard Error of Mean 0.20
Statistical Analysis 26: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 16, analysis 25]; Test type: Superiority; p = 0.2754, ANCOVA; LS Mean Difference = -0.21, 95% CI 2-sided [-0.60 to 0.17], Standard Error of Mean 0.20
Statistical Analysis 27: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Change at Week 48: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf average pain, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.5861, ANCOVA; LS Mean Difference = -0.11, 95% CI 2-sided [-0.50 to 0.29], Standard Error of Mean 0.20
Statistical Analysis 28: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 16, analysis 27]; Test type: Superiority; p = 0.4346, ANCOVA; LS Mean Difference = -0.16, 95% CI 2-sided [-0.54 to 0.23], Standard Error of Mean 0.20
Statistical Analysis 29: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Change at Week 56: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf average pain, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.8752, ANCOVA; LS Mean Difference = -0.03, 95% CI 2-sided [-0.42 to 0.36], Standard Error of Mean 0.20
Statistical Analysis 30: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 16, analysis 29]; Test type: Superiority; p = 0.2663, ANCOVA; LS Mean Difference = -0.22, 95% CI 2-sided [-0.60 to 0.17], Standard Error of Mean 0.20

17. Secondary Outcome: Change From Baseline in Brief Pain Inventory-Short Form (BPI-sf) Score Average Pain at Week 64: Observed Data
Description: BPI-sf is a self-administered questionnaire developed to assess the severity of pain and pain interference on daily functions during 24 hours prior to evaluation. Severity of pain was measured based on questions 1 to 4 of pain at its 'worst', 'least', 'average' and 'right now'. For the Average Pain item of the BPI-sf scale (11 point NRS scale; range: 0 [no pain] to 10 [pain as bad as you can imagine]), participants were asked to rate their pain by marking an "X" in one of the boxes that best described their pain during 24 hours prior to evaluation, higher scores indicated greater pain severity. Question 5 (7-items) assessed level of pain interference on daily activities.
Time Frame: Baseline, Week 64
Population: ITT population included all randomized participants who received at least one dose of SC study medication (either tanezumab or matching placebo). Here, 'number analyzed' = participants evaluable for this OM at specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Followed by Tanezumab 5 mg | Placebo Followed by Tanezumab 10 mg | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 202 | 204 | 407 | 407 | 605
units on a scale
  Baseline: number analyzed (Participants) | 202 | 204 | 405 | 407 | 605
  Baseline | 6.87 (1.20) | 7.02 (1.15) | 7.00 (1.18) | 6.88 (1.21) | 6.97 (1.21)
  Change at Week 64: number analyzed (Participants) | 63 | 57 | 140 | 147 | 200
  Change at Week 64 | -3.75 (2.37) | -4.09 (1.82) | -3.84 (2.23) | -3.39 (2.38) | -4.04 (2.06)

18. Secondary Outcome: Change From Baseline in Brief Pain Inventory-Short Form (BPI-sf) Score Pain Interference Index at Weeks 2, 4, 8, 16, 24, 32, 40, 48 and 56: Observed Data
Description: BPI-sf is a self-administered questionnaire developed to assess the severity of pain and pain interference on daily functions during 24 hours prior to evaluation. Severity of pain was measured based on questions 1 to 4. Question 5 (7-items) assessed level of pain interference on daily activities. Pain interference index was calculated as the mean of the seven BPI-sf pain interference items (question 5a to g), being pain interference with general activity; mood; walking ability; normal work (outside home and housework); relations with other people; sleep and enjoyment of life. Responses were given on an 11-point NRS with score ranging from 0 (does not interfere) to 10 (completely interferes), lower scores indicated less pain or pain interference.Pre-specified intent of study for efficacy data up to W16 was to analyze participants who received placebo from Day1 and then received tanezumab 5/10 mg at W16,together,in placebo arm.Data has been reported per four arms.
Time Frame: Baseline, Weeks 2, 4, 8, 16, 24, 32, 40, 48 and 56
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 406 | 407 | 407 | 605
units on a scale
  Change at Week 2 | -1.40 (0.11) | -1.88 (0.11) | -1.97 (0.11) | -1.57 (0.10)
  Change at Week 4 | -1.90 (0.13) | -2.50 (0.13) | -2.68 (0.13) | -2.14 (0.11)
  Change at Week 8 | -2.26 (0.13) | -2.70 (0.13) | -2.83 (0.13) | -2.44 (0.11)
  Change at Week 16 | -2.65 (0.14) | -3.06 (0.14) | -3.23 (0.14) | -2.80 (0.12)
  Change at Week 24: number analyzed (Participants) | 0 | 407 | 407 | 605
  Change at Week 24 |  | -2.67 (0.17) | -2.75 (0.16) | -2.44 (0.14)
  Change at Week 32: number analyzed (Participants) | 0 | 407 | 407 | 605
  Change at Week 32 |  | -2.64 (0.16) | -2.64 (0.16) | -2.37 (0.14)
  Change at Week 40: number analyzed (Participants) | 0 | 407 | 407 | 605
  Change at Week 40 |  | -2.44 (0.17) | -2.48 (0.17) | -2.24 (0.14)
  Change at Week 48: number analyzed (Participants) | 0 | 407 | 407 | 605
  Change at Week 48 |  | -2.37 (0.17) | -2.37 (0.17) | -2.18 (0.14)
  Change at Week 56: number analyzed (Participants) | 0 | 407 | 407 | 605
  Change at Week 56 |  | -2.32 (0.17) | -2.44 (0.17) | -2.21 (0.15)
Statistical Analysis 1: Comparison: Placebo vs Pooled Tanezumab 5 mg; Change at Week 2: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf pain interference index, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.0013, ANCOVA; LS Mean Difference = -0.48, 95% CI 2-sided [-0.77 to -0.19], Standard Error of Mean 0.15
Statistical Analysis 2: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 18, analysis 1]; Test type: Superiority; p = 0.0001, ANCOVA; LS Mean Difference = -0.57, 95% CI 2-sided [-0.87 to -0.28], Standard Error of Mean 0.15
Statistical Analysis 3: Comparison: Placebo vs Tramadol; [analysis description as in outcome 18, analysis 1]; Test type: Superiority; p = 0.2272, ANCOVA; LS Mean Difference = -0.17, 95% CI 2-sided [-0.43 to -0.10], Standard Error of Mean 0.14
Statistical Analysis 4: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 18, analysis 1]; Test type: Superiority; p = 0.0209, ANCOVA; LS Mean Difference = -0.31, 95% CI 2-sided [-0.58 to -0.05], Standard Error of Mean 0.14
Statistical Analysis 5: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 18, analysis 1]; Test type: Superiority; p = 0.0029, ANCOVA; LS Mean Difference = -0.41, 95% CI 2-sided [-0.67 to -0.14], Standard Error of Mean 0.14
Statistical Analysis 6: Comparison: Placebo vs Pooled Tanezumab 5 mg; Change at Week 4: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf pain interference index, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.0002, ANCOVA; LS Mean Difference = -0.60, 95% CI 2-sided [-0.92 to -0.28], Standard Error of Mean 0.16
Statistical Analysis 7: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 18, analysis 6]; Test type: Superiority; p < .0001, ANCOVA; LS Mean Difference = -0.78, 95% CI 2-sided [-1.10 to -0.46], Standard Error of Mean 0.16
Statistical Analysis 8: Comparison: Placebo vs Tramadol; [analysis description as in outcome 18, analysis 6]; Test type: Superiority; p = 0.1198, ANCOVA; LS Mean Difference = -0.23, 95% CI 2-sided [-0.53 to 0.06], Standard Error of Mean 0.15
Statistical Analysis 9: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 18, analysis 6]; Test type: Superiority; p = 0.0160, ANCOVA; LS Mean Difference = -0.37, 95% CI 2-sided [-0.66 to -0.07], Standard Error of Mean 0.15
Statistical Analysis 10: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 18, analysis 6]; Test type: Superiority; p = 0.0003, ANCOVA; LS Mean Difference = -0.55, 95% CI 2-sided [-0.85 to -0.25], Standard Error of Mean 0.15
Statistical Analysis 11: Comparison: Placebo vs Pooled Tanezumab 5 mg; Change at Week 8: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf pain interference index, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.0091, ANCOVA; LS Mean Difference = -0.44, 95% CI 2-sided [-0.77 to -0.11], Standard Error of Mean 0.17
Statistical Analysis 12: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 18, analysis 11]; Test type: Superiority; p = 0.0007, ANCOVA; LS Mean Difference = -0.57, 95% CI 2-sided [-0.90 to -0.24], Standard Error of Mean 0.17
Statistical Analysis 13: Comparison: Placebo vs Tramadol; [analysis description as in outcome 18, analysis 11]; Test type: Superiority; p = 0.2264, ANCOVA; LS Mean Difference = -0.18, 95% CI 2-sided [-0.48 to 0.11], Standard Error of Mean 0.15
Statistical Analysis 14: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 18, analysis 11]; Test type: Superiority; p = 0.0961, ANCOVA; LS Mean Difference = -0.26, 95% CI 2-sided [-0.56 to 0.05], Standard Error of Mean 0.15
Statistical Analysis 15: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 18, analysis 11]; Test type: Superiority; p = 0.0121, ANCOVA; LS Mean Difference = -0.39, 95% CI 2-sided [-0.69 to -0.08], Standard Error of Mean 0.15
Statistical Analysis 16: Comparison: Placebo vs Pooled Tanezumab 5 mg; Change at Week 16: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf pain interference index, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.0270, ANCOVA; LS Mean Difference = -0.41, 95% CI 2-sided [-0.77 to -0.05], Standard Error of Mean 0.18
Statistical Analysis 17: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 18, analysis 16]; Test type: Superiority; p = 0.0019, ANCOVA; LS Mean Difference = -0.58, 95% CI 2-sided [-0.94 to -0.21], Standard Error of Mean 0.18
Statistical Analysis 18: Comparison: Placebo vs Tramadol; [analysis description as in outcome 18, analysis 16]; Test type: Superiority; p = 0.3906, ANCOVA; LS Mean Difference = -0.15, 95% CI 2-sided [-0.48 to 0.19], Standard Error of Mean 0.17
Statistical Analysis 19: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 18, analysis 16]; Test type: Superiority; p = 0.1209, ANCOVA; LS Mean Difference = -0.26, 95% CI 2-sided [-0.59 to 0.07], Standard Error of Mean 0.17
Statistical Analysis 20: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 18, analysis 16]; Test type: Superiority; p = 0.0107, ANCOVA; LS Mean Difference = -0.43, 95% CI 2-sided [-0.76 to -0.10], Standard Error of Mean 0.17
Statistical Analysis 21: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Change at Week 24: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf pain interference index, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.2396, ANCOVA; LS Mean Difference = -0.23, 95% CI 2-sided [-0.61 to 0.15], Standard Error of Mean 0.19
Statistical Analysis 22: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 18, analysis 21]; Test type: Superiority; p = 0.1088, ANCOVA; LS Mean Difference = -0.31, 95% CI 2-sided [-0.69 to 0.07], Standard Error of Mean 0.19
Statistical Analysis 23: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Change at Week 32: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf pain interference index, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.1673, ANCOVA; LS Mean Difference = -0.27, 95% CI 2-sided [-0.65 to 0.11], Standard Error of Mean 0.20
Statistical Analysis 24: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 18, analysis 23]; Test type: Superiority; p = 0.1751, ANCOVA; LS Mean Difference = -0.27, 95% CI 2-sided [-0.66 to 0.12], Standard Error of Mean 0.20
Statistical Analysis 25: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Change at Week 40: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf pain interference index, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.3164, ANCOVA; LS Mean Difference = -0.20, 95% CI 2-sided [-0.59 to 0.19], Standard Error of Mean 0.20
Statistical Analysis 26: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 18, analysis 25]; Test type: Superiority; p = 0.2253, ANCOVA; LS Mean Difference = -0.24, 95% CI 2-sided [-0.62 to 0.15], Standard Error of Mean 0.20
Statistical Analysis 27: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Change at Week 48: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf pain interference index, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.3408, ANCOVA; LS Mean Difference = -0.19, 95% CI 2-sided [-0.58 to 0.20], Standard Error of Mean 0.20
Statistical Analysis 28: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 18, analysis 27]; Test type: Superiority; p = 0.3391, ANCOVA; LS Mean Difference = -0.19, 95% CI 2-sided [-0.58 to 0.20], Standard Error of Mean 0.20
Statistical Analysis 29: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Change at Week 56: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf pain interference index, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.5818, ANCOVA; LS Mean Difference = -0.11, 95% CI 2-sided [-0.50 to 0.28], Standard Error of Mean 0.20
Statistical Analysis 30: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 18, analysis 29]; Test type: Superiority; p = 0.2562, ANCOVA; LS Mean Difference = -0.23, 95% CI 2-sided [-0.62 to 0.16], Standard Error of Mean 0.20

19. Secondary Outcome: Change From Baseline in Brief Pain Inventory-Short Form (BPI-sf) Score Pain Interference Index at Week 64: Observed Data
Description: BPI-sf is a self-administered questionnaire developed to assess the severity of pain and pain interference on daily functions during 24 hours prior to evaluation. Severity of pain was measured based on questions 1 to 4. Question 5 (7-items) assessed level of pain interference on daily activities. Pain interference index was calculated as the mean of the seven BPI-sf pain interference items (question 5a to g), being pain interference with general activity; mood; walking ability; normal work (outside home and housework); relations with other people; sleep and enjoyment of life. Responses were given on an 11-point NRS with score ranging from 0 (does not interfere) to 10 (completely interferes), lower scores indicated less pain or pain interference.
Time Frame: Baseline, Week 64
Population: ITT population included all randomized participants who received at least one dose of SC study medication (either tanezumab or matching placebo). Here, 'n' = participants evaluable for this OM at specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Followed by Tanezumab 5 mg | Placebo Followed by Tanezumab 10 mg | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 202 | 204 | 407 | 407 | 605
units on a scale
  Baseline: number analyzed (Participants) | 202 | 204 | 405 | 407 | 605
  Baseline | 5.85 (1.90) | 6.20 (1.88) | 6.28 (1.81) | 6.16 (1.93) | 6.21 (1.88)
  Change at Week 64: number analyzed (Participants) | 63 | 57 | 140 | 147 | 200
  Change at Week 64 | -3.87 (2.63) | -4.21 (1.98) | -4.00 (2.44) | -3.60 (2.30) | -3.98 (2.10)

20. Secondary Outcome: Change From Baseline in Brief Pain Inventory-Short Form (BPI-sf) Score Pain Interference With General Activity at Weeks 2, 4, 8, 16, 24, 32, 40, 48 and 56: Observed Data
Description: as for outcome 18
Time Frame: Baseline, Weeks 2, 4, 8, 16, 24, 32, 40, 48 and 56
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 406 | 407 | 407 | 605
units on a scale
  Change at Week 2 | -1.46 (0.12) | -1.84 (0.12) | -1.91 (0.12) | -1.53 (0.10)
  Change at Week 4 | -1.92 (0.13) | -2.45 (0.13) | -2.71 (0.13) | -2.14 (0.12)
  Change at Week 8 | -2.37 (0.14) | -2.68 (0.14) | -2.86 (0.14) | -2.54 (0.12)
  Change at Week 16 | -2.70 (0.15) | -3.20 (0.15) | -3.35 (0.15) | -2.89 (0.13)
  Change at Week 24: number analyzed (Participants) | 0 | 407 | 407 | 605
  Change at Week 24 |  | -2.78 (0.17) | -2.87 (0.17) | -2.60 (0.14)
  Change at Week 32: number analyzed (Participants) | 0 | 407 | 407 | 605
  Change at Week 32 |  | -2.74 (0.18) | -2.76 (0.17) | -2.52 (0.15)
  Change at Week 40: number analyzed (Participants) | 0 | 407 | 407 | 605
  Change at Week 40 |  | -2.54 (0.18) | -2.58 (0.18) | -2.40 (0.15)
  Change at Week 48: number analyzed (Participants) | 0 | 407 | 407 | 605
  Change at Week 48 |  | -2.47 (0.18) | -2.47 (0.18) | -2.33 (0.15)
  Change at Week 56: number analyzed (Participants) | 0 | 407 | 407 | 605
  Change at Week 56 |  | -2.44 (0.18) | -2.53 (0.18) | -2.39 (0.15)
Statistical Analysis 1: Comparison: Placebo vs Pooled Tanezumab 5 mg; Change at Week 2: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf pain interference with general activity, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.0137, ANCOVA; LS Mean Difference = -0.39, 95% CI 2-sided [-0.69 to -0.08], Standard Error of Mean 0.16
Statistical Analysis 2: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.0044, ANCOVA; LS Mean Difference = -0.45, 95% CI 2-sided [-0.76 to -0.14], Standard Error of Mean 0.16
Statistical Analysis 3: Comparison: Placebo vs Tramadol; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.6194, ANCOVA; LS Mean Difference = -0.07, 95% CI 2-sided [-0.35 to 0.21], Standard Error of Mean 0.14
Statistical Analysis 4: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.0271, ANCOVA; LS Mean Difference = -0.31, 95% CI 2-sided [-0.59 to -0.04], Standard Error of Mean 0.14
Statistical Analysis 5: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 20, analysis 1]; Test type: Superiority; p = 0.0085, ANCOVA; LS Mean Difference = -0.38, 95% CI 2-sided [-0.66 to -0.10], Standard Error of Mean 0.14
Statistical Analysis 6: Comparison: Placebo vs Pooled Tanezumab 5 mg; Change at Week 4: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf pain interference with general activity, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.0027, ANCOVA; LS Mean Difference = -0.53, 95% CI 2-sided [-0.87 to -0.18], Standard Error of Mean 0.18
Statistical Analysis 7: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 20, analysis 6]; Test type: Superiority; p < .0001, ANCOVA; LS Mean Difference = -0.78, 95% CI 2-sided [-1.13 to -0.44], Standard Error of Mean 0.18
Statistical Analysis 8: Comparison: Placebo vs Tramadol; [analysis description as in outcome 20, analysis 6]; Test type: Superiority; p = 0.1859, ANCOVA; LS Mean Difference = -0.22, 95% CI 2-sided [-0.54 to 0.10], Standard Error of Mean 0.16
Statistical Analysis 9: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 20, analysis 6]; Test type: Superiority; p = 0.0573, ANCOVA; LS Mean Difference = -0.31, 95% CI 2-sided [-0.63 to 0.01], Standard Error of Mean 0.16
Statistical Analysis 10: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 20, analysis 6]; Test type: Superiority; p = 0.0005, ANCOVA; LS Mean Difference = -0.56, 95% CI 2-sided [-0.88 to -0.25], Standard Error of Mean 0.16
Statistical Analysis 11: Comparison: Placebo vs Pooled Tanezumab 5 mg; Change at Week 8: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf pain interference with general activity, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.0841, ANCOVA; LS Mean Difference = -0.31, 95% CI 2-sided [-0.66 to 0.04], Standard Error of Mean 0.18
Statistical Analysis 12: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 20, analysis 11]; Test type: Superiority; p = 0.0074, ANCOVA; LS Mean Difference = -0.49, 95% CI 2-sided [-0.85 to -0.13], Standard Error of Mean 0.18
Statistical Analysis 13: Comparison: Placebo vs Tramadol; [analysis description as in outcome 20, analysis 11]; Test type: Superiority; p = 0.3160, ANCOVA; LS Mean Difference = -0.17, 95% CI 2-sided [-0.49 to 0.16], Standard Error of Mean 0.16
Statistical Analysis 14: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 20, analysis 11]; Test type: Superiority; p = 0.3763, ANCOVA; LS Mean Difference = -0.15, 95% CI 2-sided [-0.47 to 0.18], Standard Error of Mean 0.17
Statistical Analysis 15: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 20, analysis 11]; Test type: Superiority; p = 0.0505, ANCOVA; LS Mean Difference = -0.32, 95% CI 2-sided [-0.65 to 0.00], Standard Error of Mean 0.17
Statistical Analysis 16: Comparison: Placebo vs Pooled Tanezumab 5 mg; Change at Week 16: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf pain interference with general activity, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.0118, ANCOVA; LS Mean Difference = -0.49, 95% CI 2-sided [-0.88 to -0.11], Standard Error of Mean 0.20
Statistical Analysis 17: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 20, analysis 16]; Test type: Superiority; p = 0.0012, ANCOVA; LS Mean Difference = -0.64, 95% CI 2-sided [-1.03 to -0.25], Standard Error of Mean 0.20
Statistical Analysis 18: Comparison: Placebo vs Tramadol; [analysis description as in outcome 20, analysis 16]; Test type: Superiority; p = 0.2966, ANCOVA; LS Mean Difference = -0.19, 95% CI 2-sided [-0.54 to 0.17], Standard Error of Mean 0.18
Statistical Analysis 19: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 20, analysis 16]; Test type: Superiority; p = 0.0956, ANCOVA; LS Mean Difference = -0.30, 95% CI 2-sided [-0.66 to 0.05], Standard Error of Mean 0.18
Statistical Analysis 20: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 20, analysis 16]; Test type: Superiority; p = 0.0117, ANCOVA; LS Mean Difference = -0.45, 95% CI 2-sided [-0.81 to -0.10], Standard Error of Mean 0.18
Statistical Analysis 21: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Change at Week 24: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf pain interference with general activity, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.3732, ANCOVA; LS Mean Difference = -0.18, 95% CI 2-sided [-0.57 to 0.21], Standard Error of Mean 0.20
Statistical Analysis 22: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 20, analysis 21]; Test type: Superiority; p = 0.1922, ANCOVA; LS Mean Difference = -0.26, 95% CI 2-sided [-0.66 to 0.13], Standard Error of Mean 0.20
Statistical Analysis 23: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Change at Week 32: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf pain interference with general activity, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.2986, ANCOVA; LS Mean Difference = -0.22, 95% CI 2-sided [-0.63 to 0.19], Standard Error of Mean 0.21
Statistical Analysis 24: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 20, analysis 23]; Test type: Superiority; p = 0.2584, ANCOVA; LS Mean Difference = -0.24, 95% CI 2-sided [-0.65 to 0.17], Standard Error of Mean 0.21
Statistical Analysis 25: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Change at Week 40: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf pain interference with general activity, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.5195, ANCOVA; LS Mean Difference = -0.14, 95% CI 2-sided [-0.57 to 0.29], Standard Error of Mean 0.22
Statistical Analysis 26: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 20, analysis 25]; Test type: Superiority; p = 0.3752, ANCOVA; LS Mean Difference = -0.19, 95% CI 2-sided [-0.60 to 0.22], Standard Error of Mean 0.21
Statistical Analysis 27: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Change at Week 48: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf pain interference with general activity, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.5157, ANCOVA; LS Mean Difference = -0.14, 95% CI 2-sided [-0.56 to 0.28], Standard Error of Mean 0.22
Statistical Analysis 28: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 20, analysis 27]; Test type: Superiority; p = 0.5065, ANCOVA; LS Mean Difference = -0.14, 95% CI 2-sided [-0.56 to 0.28], Standard Error of Mean 0.21
Statistical Analysis 29: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Change at Week 56: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf pain interference with general activity, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.8373, ANCOVA; LS Mean Difference = -0.04, 95% CI 2-sided [-0.47 to 0.38], Standard Error of Mean 0.21
Statistical Analysis 30: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 20, analysis 29]; Test type: Superiority; p = 0.5146, ANCOVA; LS Mean Difference = -0.14, 95% CI 2-sided [-0.56 to 0.28], Standard Error of Mean 0.22

21. Secondary Outcome: Change From Baseline in Brief Pain Inventory-Short Form (BPI-sf) Score Pain Interference With General Activity at Week 64: Observed Data
Description: as for outcome 19
Time Frame: Baseline, Week 64
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Followed by Tanezumab 5 mg | Placebo Followed by Tanezumab 10 mg | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 202 | 204 | 407 | 407 | 605
units on a scale
  Baseline: number analyzed (Participants) | 202 | 204 | 405 | 407 | 605
  Baseline | 6.40 (1.81) | 6.69 (1.75) | 6.69 (1.70) | 6.66 (1.82) | 6.67 (1.75)
  Change at Week 64: number analyzed (Participants) | 63 | 57 | 140 | 147 | 200
  Change at Week 64 | -3.87 (2.79) | -4.46 (2.19) | -4.03 (2.74) | -3.72 (2.57) | -4.16 (2.33)

22. Secondary Outcome: Change From Baseline in Brief Pain Inventory-Short Form (BPI-sf) Score Pain Interference With Walking Ability at Weeks 2, 4, 8, 16, 24, 32, 40, 48 and 56: Observed Data
Description: as for outcome 18
Time Frame: Baseline, Weeks 2, 4, 8, 16, 24, 32, 40, 48 and 56
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 406 | 407 | 407 | 605
units on a scale
  Change at Week 2 | -1.28 (0.12) | -1.72 (0.12) | -1.89 (0.12) | -1.54 (0.10)
  Change at Week 4 | -1.81 (0.13) | -2.38 (0.13) | -2.55 (0.13) | -2.03 (0.12)
  Change at Week 8 | -2.17 (0.14) | -2.60 (0.13) | -2.73 (0.13) | -2.30 (0.11)
  Change at Week 16 | -2.55 (0.15) | -2.90 (0.15) | -3.15 (0.15) | -2.68 (0.13)
  Change at Week 24: number analyzed (Participants) | 0 | 407 | 407 | 605
  Change at Week 24 |  | -2.54 (0.17) | -2.73 (0.17) | -2.30 (0.14)
  Change at Week 32: number analyzed (Participants) | 0 | 407 | 407 | 605
  Change at Week 32 |  | -2.50 (0.17) | -2.59 (0.17) | -2.24 (0.14)
  Change at Week 40: number analyzed (Participants) | 0 | 407 | 407 | 605
  Change at Week 40 |  | -2.31 (0.17) | -2.46 (0.17) | -2.09 (0.15)
  Change at Week 48: number analyzed (Participants) | 0 | 407 | 407 | 605
  Change at Week 48 |  | -2.24 (0.17) | -2.34 (0.17) | -2.04 (0.14)
  Change at Week 56: number analyzed (Participants) | 0 | 407 | 407 | 605
  Change at Week 56 |  | -2.24 (0.17) | -2.45 (0.17) | -2.07 (0.14)
Statistical Analysis 1: Comparison: Placebo vs Pooled Tanezumab 5 mg; Change at Week 2: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf pain interference with walking ability, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.0059, ANCOVA; LS Mean Difference = -0.45, 95% CI 2-sided [-0.76 to -0.13], Standard Error of Mean 0.16
Statistical Analysis 2: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 22, analysis 1]; Test type: Superiority; p = 0.0002, ANCOVA; LS Mean Difference = -0.61, 95% CI 2-sided [-0.93 to -0.29], Standard Error of Mean 0.16
Statistical Analysis 3: Comparison: Placebo vs Tramadol; [analysis description as in outcome 22, analysis 1]; Test type: Superiority; p = 0.0756, ANCOVA; LS Mean Difference = -0.26, 95% CI 2-sided [-0.56 to 0.03], Standard Error of Mean 0.15
Statistical Analysis 4: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 22, analysis 1]; Test type: Superiority; p = 0.2197, ANCOVA; LS Mean Difference = -0.18, 95% CI 2-sided [-0.47 to 0.11], Standard Error of Mean 0.15
Statistical Analysis 5: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 22, analysis 1]; Test type: Superiority; p = 0.0208, ANCOVA; LS Mean Difference = -0.34, 95% CI 2-sided [-0.63 to -0.05], Standard Error of Mean 0.15
Statistical Analysis 6: Comparison: Placebo vs Pooled Tanezumab 5 mg; Change at Week 4: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf pain interference with walking ability, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.0013, ANCOVA; LS Mean Difference = -0.56, 95% CI 2-sided [-0.91 to -0.22], Standard Error of Mean 0.17
Statistical Analysis 7: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 22, analysis 6]; Test type: Superiority; p < .0001, ANCOVA; LS Mean Difference = -0.74, 95% CI 2-sided [-1.08 to -0.39], Standard Error of Mean 0.18
Statistical Analysis 8: Comparison: Placebo vs Tramadol; [analysis description as in outcome 22, analysis 6]; Test type: Superiority; p = 0.1873, ANCOVA; LS Mean Difference = -0.21, 95% CI 2-sided [-0.53 to 0.10], Standard Error of Mean 0.16
Statistical Analysis 9: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 22, analysis 6]; Test type: Superiority; p = 0.0305, ANCOVA; LS Mean Difference = -0.35, 95% CI 2-sided [-0.66 to -0.03], Standard Error of Mean 0.16
Statistical Analysis 10: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 22, analysis 6]; Test type: Superiority; p = 0.0013, ANCOVA; LS Mean Difference = -0.52, 95% CI 2-sided [-0.84 to -0.20], Standard Error of Mean 0.16
Statistical Analysis 11: Comparison: Placebo vs Pooled Tanezumab 5 mg; Change at Week 8: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf pain interference with walking ability, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.0158, ANCOVA; LS Mean Difference = -0.43, 95% CI 2-sided [-0.78 to -0.08], Standard Error of Mean 0.18
Statistical Analysis 12: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 22, analysis 11]; Test type: Superiority; p = 0.0015, ANCOVA; LS Mean Difference = -0.56, 95% CI 2-sided [-0.91 to -0.21], Standard Error of Mean 0.18
Statistical Analysis 13: Comparison: Placebo vs Tramadol; [analysis description as in outcome 22, analysis 11]; Test type: Superiority; p = 0.4173, ANCOVA; LS Mean Difference = -0.13, 95% CI 2-sided [-0.45 to 0.19], Standard Error of Mean 0.16
Statistical Analysis 14: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 22, analysis 11]; Test type: Superiority; p = 0.0659, ANCOVA; LS Mean Difference = -0.30, 95% CI 2-sided [-0.62 to 0.02], Standard Error of Mean 0.16
Statistical Analysis 15: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 22, analysis 11]; Test type: Superiority; p = 0.0078, ANCOVA; LS Mean Difference = -0.43, 95% CI 2-sided [-0.74 to -0.11], Standard Error of Mean 0.16
Statistical Analysis 16: Comparison: Placebo vs Pooled Tanezumab 5 mg; Change at Week 16: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf pain interference with walking ability, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.0737, ANCOVA; LS Mean Difference = -0.35, 95% CI 2-sided [-0.72 to 0.03], Standard Error of Mean 0.19
Statistical Analysis 17: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 22, analysis 16]; Test type: Superiority; p = 0.0021, ANCOVA; LS Mean Difference = -0.59, 95% CI 2-sided [-0.97 to -0.22], Standard Error of Mean 0.19
Statistical Analysis 18: Comparison: Placebo vs Tramadol; [analysis description as in outcome 22, analysis 16]; Test type: Superiority; p = 0.4535, ANCOVA; LS Mean Difference = -0.13, 95% CI 2-sided [-0.48 to 0.21], Standard Error of Mean 0.18
Statistical Analysis 19: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 22, analysis 16]; Test type: Superiority; p = 0.2271, ANCOVA; LS Mean Difference = -0.21, 95% CI 2-sided [-0.56 to 0.13], Standard Error of Mean 0.18
Statistical Analysis 20: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 22, analysis 16]; Test type: Superiority; p = 0.0086, ANCOVA; LS Mean Difference = -0.46, 95% CI 2-sided [-0.81 to -0.12], Standard Error of Mean 0.18
Statistical Analysis 21: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Change at Week 24: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf pain interference with walking ability, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.2243, ANCOVA; LS Mean Difference = -0.24, 95% CI 2-sided [-0.63 to 0.15], Standard Error of Mean 0.20
Statistical Analysis 22: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 22, analysis 21]; Test type: Superiority; p = 0.0331, ANCOVA; LS Mean Difference = -0.42, 95% CI 2-sided [-0.81 to -0.03], Standard Error of Mean 0.20
Statistical Analysis 23: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Change at Week 32: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf pain interference with walking ability, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.1838, ANCOVA; LS Mean Difference = -0.27, 95% CI 2-sided [-0.66 to 0.13], Standard Error of Mean 0.20
Statistical Analysis 24: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 22, analysis 23]; Test type: Superiority; p = 0.0795, ANCOVA; LS Mean Difference = -0.35, 95% CI 2-sided [-0.75 to 0.04], Standard Error of Mean 0.20
Statistical Analysis 25: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Change at Week 40: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf pain interference with walking ability, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.2847, ANCOVA; LS Mean Difference = -0.22, 95% CI 2-sided [-0.63 to 0.18], Standard Error of Mean 0.21
Statistical Analysis 26: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 22, analysis 25]; Test type: Superiority; p = 0.0745, ANCOVA; LS Mean Difference = -0.36, 95% CI 2-sided [-0.76 to 0.04], Standard Error of Mean 0.20
Statistical Analysis 27: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Change at Week 48: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf pain interference with walking ability, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.3110, ANCOVA; LS Mean Difference = -0.20, 95% CI 2-sided [-0.59 to 0.19], Standard Error of Mean 0.20
Statistical Analysis 28: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 22, analysis 27]; Test type: Superiority; p = 0.1375, ANCOVA; LS Mean Difference = -0.30, 95% CI 2-sided [-0.70 to 0.10], Standard Error of Mean 0.20
Statistical Analysis 29: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Change at Week 56: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf pain interference with walking ability, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.4036, ANCOVA; LS Mean Difference = -0.17, 95% CI 2-sided [-0.58 to 0.23], Standard Error of Mean 0.21
Statistical Analysis 30: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 22, analysis 29]; Test type: Superiority; p = 0.0641, ANCOVA; LS Mean Difference = -0.38, 95% CI 2-sided [-0.79 to 0.02], Standard Error of Mean 0.21

23. Secondary Outcome: Change From Baseline in Brief Pain Inventory-Short Form (BPI-sf) Score Pain Interference With Walking Ability at Week 64: Observed Data
Description: as for outcome 19
Time Frame: Baseline, Week 64
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Followed by Tanezumab 5 mg | Placebo Followed by Tanezumab 10 mg | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 202 | 204 | 407 | 407 | 605
units on a scale
  Baseline: number analyzed (Participants) | 202 | 204 | 405 | 407 | 605
  Baseline | 5.66 (2.28) | 6.07 (2.14) | 5.95 (2.22) | 6.01 (2.24) | 6.04 (2.03)
  Change at Week 64: number analyzed (Participants) | 63 | 57 | 140 | 147 | 200
  Change at Week 64 | -3.78 (2.91) | -4.14 (2.37) | -3.65 (2.79) | -3.61 (2.65) | -3.78 (2.37)

24. Secondary Outcome: Change From Baseline in Brief Pain Inventory-Short Form (BPI-sf) Score Pain Interference With Sleep at Weeks 2, 4, 8, 16, 24, 32, 40, 48 and 56: Observed Data
Description: as for outcome 18
Time Frame: Baseline, Weeks 2, 4, 8, 16, 24, 32, 40, 48 and 56
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 406 | 407 | 407 | 605
units on a scale
  Change at Week 2 | -1.58 (0.14) | -2.09 (0.13) | -2.15 (0.14) | -1.80 (0.11)
  Change at Week 4 | -2.13 (0.15) | -2.79 (0.15) | -2.98 (0.15) | -2.34 (0.13)
  Change at Week 8 | -2.42 (0.15) | -2.94 (0.15) | -3.13 (0.15) | -2.70 (0.13)
  Change at Week 16 | -2.92 (0.16) | -3.38 (0.16) | -3.44 (0.16) | -3.00 (0.14)
  Change at Week 24: number analyzed (Participants) | 0 | 407 | 407 | 605
  Change at Week 24 |  | -2.89 (0.18) | -3.09 (0.18) | -2.59 (0.15)
  Change at Week 32: number analyzed (Participants) | 0 | 407 | 407 | 605
  Change at Week 32 |  | -2.88 (0.18) | -2.94 (0.18) | -2.54 (0.15)
  Change at Week 40: number analyzed (Participants) | 0 | 407 | 407 | 605
  Change at Week 40 |  | -2.64 (0.18) | -2.81 (0.19) | -2.41 (0.15)
  Change at Week 48: number analyzed (Participants) | 0 | 407 | 407 | 605
  Change at Week 48 |  | -2.61 (0.19) | -2.73 (0.19) | -2.34 (0.16)
  Change at Week 56: number analyzed (Participants) | 0 | 407 | 407 | 605
  Change at Week 56 |  | -2.57 (0.18) | -2.74 (0.18) | -2.37 (0.16)
Statistical Analysis 1: Comparison: Placebo vs Pooled Tanezumab 5 mg; Change at Week 2: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf pain interference with sleep, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.0037, ANCOVA; LS Mean Difference = -0.51, 95% CI 2-sided [-0.85 to -0.17], Standard Error of Mean 0.18
Statistical Analysis 2: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 24, analysis 1]; Test type: Superiority; p = 0.0013, ANCOVA; LS Mean Difference = -0.57, 95% CI 2-sided [-0.91 to -0.22], Standard Error of Mean 0.18
Statistical Analysis 3: Comparison: Placebo vs Tramadol; [analysis description as in outcome 24, analysis 1]; Test type: Superiority; p = 0.1712, ANCOVA; LS Mean Difference = -0.22, 95% CI 2-sided [-0.53 to 0.09], Standard Error of Mean 0.16
Statistical Analysis 4: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 24, analysis 1]; Test type: Superiority; p = 0.0686, ANCOVA; LS Mean Difference = -0.29, 95% CI 2-sided [-0.60 to 0.02], Standard Error of Mean 0.16
Statistical Analysis 5: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 24, analysis 1]; Test type: Superiority; p = 0.0289, ANCOVA; LS Mean Difference = -0.35, 95% CI 2-sided [-0.66 to -0.04], Standard Error of Mean 0.16
Statistical Analysis 6: Comparison: Placebo vs Pooled Tanezumab 5 mg; Change at Week 4: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf pain interference with sleep, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.0003, ANCOVA; LS Mean Difference = -0.66, 95% CI 2-sided [-1.02 to -0.30], Standard Error of Mean 0.18
Statistical Analysis 7: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 24, analysis 6]; Test type: Superiority; p < .0001, ANCOVA; LS Mean Difference = -0.86, 95% CI 2-sided [-1.22 to -0.49], Standard Error of Mean 0.19
Statistical Analysis 8: Comparison: Placebo vs Tramadol; [analysis description as in outcome 24, analysis 6]; Test type: Superiority; p = 0.2056, ANCOVA; LS Mean Difference = -0.22, 95% CI 2-sided [-0.55 to 0.12], Standard Error of Mean 0.17
Statistical Analysis 9: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 24, analysis 6]; Test type: Superiority; p = 0.0084, ANCOVA; LS Mean Difference = -0.45, 95% CI 2-sided [-0.78 to -0.11], Standard Error of Mean 0.17
Statistical Analysis 10: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 24, analysis 6]; Test type: Superiority; p = 0.0002, ANCOVA; LS Mean Difference = -0.64, 95% CI 2-sided [-0.98 to -0.31], Standard Error of Mean 0.17
Statistical Analysis 11: Comparison: Placebo vs Pooled Tanezumab 5 mg; Change at Week 8: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf pain interference with sleep, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.0063, ANCOVA; LS Mean Difference = -0.52, 95% CI 2-sided [-0.90 to -0.15], Standard Error of Mean 0.19
Statistical Analysis 12: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 24, analysis 11]; Test type: Superiority; p = 0.0002, ANCOVA; LS Mean Difference = -0.72, 95% CI 2-sided [-1.09 to -0.34], Standard Error of Mean 0.19
Statistical Analysis 13: Comparison: Placebo vs Tramadol; [analysis description as in outcome 24, analysis 11]; Test type: Superiority; p = 0.1155, ANCOVA; LS Mean Difference = -0.28, 95% CI 2-sided [-0.63 to 0.07], Standard Error of Mean 0.18
Statistical Analysis 14: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 24, analysis 11]; Test type: Superiority; p = 0.1652, ANCOVA; LS Mean Difference = -0.24, 95% CI 2-sided [-0.59 to 0.10], Standard Error of Mean 0.18
Statistical Analysis 15: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 24, analysis 11]; Test type: Superiority; p = 0.0129, ANCOVA; LS Mean Difference = -0.44, 95% CI 2-sided [-0.78 to -0.09], Standard Error of Mean 0.18
Statistical Analysis 16: Comparison: Placebo vs Pooled Tanezumab 5 mg; Change at Week 16: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf pain interference with sleep, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.0236, ANCOVA; LS Mean Difference = -0.46, 95% CI 2-sided [-0.87 to -0.06], Standard Error of Mean 0.21
Statistical Analysis 17: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 24, analysis 16]; Test type: Superiority; p = 0.0136, ANCOVA; LS Mean Difference = -0.52, 95% CI 2-sided [-0.93 to -0.11], Standard Error of Mean 0.21
Statistical Analysis 18: Comparison: Placebo vs Tramadol; [analysis description as in outcome 24, analysis 16]; Test type: Superiority; p = 0.6624, ANCOVA; LS Mean Difference = -0.09, 95% CI 2-sided [-0.47 to 0.30], Standard Error of Mean 0.20
Statistical Analysis 19: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 24, analysis 16]; Test type: Superiority; p = 0.0468, ANCOVA; LS Mean Difference = -0.38, 95% CI 2-sided [-0.75 to -0.01], Standard Error of Mean 0.19
Statistical Analysis 20: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 24, analysis 16]; Test type: Superiority; p = 0.0250, ANCOVA; LS Mean Difference = -0.43, 95% CI 2-sided [-0.81 to -0.05], Standard Error of Mean 0.19
Statistical Analysis 21: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Change at Week 24: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf pain interference with sleep, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.1539, ANCOVA; LS Mean Difference = -0.30, 95% CI 2-sided [-0.72 to 0.11], Standard Error of Mean 0.21
Statistical Analysis 22: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 24, analysis 21]; Test type: Superiority; p = 0.0169, ANCOVA; LS Mean Difference = -0.50, 95% CI 2-sided [-0.91 to -0.09], Standard Error of Mean 0.21
Statistical Analysis 23: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Change at Week 32: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf pain interference with sleep, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.1049, ANCOVA; LS Mean Difference = -0.35, 95% CI 2-sided [-0.77 to 0.07], Standard Error of Mean 0.21
Statistical Analysis 24: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 24, analysis 23]; Test type: Superiority; p = 0.0599, ANCOVA; LS Mean Difference = -0.40, 95% CI 2-sided [-0.82 to 0.02], Standard Error of Mean 0.21
Statistical Analysis 25: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Change at Week 40: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf pain interference with sleep, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.3041, ANCOVA; LS Mean Difference = -0.22, 95% CI 2-sided [-0.65 to 0.20], Standard Error of Mean 0.22
Statistical Analysis 26: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 24, analysis 25]; Test type: Superiority; p = 0.0737, ANCOVA; LS Mean Difference = -0.40, 95% CI 2-sided [-0.83 to 0.04], Standard Error of Mean 0.22
Statistical Analysis 27: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Change at Week 48: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf pain interference with sleep, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.2293, ANCOVA; LS Mean Difference = -0.27, 95% CI 2-sided [-0.71 to 0.17], Standard Error of Mean 0.23
Statistical Analysis 28: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 24, analysis 27]; Test type: Superiority; p = 0.0806, ANCOVA; LS Mean Difference = -0.39, 95% CI 2-sided [-0.82 to 0.05], Standard Error of Mean 0.22
Statistical Analysis 29: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Change at Week 56: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf pain interference with sleep, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.3680, ANCOVA; LS Mean Difference = -0.20, 95% CI 2-sided [-0.62 to 0.23], Standard Error of Mean 0.22
Statistical Analysis 30: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 24, analysis 29]; Test type: Superiority; p = 0.0893, ANCOVA; LS Mean Difference = -0.36, 95% CI 2-sided [-0.79 to 0.06], Standard Error of Mean 0.21

25. Secondary Outcome: Change From Baseline in Brief Pain Inventory-Short Form (BPI-sf) Score Pain Interference With Sleep at Week 64: Observed Data
Description: as for outcome 19
Time Frame: Baseline, Week 64
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Followed by Tanezumab 5 mg | Placebo Followed by Tanezumab 10 mg | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 202 | 204 | 407 | 407 | 605
units on a scale
  Baseline: number analyzed (Participants) | 202 | 204 | 405 | 407 | 605
  Baseline | 6.45 (2.49) | 6.73 (2.37) | 6.88 (2.31) | 6.67 (2.39) | 6.82 (2.38)
  Change at Week 64: number analyzed (Participants) | 63 | 57 | 140 | 147 | 200
  Change at Week 64 | -4.29 (3.17) | -4.54 (2.80) | -4.19 (2.95) | -4.05 (2.70) | -4.11 (2.78)

26. Secondary Outcome: Change From Baseline in Brief Pain Inventory-Short Form (BPI-sf) Score Pain Interference With Normal Work at Weeks 2, 4, 8, 16, 24, 32, 40, 48 and 56: Observed Data
Description: as for outcome 18
Time Frame: Baseline, Weeks 2, 4, 8, 16, 24, 32, 40, 48 and 56
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 406 | 407 | 407 | 605
units on a scale
  Change at Week 2 | -1.30 (0.12) | -1.86 (0.12) | -2.01 (0.12) | -1.53 (0.10)
  Change at Week 4 | -1.92 (0.14) | -2.43 (0.14) | -2.81 (0.14) | -2.14 (0.12)
  Change at Week 8 | -2.32 (0.14) | -2.70 (0.14) | -2.96 (0.14) | -2.51 (0.12)
  Change at Week 16 | -2.64 (0.15) | -3.15 (0.15) | -3.33 (0.16) | -2.87 (0.13)
  Change at Week 24: number analyzed (Participants) | 0 | 407 | 407 | 605
  Change at Week 24 |  | -2.78 (0.17) | -2.89 (0.17) | -2.53 (0.15)
  Change at Week 32: number analyzed (Participants) | 0 | 407 | 407 | 605
  Change at Week 32 |  | -2.72 (0.18) | -2.75 (0.18) | -2.52 (0.15)
  Change at Week 40: number analyzed (Participants) | 0 | 407 | 407 | 605
  Change at Week 40 |  | -2.57 (0.18) | -2.60 (0.18) | -2.37 (0.15)
  Change at Week 48: number analyzed (Participants) | 0 | 407 | 407 | 605
  Change at Week 48 |  | -2.48 (0.18) | -2.49 (0.18) | -2.33 (0.15)
  Change at Week 56: number analyzed (Participants) | 0 | 407 | 407 | 605
  Change at Week 56 |  | -2.46 (0.18) | -2.58 (0.18) | -2.33 (0.16)
Statistical Analysis 1: Comparison: Placebo vs Pooled Tanezumab 5 mg; Change at Week 2: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf pain interference with normal work, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.0007, ANCOVA; LS Mean Difference = -0.56, 95% CI 2-sided [-0.88 to -0.24], Standard Error of Mean 0.16
Statistical Analysis 2: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 26, analysis 1]; Test type: Superiority; p < .0001, ANCOVA; LS Mean Difference = -0.71, 95% CI 2-sided [-1.03 to -0.38], Standard Error of Mean 0.17
Statistical Analysis 3: Comparison: Placebo vs Tramadol; [analysis description as in outcome 26, analysis 1]; Test type: Superiority; p = 0.1291, ANCOVA; LS Mean Difference = -0.23, 95% CI 2-sided [-0.53 to 0.07], Standard Error of Mean 0.15
Statistical Analysis 4: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 26, analysis 1]; Test type: Superiority; p = 0.0290, ANCOVA; LS Mean Difference = -0.33, 95% CI 2-sided [-0.63 to -0.03], Standard Error of Mean 0.15
Statistical Analysis 5: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 26, analysis 1]; Test type: Superiority; p = 0.0015, ANCOVA; LS Mean Difference = -0.48, 95% CI 2-sided [-0.77 to -0.18], Standard Error of Mean 0.15
Statistical Analysis 6: Comparison: Placebo vs Pooled Tanezumab 5 mg; Change at Week 4: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf pain interference with normal work, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.0041, ANCOVA; LS Mean Difference = -0.52, 95% CI 2-sided [-0.87 to -0.17], Standard Error of Mean 0.18
Statistical Analysis 7: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 26, analysis 6]; Test type: Superiority; p < .0001, ANCOVA; LS Mean Difference = -0.89, 95% CI 2-sided [-1.25 to -0.54], Standard Error of Mean 0.18
Statistical Analysis 8: Comparison: Placebo vs Tramadol; [analysis description as in outcome 26, analysis 6]; Test type: Superiority; p = 0.1799, ANCOVA; LS Mean Difference = -0.22, 95% CI 2-sided [-0.55 to 0.10], Standard Error of Mean 0.17
Statistical Analysis 9: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 26, analysis 6]; Test type: Superiority; p = 0.0696, ANCOVA; LS Mean Difference = -0.30, 95% CI 2-sided [-0.62 to 0.02], Standard Error of Mean 0.16
Statistical Analysis 10: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 26, analysis 6]; Test type: Superiority; p < .0001, ANCOVA; LS Mean Difference = -0.67, 95% CI 2-sided [-0.99 to -0.35], Standard Error of Mean 0.16
Statistical Analysis 11: Comparison: Placebo vs Pooled Tanezumab 5 mg; Change at Week 8: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf pain interference with normal work, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.0387, ANCOVA; LS Mean Difference = -0.38, 95% CI 2-sided [-0.74 to -0.02], Standard Error of Mean 0.18
Statistical Analysis 12: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 26, analysis 11]; Test type: Superiority; p = 0.0005, ANCOVA; LS Mean Difference = -0.64, 95% CI 2-sided [-1.00 to -0.28], Standard Error of Mean 0.18
Statistical Analysis 13: Comparison: Placebo vs Tramadol; [analysis description as in outcome 26, analysis 11]; Test type: Superiority; p = 0.2768, ANCOVA; LS Mean Difference = -0.18, 95% CI 2-sided [-0.51 to 0.15], Standard Error of Mean 0.17
Statistical Analysis 14: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 26, analysis 11]; Test type: Superiority; p = 0.2408, ANCOVA; LS Mean Difference = -0.20, 95% CI 2-sided [-0.53 to 0.13], Standard Error of Mean 0.17
Statistical Analysis 15: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 26, analysis 11]; Test type: Superiority; p = 0.0064, ANCOVA; LS Mean Difference = -0.46, 95% CI 2-sided [-0.78 to -0.13], Standard Error of Mean 0.17
Statistical Analysis 16: Comparison: Placebo vs Pooled Tanezumab 5 mg; Change at Week 16: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf pain interference with normal work, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.0115, ANCOVA; LS Mean Difference = -0.51, 95% CI 2-sided [-0.90 to -0.11], Standard Error of Mean 0.20
Statistical Analysis 17: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 26, analysis 16]; Test type: Superiority; p = 0.0006, ANCOVA; LS Mean Difference = -0.69, 95% CI 2-sided [-1.08 to -0.29], Standard Error of Mean 0.20
Statistical Analysis 18: Comparison: Placebo vs Tramadol; [analysis description as in outcome 26, analysis 16]; Test type: Superiority; p = 0.2028, ANCOVA; LS Mean Difference = -0.23, 95% CI 2-sided [-0.59 to 0.13], Standard Error of Mean 0.18
Statistical Analysis 19: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 26, analysis 16]; Test type: Superiority; p = 0.1351, ANCOVA; LS Mean Difference = -0.28, 95% CI 2-sided [-0.64 to 0.09], Standard Error of Mean 0.18
Statistical Analysis 20: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 26, analysis 16]; Test type: Superiority; p = 0.0133, ANCOVA; LS Mean Difference = -0.46, 95% CI 2-sided [-0.82 to -0.09], Standard Error of Mean 0.18
Statistical Analysis 21: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Change at Week 24: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf pain interference with normal work, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.2157, ANCOVA; LS Mean Difference = -0.25, 95% CI 2-sided [-0.65 to 0.15], Standard Error of Mean 0.20
Statistical Analysis 22: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 26, analysis 21]; Test type: Superiority; p = 0.0781, ANCOVA; LS Mean Difference = -0.36, 95% CI 2-sided [-0.76 to 0.04], Standard Error of Mean 0.20
Statistical Analysis 23: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Change at Week 32: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf pain interference with normal work, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.3527, ANCOVA; LS Mean Difference = -0.20, 95% CI 2-sided [-0.62 to 0.22], Standard Error of Mean 0.21
Statistical Analysis 24: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 26, analysis 23]; Test type: Superiority; p = 0.2994, ANCOVA; LS Mean Difference = -0.22, 95% CI 2-sided [-0.65 to 0.20], Standard Error of Mean 0.22
Statistical Analysis 25: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Change at Week 40: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf pain interference with normal work, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.3326, ANCOVA; LS Mean Difference = -0.21, 95% CI 2-sided [-0.63 to 0.21], Standard Error of Mean 0.22
Statistical Analysis 26: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 26, analysis 25]; Test type: Superiority; p = 0.2822, ANCOVA; LS Mean Difference = -0.23, 95% CI 2-sided [-0.65 to 0.19], Standard Error of Mean 0.21
Statistical Analysis 27: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Change at Week 48: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf pain interference with normal work, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.4932, ANCOVA; LS Mean Difference = -0.15, 95% CI 2-sided [-0.57 to 0.28], Standard Error of Mean 0.22
Statistical Analysis 28: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 26, analysis 27]; Test type: Superiority; p = 0.4571, ANCOVA; LS Mean Difference = -0.16, 95% CI 2-sided [-0.58 to 0.26], Standard Error of Mean 0.22
Statistical Analysis 29: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Change at Week 56: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline BPI-sf pain interference with normal work, and baseline average LBPI as covariates, and study site as a random effect; Test type: Superiority; p = 0.5586, ANCOVA; LS Mean Difference = -0.13, 95% CI 2-sided [-0.56 to 0.30], Standard Error of Mean 0.22
Statistical Analysis 30: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 26, analysis 29]; Test type: Superiority; p = 0.2664, ANCOVA; LS Mean Difference = -0.24, 95% CI 2-sided [-0.67 to 0.19], Standard Error of Mean 0.22

27. Secondary Outcome: Change From Baseline in Brief Pain Inventory-Short Form (BPI-sf) Score Pain Interference With Normal Work at Week 64: Observed Data
Description: as for outcome 19
Time Frame: Baseline, Week 64
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Followed by Tanezumab 5 mg | Placebo Followed by Tanezumab 10 mg | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 202 | 204 | 407 | 407 | 605
units on a scale
  Baseline: number analyzed (Participants) | 202 | 204 | 405 | 407 | 605
  Baseline | 6.31 (2.12) | 6.62 (2.03) | 6.65 (1.91) | 6.65 (1.90) | 6.56 (2.07)
  Change at Week 64: number analyzed (Participants) | 63 | 57 | 140 | 147 | 200
  Change at Week 64 | -3.95 (2.99) | -4.60 (2.46) | -4.15 (2.86) | -3.80 (2.71) | -4.08 (2.39)

28. Secondary Outcome: Number of Participants Who Responded for Chronic Low Back Pain Responder Index at Weeks 2, 4, 8, 16, 24, 32, 40, 48 and 56
Description: Chronic Low Back Pain Responder Index analysis is a composite endpoint of average low back pain intensity (aLBPI) score, PGA of Low Back Pain, and RMDQ total score. Participants were successful responders if they had: >=30 percent reduction in mean daily average LBPI from baseline to particular week; decrease of >=30 percent in PGA of low back pain from baseline to particular week or no worsening (increase) in RMDQ total score from baseline to particular week. Pre-specified intent of study for efficacy data up to W16 was to analyze participants who received placebo from Day1 and then received tanezumab 5/10 mg at W16,together,in placebo arm.Data has been reported per four arms. Also, intent of study was to compare tanezumab Vs placebo for data up to & including W16 & comparisons of tanezumab Vs tramadol for data up to & including W56.
Time Frame: Weeks 2, 4, 8, 16, 24, 32, 40, 48 and 56
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 404 | 404 | 406 | 605
Participants
  Week 2 | 32 | 62 | 76 | 74
  Week 4 | 67 | 115 | 130 | 134
  Week 8 | 86 | 131 | 151 | 178
  Week 16 | 136 | 168 | 179 | 211
  Week 24: number analyzed (Participants) | 0 | 404 | 406 | 605
  Week 24 |  | 166 | 158 | 207
  Week 32: number analyzed (Participants) | 0 | 404 | 406 | 605
  Week 32 |  | 158 | 160 | 204
  Week 40: number analyzed (Participants) | 0 | 404 | 406 | 605
  Week 40 |  | 158 | 149 | 202
  Week 48: number analyzed (Participants) | 0 | 404 | 406 | 605
  Week 48 |  | 148 | 140 | 197
  Week 56: number analyzed (Participants) | 0 | 404 | 406 | 605
  Week 56 |  | 140 | 144 | 192
Statistical Analysis 1: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 2: OR and 95% CI estimated from logistic regression model. Logistic regression model included treatment as fixed effect and baseline average LBPI, baseline PGA, and baseline RMDQ as covariates; Test type: Superiority; p = 0.0010, Regression, Logistic; Odds Ratio (OR) = 2.14, 95% CI 2-sided [1.36 to 3.36]
Statistical Analysis 2: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 28, analysis 1]; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 2.68, 95% CI 2-sided [1.73 to 4.16]
Statistical Analysis 3: Comparison: Placebo vs Tramadol; [analysis description as in outcome 28, analysis 1]; Test type: Superiority; p = 0.0300, Regression, Logistic; Odds Ratio (OR) = 1.62, 95% CI 2-sided [1.05 to 2.51]
Statistical Analysis 4: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 4: OR and 95% CI estimated from logistic regression model. Logistic regression model included treatment as fixed effect and baseline average LBPI, baseline PGA, and baseline RMDQ as covariates; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 2.03, 95% CI 2-sided [1.44 to 2.86]
Statistical Analysis 5: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 28, analysis 4]; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 2.37, 95% CI 2-sided [1.69 to 3.32]
Statistical Analysis 6: Comparison: Placebo vs Tramadol; [analysis description as in outcome 28, analysis 4]; Test type: Superiority; p = 0.0290, Regression, Logistic; Odds Ratio (OR) = 1.44, 95% CI 2-sided [1.04 to 1.99]
Statistical Analysis 7: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 8: OR and 95% CI estimated from logistic regression model. Logistic regression model included treatment as fixed effect and baseline average LBPI, baseline PGA, and baseline RMDQ as covariates; Test type: Superiority; p = 0.0003, Regression, Logistic; Odds Ratio (OR) = 1.80, 95% CI 2-sided [1.31 to 2.47]
Statistical Analysis 8: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 28, analysis 7]; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 2.21, 95% CI 2-sided [1.62 to 3.03]
Statistical Analysis 9: Comparison: Placebo vs Tramadol; [analysis description as in outcome 28, analysis 7]; Test type: Superiority; p = 0.0033, Regression, Logistic; Odds Ratio (OR) = 1.56, 95% CI 2-sided [1.16 to 2.10]
Statistical Analysis 10: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 16: OR and 95% CI estimated from logistic regression model. Logistic regression model included treatment as fixed effect and baseline average LBPI, baseline PGA, and baseline RMDQ as covariates; Test type: Superiority; p = 0.0179, Regression, Logistic; Odds Ratio (OR) = 1.41, 95% CI 2-sided [1.06 to 1.88]
Statistical Analysis 11: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 28, analysis 10]; Test type: Superiority; p = 0.0021, Regression, Logistic; Odds Ratio (OR) = 1.56, 95% CI 2-sided [1.18 to 2.08]
Statistical Analysis 12: Comparison: Placebo vs Tramadol; [analysis description as in outcome 28, analysis 10]; Test type: Superiority; p = 0.6629, Regression, Logistic; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.81 to 1.38]
Statistical Analysis 13: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 24: OR and 95% CI estimated from logistic regression model. Logistic regression model included treatment as fixed effect and baseline average LBPI, baseline PGA, and baseline RMDQ as covariates; Test type: Superiority; p = 0.0251, Regression, Logistic; Odds Ratio (OR) = 1.35, 95% CI 2-sided [1.04 to 1.75]
Statistical Analysis 14: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 28, analysis 13]; Test type: Superiority; p = 0.1278, Regression, Logistic; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.94 to 1.59]
Statistical Analysis 15: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 32: OR and 95% CI estimated from logistic regression model. Logistic regression model included treatment as fixed effect and baseline average LBPI, baseline PGA, and baseline RMDQ as covariates; Test type: Superiority; p = 0.0749, Regression, Logistic; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.98 to 1.65]
Statistical Analysis 16: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 28, analysis 15]; Test type: Superiority; p = 0.0633, Regression, Logistic; Odds Ratio (OR) = 1.28, 95% CI 2-sided [0.99 to 1.66]
Statistical Analysis 17: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 40: OR and 95% CI estimated from logistic regression model. Logistic regression model included treatment as fixed effect and baseline average LBPI, baseline PGA, and baseline RMDQ as covariates; Test type: Superiority; p = 0.0626, Regression, Logistic; Odds Ratio (OR) = 1.28, 95% CI 2-sided [0.99 to 1.67]
Statistical Analysis 18: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 28, analysis 17]; Test type: Superiority; p = 0.2727, Regression, Logistic; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.89 to 1.51]
Statistical Analysis 19: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 48: OR and 95% CI estimated from logistic regression model. Logistic regression model included treatment as fixed effect and baseline average LBPI, baseline PGA, and baseline RMDQ as covariates; Test type: Superiority; p = 0.1749, Regression, Logistic; Odds Ratio (OR) = 1.20, 95% CI 2-sided [0.92 to 1.57]
Statistical Analysis 20: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 28, analysis 19]; Test type: Superiority; p = 0.5239, Regression, Logistic; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.84 to 1.42]
Statistical Analysis 21: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 56: OR and 95% CI estimated from logistic regression model. Logistic regression model included treatment as fixed effect and baseline average LBPI, baseline PGA, and baseline RMDQ as covariates; Test type: Superiority; p = 0.3336, Regression, Logistic; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.87 to 1.49]
Statistical Analysis 22: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 28, analysis 21]; Test type: Superiority; p = 0.2163, Regression, Logistic; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.91 to 1.54]

29. Secondary Outcome: Percentage of Participants Achieving Improvement of >=2 Points in Patient's Global Assessment (PGA) of Low Back Pain From Baseline at Weeks 2, 4, 8, 16, 24, 32, 40, 48 and 56: Mixed Baseline Observation Carried Forward (BOCF)/ Last Observation CF (LOCF)
Description: PGA of LBP assessed by asking question to participants:Considering all ways your low back pain affects you,how are you doing today? They responded on 5 point Likert scale ranging from 1-5, using IRT, where 1=very good (asymptomatic & no limitation of normal activities);2=good (mild symptoms and no limitation of normal activities);3=fair (moderate symptoms and limitation of some normal activities);4=poor (severe symptoms & inability to carry out most normal activities); & 5=very poor (very severe symptoms which are intolerable and inability to carry out all normal activities). Higher scores indicated worsening of condition. % of participants with improvement of at least 2 points from baseline in PGA of LBP were reported. Missing data was imputed using BOCF/LOCF. Pre-specified intent of study for efficacy data up to W16 was to analyze participants who received placebo from Day1 and then received tanezumab 5/10 mg at W16,together,in placebo arm.Data has been reported per four arms.
Time Frame: Baseline, Weeks 2, 4, 8, 16, 24, 32, 40, 48 and 56
Population: ITT population.Data were not collected after W16 in placebo arm for this OM, as those who met criteria to continue, switched to active treatment with tan after W16. N =participants evaluable for this OM. intent of study was to compare tan Vs placebo for data up to & including W16 & comparisons of tan Vs tramadol for data up to & including W56.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 406 | 405 | 407 | 605
percentage of participants
  Week 2 | 9.4 | 11.1 | 14.7 | 10.1
  Week 4 | 13.8 | 20.5 | 21.4 | 15.0
  Week 8 | 15.3 | 20.2 | 24.1 | 18.8
  Week 16 | 22.7 | 27.4 | 30.0 | 22.5
  Week 24: number analyzed (Participants) | 0 | 405 | 407 | 605
  Week 24 |  | 25.9 | 25.1 | 21.5
  Week 32: number analyzed (Participants) | 0 | 405 | 407 | 605
  Week 32 |  | 25.2 | 23.1 | 20.7
  Week 40: number analyzed (Participants) | 0 | 405 | 407 | 605
  Week 40 |  | 25.9 | 22.9 | 20.7
  Week 48: number analyzed (Participants) | 0 | 405 | 407 | 605
  Week 48 |  | 23.2 | 22.4 | 20.5
  Week 56: number analyzed (Participants) | 0 | 405 | 407 | 605
  Week 56 |  | 24.2 | 21.1 | 20.5
Statistical Analysis 1: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 2: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline PGA of low back pain, baseline average LBPI, and treatment; Test type: Superiority; p = 0.3260, Regression, Logistic; Odds Ratio (OR) = 1.28, 95% CI 2-sided [0.78 to 2.08]
Statistical Analysis 2: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 29, analysis 1]; Test type: Superiority; p = 0.0445, Regression, Logistic; Odds Ratio (OR) = 1.61, 95% CI 2-sided [1.01 to 2.56]
Statistical Analysis 3: Comparison: Placebo vs Tramadol; [analysis description as in outcome 29, analysis 1]; Test type: Superiority; p = 0.9263, Regression, Logistic; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.65 to 1.61]
Statistical Analysis 4: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 29, analysis 1]; Test type: Superiority; p = 0.3194, Regression, Logistic; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.81 to 1.94]
Statistical Analysis 5: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 29, analysis 1]; Test type: Superiority; p = 0.0308, Regression, Logistic; Odds Ratio (OR) = 1.58, 95% CI 2-sided [1.04 to 2.38]
Statistical Analysis 6: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 4: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline PGA of low back pain, baseline average LBPI, and treatment; Test type: Superiority; p = 0.0048, Regression, Logistic; Odds Ratio (OR) = 1.79, 95% CI 2-sided [1.20 to 2.69]
Statistical Analysis 7: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 29, analysis 6]; Test type: Superiority; p = 0.0114, Regression, Logistic; Odds Ratio (OR) = 1.68, 95% CI 2-sided [1.12 to 2.51]
Statistical Analysis 8: Comparison: Placebo vs Tramadol; [analysis description as in outcome 29, analysis 6]; Test type: Superiority; p = 0.7857, Regression, Logistic; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.71 to 1.56]
Statistical Analysis 9: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 29, analysis 6]; Test type: Superiority; p = 0.0041, Regression, Logistic; Odds Ratio (OR) = 1.70, 95% CI 2-sided [1.18 to 2.44]
Statistical Analysis 10: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 29, analysis 6]; Test type: Superiority; p = 0.0109, Regression, Logistic; Odds Ratio (OR) = 1.59, 95% CI 2-sided [1.11 to 2.28]
Statistical Analysis 11: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 8: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline PGA of low back pain, baseline average LBPI, and treatment; Test type: Superiority; p = 0.0363, Regression, Logistic; Odds Ratio (OR) = 1.53, 95% CI 2-sided [1.03 to 2.27]
Statistical Analysis 12: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 29, analysis 11]; Test type: Superiority; p = 0.0040, Regression, Logistic; Odds Ratio (OR) = 1.76, 95% CI 2-sided [1.20 to 2.59]
Statistical Analysis 13: Comparison: Placebo vs Tramadol; [analysis description as in outcome 29, analysis 11]; Test type: Superiority; p = 0.1992, Regression, Logistic; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.88 to 1.84]
Statistical Analysis 14: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 29, analysis 11]; Test type: Superiority; p = 0.3084, Regression, Logistic; Odds Ratio (OR) = 1.20, 95% CI 2-sided [0.85 to 1.70]
Statistical Analysis 15: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 29, analysis 11]; Test type: Superiority; p = 0.0586, Regression, Logistic; Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.99 to 1.94]
Statistical Analysis 16: Comparison: Placebo vs Pooled Tanezumab 5 mg; Week 16: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline PGA of low back pain, baseline average LBPI, and treatment; Test type: Superiority; p = 0.0630, Regression, Logistic; Odds Ratio (OR) = 1.39, 95% CI 2-sided [0.98 to 1.97]
Statistical Analysis 17: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 29, analysis 16]; Test type: Superiority; p = 0.0347, Regression, Logistic; Odds Ratio (OR) = 1.45, 95% CI 2-sided [1.03 to 2.04]
Statistical Analysis 18: Comparison: Placebo vs Tramadol; [analysis description as in outcome 29, analysis 16]; Test type: Superiority; p = 0.7900, Regression, Logistic; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.69 to 1.33]
Statistical Analysis 19: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 29, analysis 16]; Test type: Superiority; p = 0.0207, Regression, Logistic; Odds Ratio (OR) = 1.45, 95% CI 2-sided [1.06 to 2.00]
Statistical Analysis 20: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 29, analysis 16]; Test type: Superiority; p = 0.0093, Regression, Logistic; Odds Ratio (OR) = 1.51, 95% CI 2-sided [1.11 to 2.07]
Statistical Analysis 21: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 24: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline PGA of low back pain, baseline average LBPI, and treatment; Test type: Superiority; p = 0.0400, Regression, Logistic; Odds Ratio (OR) = 1.39, 95% CI 2-sided [1.02 to 1.91]
Statistical Analysis 22: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 29, analysis 21]; Test type: Superiority; p = 0.2478, Regression, Logistic; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.88 to 1.65]
Statistical Analysis 23: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 32: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline PGA of low back pain, baseline average LBPI, and treatment; Test type: Superiority; p = 0.0304, Regression, Logistic; Odds Ratio (OR) = 1.42, 95% CI 2-sided [1.03 to 1.96]
Statistical Analysis 24: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 29, analysis 23]; Test type: Superiority; p = 0.4763, Regression, Logistic; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.81 to 1.56]
Statistical Analysis 25: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 40: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline PGA of low back pain, baseline average LBPI, and treatment; Test type: Superiority; p = 0.0178, Regression, Logistic; Odds Ratio (OR) = 1.47, 95% CI 2-sided [1.07 to 2.01]
Statistical Analysis 26: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 29, analysis 25]; Test type: Superiority; p = 0.5223, Regression, Logistic; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.80 to 1.53]
Statistical Analysis 27: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 48: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline PGA of low back pain, baseline average LBPI, and treatment; Test type: Superiority; p = 0.1708, Regression, Logistic; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.91 to 1.72]
Statistical Analysis 28: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 29, analysis 27]; Test type: Superiority; p = 0.6022, Regression, Logistic; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.79 to 1.50]
Statistical Analysis 29: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 56: OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline PGA of low back pain, baseline average LBPI, and treatment; Test type: Superiority; p = 0.0846, Regression, Logistic; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.96 to 1.81]
Statistical Analysis 30: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 29, analysis 29]; Test type: Superiority; p = 0.9626, Regression, Logistic; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.73 to 1.39]

30. Secondary Outcome: European Quality of Life- 5 Dimension-5 Levels (EQ-5D-5L) Dimensions Score
Description: EQ-5D-5L is a standardized participant completed questionnaire that measures health-related quality of life and translates that score into an index value or utility score. EQ-5D-5L consists of two components: a health state profile and an optional visual analogue scale (VAS). EQ-5D health state profile is comprised of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Individual dimension scores ranged from 1.0 (least impairment of health state) to 5.0 (most impairment of health state). Each dimension has 5 levels: 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, and 5=extreme problems. The health utility score for a participant with no problems in all 5 items is 1 for all countries (except for Zimbabwe where it is 0.9), and is reduced where a participant reports greater levels of problems across the five dimensions.
Time Frame: Baseline, Weeks 8, 16, 24, 40 and 56
Population: ITT population included all randomized participants who received at least one dose of SC study medication (either tanezumab or matching placebo). Here, 'n' = Participants evaluable for this OM for specified categories.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Followed by Tanezumab 5 mg | Placebo Followed by Tanezumab 10 mg | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 202 | 204 | 407 | 407 | 605
units on a scale
  Baseline: Mobility: number analyzed (Participants) | 202 | 204 | 405 | 407 | 605
  Baseline: Mobility | 2.5 (0.84) | 2.6 (0.88) | 2.5 (0.83) | 2.6 (0.82) | 2.6 (0.86)
  Baseline: Self-care: number analyzed (Participants) | 202 | 204 | 405 | 407 | 605
  Baseline: Self-care | 2.0 (0.95) | 2.1 (0.97) | 2.0 (0.95) | 2.0 (0.92) | 2.0 (0.95)
  Baseline: Usual activities: number analyzed (Participants) | 202 | 204 | 405 | 407 | 605
  Baseline: Usual activities | 2.8 (0.90) | 2.8 (0.83) | 2.8 (0.82) | 2.8 (0.80) | 2.8 (0.84)
  Baseline: Pain/Discomfort: number analyzed (Participants) | 202 | 204 | 405 | 407 | 605
  Baseline: Pain/Discomfort | 3.3 (0.73) | 3.4 (0.71) | 3.4 (0.68) | 3.3 (0.69) | 3.3 (0.70)
  Baseline: Anxiety/Depression: number analyzed (Participants) | 202 | 204 | 405 | 407 | 605
  Baseline: Anxiety/Depression | 1.8 (0.99) | 1.9 (1.03) | 1.9 (1.01) | 1.9 (0.98) | 1.9 (1.00)
  Week 8: Mobility: number analyzed (Participants) | 183 | 184 | 374 | 375 | 557
  Week 8: Mobility | 1.9 (0.78) | 2.0 (0.90) | 1.8 (0.85) | 1.8 (0.81) | 1.9 (0.87)
  Week 8: Self-care: number analyzed (Participants) | 183 | 184 | 374 | 375 | 557
  Week 8: Self-care | 1.5 (0.71) | 1.7 (0.79) | 1.4 (0.66) | 1.4 (0.65) | 1.5 (0.73)
  Week 8: Usual activities: number analyzed (Participants) | 183 | 184 | 374 | 375 | 557
  Week 8: Usual activities | 2.2 (0.81) | 2.2 (0.89) | 2.0 (0.85) | 2.0 (0.82) | 2.1 (0.91)
  Week 8: Pain/Discomfort: number analyzed (Participants) | 183 | 184 | 374 | 375 | 557
  Week 8: Pain/Discomfort | 2.7 (0.82) | 2.6 (0.84) | 2.5 (0.80) | 2.4 (0.80) | 2.5 (0.79)
  Week 8: Anxiety/Depression: number analyzed (Participants) | 183 | 184 | 374 | 375 | 557
  Week 8: Anxiety/Depression | 1.5 (0.81) | 1.6 (0.92) | 1.5 (0.83) | 1.5 (0.78) | 1.6 (0.84)
  Week 16: Mobility: number analyzed (Participants) | 161 | 163 | 333 | 338 | 452
  Week 16: Mobility | 1.7 (0.82) | 1.8 (0.85) | 1.7 (0.78) | 1.6 (0.75) | 1.8 (0.79)
  Week 16: Self-care: number analyzed (Participants) | 161 | 163 | 333 | 338 | 452
  Week 16: Self-care | 1.4 (0.64) | 1.5 (0.72) | 1.3 (0.62) | 1.3 (0.61) | 1.5 (0.69)
  Week 16: Usual activities: number analyzed (Participants) | 161 | 163 | 333 | 338 | 452
  Week 16: Usual activities | 1.9 (0.81) | 2.0 (0.85) | 1.8 (0.84) | 1.8 (0.80) | 1.9 (0.82)
  Week 16: Pain/Discomfort: number analyzed (Participants) | 161 | 163 | 333 | 338 | 452
  Week 16: Pain/Discomfort | 2.3 (0.90) | 2.4 (0.86) | 2.2 (0.83) | 2.2 (0.75) | 2.3 (0.76)
  Week 16: Anxiety/Depression: number analyzed (Participants) | 161 | 163 | 333 | 338 | 452
  Week 16: Anxiety/Depression | 1.4 (0.68) | 1.5 (0.82) | 1.5 (0.83) | 1.4 (0.77) | 1.5 (0.79)
  Week 24: Mobility: number analyzed (Participants) | 86 | 88 | 222 | 227 | 285
  Week 24: Mobility | 1.5 (0.63) | 1.6 (0.79) | 1.6 (0.75) | 1.5 (0.66) | 1.7 (0.75)
  Week 24: Self-care: number analyzed (Participants) | 86 | 88 | 222 | 227 | 285
  Week 24: Self-care | 1.3 (0.47) | 1.4 (0.75) | 1.3 (0.58) | 1.2 (0.51) | 1.3 (0.59)
  Week 24: Usual activities: number analyzed (Participants) | 86 | 88 | 222 | 227 | 285
  Week 24: Usual activities | 1.6 (0.68) | 1.7 (0.71) | 1.6 (0.71) | 1.7 (0.67) | 1.7 (0.72)
  Week 24: Pain/Discomfort: number analyzed (Participants) | 86 | 88 | 222 | 227 | 285
  Week 24: Pain/Discomfort | 2.0 (0.64) | 1.9 (0.70) | 2.1 (0.76) | 2.0 (0.74) | 2.1 (0.75)
  Week 24: Anxiety/Depression: number analyzed (Participants) | 86 | 88 | 222 | 227 | 285
  Week 24: Anxiety/Depression | 1.2 (0.44) | 1.3 (0.64) | 1.4 (0.73) | 1.3 (0.65) | 1.3 (0.66)
  Week 40: Mobility: number analyzed (Participants) | 70 | 73 | 162 | 174 | 225
  Week 40: Mobility | 1.5 (0.76) | 1.5 (0.62) | 1.5 (0.75) | 1.5 (0.70) | 1.6 (0.73)
  Week 40: Self-care: number analyzed (Participants) | 70 | 73 | 162 | 174 | 225
  Week 40: Self-care | 1.2 (0.62) | 1.3 (0.53) | 1.2 (0.46) | 1.2 (0.45) | 1.3 (0.62)
  Week 40: Usual activities: number analyzed (Participants) | 70 | 73 | 162 | 174 | 225
  Week 40: Usual activities | 1.6 (0.69) | 1.6 (0.73) | 1.6 (0.72) | 1.7 (0.68) | 1.7 (0.76)
  Week 40: Pain/Discomfort: number analyzed (Participants) | 70 | 73 | 162 | 174 | 225
  Week 40: Pain/Discomfort | 1.9 (0.62) | 1.9 (0.64) | 2.0 (0.73) | 1.9 (0.75) | 2.0 (0.72)
  Week 40: Anxiety/Depression: number analyzed (Participants) | 70 | 73 | 162 | 174 | 225
  Week 40: Anxiety/Depression | 1.2 (0.49) | 1.3 (0.60) | 1.3 (0.64) | 1.3 (0.68) | 1.4 (0.63)
  Week 56: Mobility: number analyzed (Participants) | 62 | 62 | 134 | 154 | 197
  Week 56: Mobility | 1.4 (0.61) | 1.5 (0.72) | 1.5 (0.69) | 1.4 (0.67) | 1.6 (0.83)
  Week 56: Self-care: number analyzed (Participants) | 62 | 62 | 134 | 154 | 197
  Week 56: Self-care | 1.1 (0.44) | 1.3 (0.52) | 1.2 (0.55) | 1.2 (0.43) | 1.4 (0.66)
  Week 56: Usual activities: number analyzed (Participants) | 62 | 62 | 134 | 154 | 197
  Week 56: Usual activities | 1.6 (0.82) | 1.6 (0.69) | 1.6 (0.78) | 1.6 (0.73) | 1.7 (0.82)
  Week 56: Pain/Discomfort: number analyzed (Participants) | 62 | 62 | 134 | 154 | 197
  Week 56: Pain/Discomfort | 2.0 (0.77) | 1.9 (0.66) | 2.0 (0.72) | 1.9 (0.72) | 2.0 (0.74)
  Week 56: Anxiety/Depression: number analyzed (Participants) | 62 | 62 | 134 | 154 | 197
  Week 56: Anxiety/Depression | 1.3 (0.54) | 1.3 (0.55) | 1.4 (0.77) | 1.3 (0.70) | 1.3 (0.63)

31. Secondary Outcome: European Quality of Life- 5 Dimension-5 Levels (EQ-5D-5L) Overall Health Utility Score/ Index Value
Description: EQ-5D-5L: standardized participant completed questionnaire that measures health-related quality of life and translates that score into an index value or utility score.EQ-5D-5L consists of 2 components: a health state profile and an optional VAS.EQ-5D health state profile comprises of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression.Individual dimension scores ranged from 1.0(least impairment of health state) to 5.0(most impairment of health state). Each dimension has 5 levels: 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems, and 5=extreme problems.Responses from five domains were used to calculate a single utility index (Overall health utility score) where values are less than equal to (<=) 1.Overall health utility score for a participant with no problems in all 5 items is 1 for all countries (except for Zimbabwe where it is 0.9), and reduced where participant reports greater levels of problems across five dimensions.
Time Frame: Baseline, Weeks 8, 16, 24, 40, 56 and 64
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Followed by Tanezumab 5 mg | Placebo Followed by Tanezumab 10 mg | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 202 | 204 | 407 | 407 | 605
units on a scale
  Baseline: number analyzed (Participants) | 202 | 204 | 405 | 407 | 605
  Baseline | 0.62 (0.16) | 0.61 (0.15) | 0.61 (0.16) | 0.62 (0.16) | 0.61 (0.16)
  Week 8: number analyzed (Participants) | 183 | 184 | 374 | 375 | 557
  Week 8 | 0.74 (0.13) | 0.71 (0.14) | 0.75 (0.13) | 0.76 (0.14) | 0.74 (0.14)
  Week 16: number analyzed (Participants) | 161 | 163 | 333 | 338 | 452
  Week 16 | 0.77 (0.14) | 0.75 (0.14) | 0.78 (0.14) | 0.79 (0.13) | 0.77 (0.13)
  Week 24: number analyzed (Participants) | 86 | 88 | 222 | 227 | 285
  Week 24 | 0.82 (0.10) | 0.81 (0.13) | 0.80 (0.13) | 0.82 (0.12) | 0.80 (0.12)
  Week 40: number analyzed (Participants) | 70 | 73 | 162 | 174 | 225
  Week 40 | 0.83 (0.11) | 0.82 (0.12) | 0.82 (0.12) | 0.83 (0.12) | 0.80 (0.14)
  Week 56: number analyzed (Participants) | 62 | 62 | 134 | 154 | 197
  Week 56 | 0.85 (0.11) | 0.82 (0.13) | 0.82 (0.14) | 0.84 (0.12) | 0.81 (0.14)

32. Secondary Outcome: Work Productivity and Activity Impairment Questionnaire for Low Back Pain (WPAI:LBP) Scores at Baseline: Observed Data
Description: WPAI: LBP is 6-question participant rated questionnaire that measures the effect of participant's chronic low back pain (CLBP) on general health and symptom severity on work productivity and regular activities. It yields 4 sub-scores: work time missed due to pain (absenteeism), impairment while working (presenteeism), overall work impairment (work productivity) and activity impairment (daily activity impairment). These sub-scores are expressed as an impairment percentage (range from 0 to 100), with higher numbers indicating greater impairment and less productivity. Pre-specified intent of study for efficacy data up to Week 16 was to analyze, participants who received placebo from Day 1 and received tanezumab 5/10 mg at week 16 in placebo arm, in pooled manner. Hence data have been reported per four arms.
Time Frame: Baseline
Population: ITT population was analyzed.'n' = Participants evaluable for this OM for specified categories. Pre-specified intent of study was w compare tanezumab Vs placebo for data up to and including week 16 and comparisons of tanezumab Vs tramadol for data up to and including week 56. Number analyzed is 0 for placebo arm for week 16 and onwards.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 406 | 407 | 407 | 605
units on a scale
  Percent Work Time Missed: number analyzed (Participants) | 232 | 236 | 236 | 316
  Percent Work Time Missed | 8.2 (17.43) | 11.1 (21.03) | 10.8 (19.89) | 10.7 (20.12)
  Percent Impairment While Working: number analyzed (Participants) | 229 | 230 | 232 | 313
  Percent Impairment While Working | 57.9 (21.25) | 60.8 (19.68) | 60.6 (20.56) | 61.2 (19.83)
  Percent Overall Work Impairment: number analyzed (Participants) | 229 | 230 | 232 | 313
  Percent Overall Work Impairment | 60.2 (22.11) | 63.2 (20.34) | 63.1 (21.69) | 63.6 (20.93)
  Percent Activity Impairment: number analyzed (Participants) | 406 | 405 | 407 | 605
  Percent Activity Impairment | 65.7 (18.13) | 66.6 (17.57) | 65.1 (18.33) | 65.4 (18.31)

33. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment Questionnaire for Low Back Pain (WPAI:LBP) Scores at Weeks 16, 56 and 64
Description: WPAI: LBP is 6-question participant rated questionnaire that measures the effect of participant's chronic low back pain (CLBP) on general health and symptom severity on work productivity and regular activities. It yields 4 sub-scores: work time missed due to pain (absenteeism), impairment while working (presenteeism), overall work impairment (work productivity) and activity impairment (daily activity impairment). These sub-scores are expressed as an impairment percentage (range from 0 to 100), with higher numbers indicating greater impairment and less productivity. Pre-specified intent of study for efficacy data up to W16 was to analyze participants who received placebo from Day1 and then received tanezumab 5/10 mg at W16,together,in placebo arm.Data has been reported per four arms.
Time Frame: Baseline, Weeks 16, 56 and 64
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 406 | 407 | 407 | 605
units on a scale
  Change at Week 16: Percent Work Time Missed: number analyzed (Participants) | 171 | 179 | 174 | 208
  Change at Week 16: Percent Work Time Missed | -5.82 (1.18) | -5.07 (1.15) | -5.89 (1.16) | -5.68 (1.07)
  Change at Week 16:Percent Impairment While Working: number analyzed (Participants) | 166 | 173 | 170 | 204
  Change at Week 16:Percent Impairment While Working | -25.46 (1.75) | -29.49 (1.71) | -30.22 (1.72) | -27.11 (1.58)
  Change at Week 16: Percent Overall Work Impairment: number analyzed (Participants) | 166 | 173 | 170 | 204
  Change at Week 16: Percent Overall Work Impairment | -26.54 (1.80) | -30.49 (1.75) | -31.95 (1.77) | -28.29 (1.62)
  Change at Week 16: Percent Activity Impairment: number analyzed (Participants) | 329 | 337 | 343 | 457
  Change at Week 16: Percent Activity Impairment | -28.07 (1.39) | -32.25 (1.38) | -32.25 (1.38) | -30.83 (1.23)
  Change at Week 56: Percent Work Time Missed: number analyzed (Participants) | 0 | 77 | 77 | 87
  Change at Week 56: Percent Work Time Missed |  | -8.06 (1.11) | -7.48 (1.11) | -7.19 (1.05)
  Change at Week 56:Percent Impairment While Working: number analyzed (Participants) | 0 | 76 | 76 | 87
  Change at Week 56:Percent Impairment While Working |  | -39.38 (2.03) | -41.32 (2.02) | -38.51 (1.89)
  Change at Week 56: Percent Overall Work Impairment: number analyzed (Participants) | 0 | 76 | 76 | 87
  Change at Week 56: Percent Overall Work Impairment |  | -41.18 (2.18) | -42.63 (2.18) | -39.25 (2.04)
  Change at Week 56: Percent Activity Impairment: number analyzed (Participants) | 0 | 134 | 154 | 197
  Change at Week 56: Percent Activity Impairment |  | -43.53 (1.75) | -44.16 (1.63) | -43.00 (1.47)
Statistical Analysis 1: Comparison: Placebo vs Pooled Tanezumab 5 mg; Change at Week 16: Percent Work Time Missed: ANCOVA model included treatment as fixed effects, baseline WPAI score and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.6508, ANCOVA; LS Mean Difference = 0.74, 95% CI 2-sided [-2.49 to 3.98], Standard Error of Mean 1.64
Statistical Analysis 2: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 33, analysis 1]; Test type: Superiority; p = 0.9629, ANCOVA; LS Mean Difference = -0.08, 95% CI 2-sided [-3.33 to 3.18], Standard Error of Mean 1.66
Statistical Analysis 3: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 33, analysis 1]; Test type: Superiority; p = 0.7007, ANCOVA; LS Mean Difference = 0.60, 95% CI 2-sided [-2.48 to 3.69], Standard Error of Mean 1.57
Statistical Analysis 4: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 33, analysis 1]; Test type: Superiority; p = 0.8902, ANCOVA; LS Mean Difference = -0.22, 95% CI 2-sided [-3.32 to 2.88], Standard Error of Mean 1.58
Statistical Analysis 5: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Change at Week 56: Percent Work Time Missed: ANCOVA model included treatment as fixed effects, baseline WPAI score and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.5698, ANCOVA; LS Mean Difference = -0.87, 95% CI 2-sided [-3.89 to 2.15], Standard Error of Mean 1.53
Statistical Analysis 6: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 33, analysis 5]; Test type: Superiority; p = 0.8464, ANCOVA; LS Mean Difference = -0.30, 95% CI 2-sided [-3.32 to 2.72], Standard Error of Mean 1.53
Statistical Analysis 7: Comparison: Placebo vs Pooled Tanezumab 5 mg; Change at Week 16: Percent Impairment While Working: ANCOVA model included treatment as fixed effects, baseline WPAI score and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.0919, ANCOVA; LS Mean Difference = -4.03, 95% CI 2-sided [-8.72 to 0.66], Standard Error of Mean 2.39
Statistical Analysis 8: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 33, analysis 7]; Test type: Superiority; p = 0.0477, ANCOVA; LS Mean Difference = -4.76, 95% CI 2-sided [-9.47 to -0.05], Standard Error of Mean 2.40
Statistical Analysis 9: Comparison: Placebo vs Tramadol; [analysis description as in outcome 33, analysis 7]; Test type: Superiority; p = 0.4735, ANCOVA; LS Mean Difference = -1.65, 95% CI 2-sided [-6.17 to 2.87], Standard Error of Mean 2.30
Statistical Analysis 10: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 33, analysis 7]; Test type: Superiority; p = 0.2935, ANCOVA; LS Mean Difference = -2.38, 95% CI 2-sided [-6.82 to 2.06], Standard Error of Mean 2.26
Statistical Analysis 11: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 33, analysis 7]; Test type: Superiority; p = 0.1714, ANCOVA; LS Mean Difference = -3.11, 95% CI 2-sided [-7.56 to 1.35], Standard Error of Mean 2.27
Statistical Analysis 12: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Change at Week 56: Percent Impairment While Working: ANCOVA model included treatment as fixed effects, baseline WPAI score and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.7521, ANCOVA; LS Mean Difference = -0.87, 95% CI 2-sided [-6.30 to 4.56], Standard Error of Mean 2.75
Statistical Analysis 13: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 33, analysis 12]; Test type: Superiority; p = 0.3078, ANCOVA; LS Mean Difference = -2.81, 95% CI 2-sided [-8.24 to 2.61], Standard Error of Mean 2.75
Statistical Analysis 14: Comparison: Placebo vs Pooled Tanezumab 5 mg; Change at Week 16: Percent Overall Work Impairment: ANCOVA model included treatment as fixed effects, baseline WPAI score and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.1090, ANCOVA; LS Mean Difference = -3.95, 95% CI 2-sided [-8.78 to 0.88], Standard Error of Mean 2.46
Statistical Analysis 15: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 33, analysis 14]; Test type: Superiority; p = 0.0289, ANCOVA; LS Mean Difference = -5.41, 95% CI 2-sided [-10.27 to -0.56], Standard Error of Mean 2.47
Statistical Analysis 16: Comparison: Placebo vs Tramadol; [analysis description as in outcome 33, analysis 14]; Test type: Superiority; p = 0.4613, ANCOVA; LS Mean Difference = -1.75, 95% CI 2-sided [-6.41 to 2.91], Standard Error of Mean 2.37
Statistical Analysis 17: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 33, analysis 14]; Test type: Superiority; p = 0.3460, ANCOVA; LS Mean Difference = -2.20, 95% CI 2-sided [-6.78 to 2.38], Standard Error of Mean 2.33
Statistical Analysis 18: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 33, analysis 14]; Test type: Superiority; p = 0.1179, ANCOVA; LS Mean Difference = -3.66, 95% CI 2-sided [-8.26 to 0.93], Standard Error of Mean 2.34
Statistical Analysis 19: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Change at Week 56: Percent Overall Work Impairment: ANCOVA model included treatment as fixed effects, baseline WPAI score and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.5151, ANCOVA; LS Mean Difference = -1.93, 95% CI 2-sided [-7.78 to 3.92], Standard Error of Mean 2.97
Statistical Analysis 20: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 33, analysis 19]; Test type: Superiority; p = 0.2550, ANCOVA; LS Mean Difference = -3.38, 95% CI 2-sided [-9.22 to 2.46], Standard Error of Mean 2.96
Statistical Analysis 21: Comparison: Placebo vs Pooled Tanezumab 5 mg; Change at Week 16: Percent Activity Impairment: ANCOVA model included treatment as fixed effects, baseline WPAI score and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.0157, ANCOVA; LS Mean Difference = -4.18, 95% CI 2-sided [-7.57 to -0.79], Standard Error of Mean 1.73
Statistical Analysis 22: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 33, analysis 21]; Test type: Superiority; p = 0.0159, ANCOVA; LS Mean Difference = -4.18, 95% CI 2-sided [-7.57 to -0.78], Standard Error of Mean 1.73
Statistical Analysis 23: Comparison: Placebo vs Tramadol; [analysis description as in outcome 33, analysis 21]; Test type: Superiority; p = 0.0896, ANCOVA; LS Mean Difference = -2.75, 95% CI 2-sided [-5.94 to 0.43], Standard Error of Mean 1.62
Statistical Analysis 24: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 33, analysis 21]; Test type: Superiority; p = 0.3749, ANCOVA; LS Mean Difference = -1.42, 95% CI 2-sided [-4.57 to 1.72], Standard Error of Mean 1.60
Statistical Analysis 25: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 33, analysis 21]; Test type: Superiority; p = 0.3733, ANCOVA; LS Mean Difference = -1.42, 95% CI 2-sided [-4.55 to 1.71], Standard Error of Mean 1.59
Statistical Analysis 26: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Change at Week 56: Percent Activity Impairment: ANCOVA model included treatment as fixed effects, baseline WPAI score and baseline diary average pain as covariates, and study site as a random effect; Test type: Superiority; p = 0.8056, ANCOVA; LS Mean Difference = -0.53, 95% CI 2-sided [-4.80 to 3.73], Standard Error of Mean 2.17
Statistical Analysis 27: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 33, analysis 26]; Test type: Superiority; p = 0.5764, ANCOVA; LS Mean Difference = -1.16, 95% CI 2-sided [-5.25 to 2.93], Standard Error of Mean 2.08

34. Secondary Outcome: Number of Participants Who Withdrew Due to Lack of Efficacy
Description: Number of participants who withdrew from treatment due to lack of efficacy have been reported here.
Time Frame: Baseline up to Week 56
Population: ITT population included all randomized participants who received at least one dose of SC study medication (either tanezumab or matching placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Followed by Tanezumab 5 mg | Placebo Followed by Tanezumab 10 mg | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 202 | 204 | 407 | 407 | 605
Participants | 25 | 41 | 41 | 46 | 65
Statistical Analysis 1: Comparison: Pooled Tanezumab 5 mg vs Tramadol; OR and 95% CI estimated from logistic regression model. Logistic regression model included baseline average LBPI and treatment; Test type: Superiority; p = 0.7366, Regression, Logistic; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.62 to 1.41]
Statistical Analysis 2: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 34, analysis 1]; Test type: Superiority; p = 0.7710, Regression, Logistic; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.71 to 1.58]

35. Secondary Outcome: Time to Discontinuation Due to Lack of Efficacy
Description: Time to discontinuation due to lack of efficacy was defined as the time interval from the date of first study drug administration up to the date of discontinuation of participant from treatment due to lack of efficacy.
Time Frame: Baseline up to Week 56
Population: as for outcome 34
Measure: Median (Full Range); unit: days
Arm/Group | Placebo Followed by Tanezumab 5 mg | Placebo Followed by Tanezumab 10 mg | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 202 | 204 | 407 | 407 | 605
days | NA [14 to 123] — Due to the Kaplan-Meier estimate not reaching the level for discontinuation due to insufficient clinical response, lack of efficacy, median could not be calculated. | NA [8 to 122] — Due to the Kaplan-Meier estimate not reaching the level for discontinuation due to insufficient clinical response, lack of efficacy, median could not be calculated. | NA [14 to 252] — Due to the Kaplan-Meier estimate not reaching the level for discontinuation due to insufficient clinical response, lack of efficacy, median could not be calculated. | NA [2 to 175] — Due to the Kaplan-Meier estimate not reaching the level for discontinuation due to insufficient clinical response, lack of efficacy, median could not be calculated. | NA [2 to 314] — Due to the Kaplan-Meier estimate not reaching the level for discontinuation due to insufficient clinical response, lack of efficacy, median could not be calculated.
Statistical Analysis 1: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Missing data for the selected percentile(s) was due to the Kaplan-Meier estimate not reaching the level for discontinuation due to lack of efficacy; Test type: Superiority; p = 0.4724, Log Rank
Statistical Analysis 2: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 35, analysis 1]; Test type: Superiority; p = 0.7142, Log Rank

36. Secondary Outcome: Number of Participants Who Took Rescue Medication During Weeks 2, 4, 8, 12, 16, 24, 32, 40, 48, 56 and 64
Description: In case of inadequate pain relief, acetaminophen/paracetamol caplets, tablets, or capsules up to 3000 mg per day up to 3 days in a week could be taken as rescue medication between day 1 and week 56. Number of participants with any use of rescue medication during the particular study week were summarized. As pre specified intent of study, for analyses after week 16 where multiple imputation was used, data was reported per 3 arms. This is because participants who received placebo from Day 1 and received tanezumab 5/10 mg at week 16, received placebo for the first 16 weeks, and their data before week 16 were not be imputed into analyses after week 16.
Time Frame: Weeks 2, 4, 8, 12, 16, 24, 32, 40, 48, 56 and 64
Population: ITT population included all randomized participants who received at least one dose of SC study medication (either tanezumab or matching placebo). Here,"N"=participants evaluable for this OM and "n" participants evaluable for OM at specified time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 407 | 407 | 604
Participants
  Week 2: number analyzed (Participants) | 406 | 406 | 602
  Week 2 | 226 | 208 | 318
  Week 4 | 205 | 175 | 285
  Week 8 | 176 | 158 | 250
  Week 12 | 150 | 147 | 216
  Week 16 | 134 | 125 | 193
  Week 24 | 145 | 150 | 211
  Week 32 | 146 | 152 | 210
  Week 40 | 145 | 144 | 209
  Week 48 | 141 | 144 | 210
  Week 56 | 142 | 142 | 215
Statistical Analysis 1: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 2: Odds ratio and 95% CI estimated from logistic regression model. Logistic regression model included baseline LBPI and treatment; Test type: Superiority; p = 0.3960, Regression, Logistic; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.87 to 1.44]
Statistical Analysis 2: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 36, analysis 1]; Test type: Superiority; p = 0.5932, Regression, Logistic; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.73 to 1.20]
Statistical Analysis 3: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 4: Odds ratio and 95% CI estimated from logistic regression model. Logistic regression model included baseline LBPI and treatment; Test type: Superiority; p = 0.3326, Regression, Logistic; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.88 to 1.46]
Statistical Analysis 4: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 36, analysis 3]; Test type: Superiority; p = 0.1765, Regression, Logistic; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.65 to 1.08]
Statistical Analysis 5: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 8: Odds ratio and 95% CI estimated from logistic regression model. Logistic regression model included baseline LBPI and treatment; Test type: Superiority; p = 0.5619, Regression, Logistic; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.84 to 1.39]
Statistical Analysis 6: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 36, analysis 5]; Test type: Superiority; p = 0.3909, Regression, Logistic; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.69 to 1.16]
Statistical Analysis 7: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 12: Odds ratio and 95% CI estimated from logistic regression model. Logistic regression model included baseline LBPI and treatment; Test type: Superiority; p = 0.7562, Regression, Logistic; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.80 to 1.35]
Statistical Analysis 8: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 36, analysis 7]; Test type: Superiority; p = 0.9476, Regression, Logistic; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.78 to 1.31]
Statistical Analysis 9: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 16: Odds ratio and 95% CI estimated from logistic regression model. Logistic regression model included baseline LBPI and treatment; Test type: Superiority; p = 0.7746, Regression, Logistic; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.79 to 1.36]
Statistical Analysis 10: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 36, analysis 9]; Test type: Superiority; p = 0.6377, Regression, Logistic; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.71 to 1.23]
Statistical Analysis 11: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 24: Odds ratio and 95% CI estimated from logistic regression model. Logistic regression model included baseline LBPI and treatment; Test type: Superiority; p = 0.8532, Regression, Logistic; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.79 to 1.33]
Statistical Analysis 12: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 36, analysis 11]; Test type: Superiority; p = 0.5644, Regression, Logistic; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.83 to 1.40]
Statistical Analysis 13: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 32: Odds ratio and 95% CI estimated from logistic regression model. Logistic regression model included baseline LBPI and treatment; Test type: Superiority; p = 0.7690, Regression, Logistic; Odds Ratio (OR) = 1.04, 0.7690% CI 2-sided [0.80 to 1.35]
Statistical Analysis 14: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 36, analysis 13]; Test type: Superiority; p = 0.4321, Regression, Logistic; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.85 to 1.44]
Statistical Analysis 15: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 40: Odds ratio and 95% CI estimated from logistic regression model. Logistic regression model included baseline LBPI and treatment; Test type: Superiority; p = 0.7714, Regression, Logistic; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.80 to 1.35]
Statistical Analysis 16: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 36, analysis 15]; Test type: Superiority; p = 0.8389, Regression, Logistic; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.79 to 1.34]
Statistical Analysis 17: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 48: Odds ratio and 95% CI estimated from logistic regression model. Logistic regression model included baseline LBPI and treatment; Test type: Superiority; p = 0.9383, Regression, Logistic; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.76 to 1.29]
Statistical Analysis 18: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 36, analysis 17]; Test type: Superiority; p = 0.8800, Regression, Logistic; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.78 to 1.33]
Statistical Analysis 19: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 56: Odds ratio and 95% CI estimated from logistic regression model. Logistic regression model included baseline LBPI and treatment; Test type: Superiority; p = 0.7946, Regression, Logistic; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.74 to 1.26]
Statistical Analysis 20: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 36, analysis 19]; Test type: Superiority; p = 0.7803, Regression, Logistic; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.74 to 1.25]

37. Secondary Outcome: Number of Participants Who Took Rescue Medication During Week 64: Observed Data
Description: In case of inadequate pain relief, after Week 24, acetaminophen/paracetamol up to 4000 mg per day up to 5 days in a week could be taken as rescue medication and use was reported weekly via diary. Number of participants with any use of rescue medication during the 4 weeks up to and including the particular study week were summarized.
Time Frame: Week 64
Population: ITT population included all randomized participants who received at least one dose of SC study medication (either tanezumab or matching placebo). Here, 'Overall number of participants analyzed' signifies participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Followed by Tanezumab 5 mg | Placebo Followed by Tanezumab 10 mg | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 61 | 60 | 136 | 151 | 193
Participants | 35 | 26 | 59 | 70 | 99

38. Secondary Outcome: Number of Days of Rescue Medication Used at Weeks 2, 4, 8, 12, 16, 24, 32, 40, 48 and 56
Description: In case of inadequate pain relief, acetaminophen/paracetamol caplets, tablets, or capsules up to 3000 mg per day up to 3 days in a week could be taken as rescue medication between day 1 and week 56. Number of days the participants used the rescue medication during the particular study weeks were summarized. As pre specified intent of study, for analyses after week 16 where multiple imputation was used, data was reported per 3 arms. This is because participants who received placebo from Day 1 and received tanezumab 5/10 mg at week 16, received placebo for the first 16 weeks, and their data before week 16 were not be imputed into analyses after week 16.
Time Frame: Weeks 2, 4, 8, 12, 16, 24, 32, 40, 48 and 56
Population: as for outcome 37
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 407 | 407 | 605
days
  Week 2 | 2.05 (0.15) | 1.85 (0.14) | 1.76 (0.11)
  Week 4 | 1.62 (0.13) | 1.40 (0.12) | 1.46 (0.10)
  Week 8 | 1.40 (0.13) | 1.15 (0.11) | 1.23 (0.09)
  Week 12 | 1.25 (0.13) | 1.02 (0.11) | 1.11 (0.09)
  Week 16 | 1.18 (0.13) | 0.96 (0.11) | 0.99 (0.09)
  Week 24 | 1.36 (0.15) | 1.35 (0.14) | 1.32 (0.12)
  Week 32 | 1.35 (0.15) | 1.36 (0.15) | 1.38 (0.12)
  Week 40 | 1.39 (0.15) | 1.24 (0.14) | 1.37 (0.12)
  Week 48 | 1.32 (0.14) | 1.25 (0.14) | 1.37 (0.12)
  Week 56 | 1.32 (0.14) | 1.22 (0.13) | 1.42 (0.12)
Statistical Analysis 1: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 2: Analysis was performed using negative binomial model with model terms of Baseline average LBPI and treatment group; Test type: Superiority; p = 0.1272, Negative binomial model; LS Mean Ratio = 1.16, 95% CI 2-sided [0.96 to 1.41], Standard Error of Mean 0.11
Statistical Analysis 2: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 38, analysis 1]; Test type: Superiority; p = 0.6322, Negative binomial model; LS Mean Ratio = 1.05, 95% CI 2-sided [0.86 to 1.27], Standard Error of Mean 0.10
Statistical Analysis 3: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 4: Analysis was performed using negative binomial model with model terms of Baseline average LBPI and treatment group; Test type: Superiority; p = 0.3559, Negative binomial model; LS Mean Ratio = 1.10, 95% CI 2-sided [0.89 to 1.36], Standard Error of Mean 0.12
Statistical Analysis 4: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 38, analysis 3]; Test type: Superiority; p = 0.6798, Negative binomial model; LS Mean Ratio = 0.96, 95% CI 2-sided [0.77 to 1.18]
Statistical Analysis 5: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 8: Analysis was performed using negative binomial model with model terms of Baseline average LBPI and treatment group; Test type: Superiority; p = 0.2670, Negative binomial model; LS Mean Ratio = 1.14, 95% CI 2-sided [0.90 to 1.44]
Statistical Analysis 6: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 38, analysis 5]; Test type: Superiority; p = 0.5865, Negative binomial model; LS Mean Ratio = 0.94, 95% CI 2-sided [0.74 to 1.19]
Statistical Analysis 7: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 12: Analysis was performed using negative binomial model with model terms of Baseline average LBPI and treatment group; Test type: Superiority; p = 0.3378, Negative binomial model; LS Mean Ratio = 1.13, 95% CI 2-sided [0.88 to 1.47]
Statistical Analysis 8: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 38, analysis 7]; Test type: Superiority; p = 0.5510, Negative binomial model; LS Mean Ratio = 0.92, 95% CI 2-sided [0.71 to 1.20]
Statistical Analysis 9: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 16: Analysis was performed using negative binomial model with model terms of Baseline average LBPI and treatment group; Test type: Superiority; p = 0.2088, Negative binomial model; LS Mean Ratio = 1.20, 95% CI 2-sided [0.90 to 1.60], Standard Error of Mean 0.18
Statistical Analysis 10: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 38, analysis 9]; Test type: Superiority; p = 0.8692, Negative binomial model; LS Mean Ratio = 0.98, 95% CI 2-sided [0.73 to 1.30], Standard Error of Mean 0.14
Statistical Analysis 11: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 24: Analysis was performed using negative binomial model with model terms of Baseline average LBPI and treatment group; Test type: Superiority; p = 0.8444, Negative binomial model; LS Mean Ratio = 1.03, 95% CI 2-sided [0.78 to 1.35], Standard Error of Mean 0.14
Statistical Analysis 12: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 38, analysis 11]; Test type: Superiority; p = 0.8936, Negative binomial model; LS Mean Ratio = 1.02, 95% CI 2-sided [0.78 to 1.34], Standard Error of Mean 0.14
Statistical Analysis 13: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 32: Analysis was performed using negative binomial model with model terms of Baseline average LBPI and treatment group; Test type: Superiority; p = 0.8716, Negative binomial model; LS Mean Ratio = 0.98, 95% CI 2-sided [0.75 to 1.28], Standard Error of Mean 0.14
Statistical Analysis 14: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 38, analysis 13]; Test type: Superiority; p = 0.8827, Negative binomial model; LS Mean Ratio = 0.98, 95% CI 2-sided [0.75 to 1.29], Standard Error of Mean 0.14
Statistical Analysis 15: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 40: Analysis was performed using negative binomial model with model terms of Baseline average LBPI and treatment group; Test type: Superiority; p = 0.8996, Negative binomial model; LS Mean Ratio = 1.02, 95% CI 2-sided [0.77 to 1.34], Standard Error of Mean 0.14
Statistical Analysis 16: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 38, analysis 15]; Test type: Superiority; p = 0.4880, Negative binomial model; LS Mean Ratio = 0.91, 95% CI 2-sided [0.69 to 1.20], Standard Error of Mean 0.13
Statistical Analysis 17: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 48: Analysis was performed using negative binomial model with model terms of Baseline average LBPI and treatment group; Test type: Superiority; p = 0.7938, Negative binomial model; LS Mean Ratio = 0.96, 95% CI 2-sided [0.73 to 1.27], Standard Error of Mean 0.14
Statistical Analysis 18: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 38, analysis 17]; Test type: Superiority; p = 0.5092, Negative binomial model; LS Mean Ratio = 0.91, 95% CI 2-sided [0.69 to 1.20], Standard Error of Mean 0.13
Statistical Analysis 19: Comparison: Pooled Tanezumab 5 mg vs Tramadol; Week 56: Analysis was performed using negative binomial model with model terms of Baseline average LBPI and treatment group; Test type: Superiority; p = 0.6148, Negative binomial model; LS Mean Ratio = 0.93, 95% CI 2-sided [0.71 to 1.22], Standard Error of Mean 0.13
Statistical Analysis 20: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 38, analysis 19]; Test type: Superiority; p = 0.2844, Negative binomial model; LS Mean Ratio = 0.86, 95% CI 2-sided [0.66 to 1.13], Standard Error of Mean 0.12

39. Secondary Outcome: Number of Days of Rescue Medication Used at Week 64
Description: In case of inadequate pain relief, acetaminophen/paracetamol caplets, tablets, or capsules up to 3000 mg per day up to 3 days in a week could be taken as rescue medication between day 1 and week 56. Number of days per week the participants used the rescue medication during the 4 weeks up to and including the particular study week were summarized.
Time Frame: Week 64
Population: ITT population included all randomized participants who received at least one dose of SC study medication (either tanezumab or matching placebo). Here, 'Overall number of participants analyzed' signifies participants who took rescue medication.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo Followed by Tanezumab 5 mg | Placebo Followed by Tanezumab 10 mg | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 61 | 60 | 136 | 151 | 193
days | 1.3 (1.59) | 1.3 (2.02) | 1.3 (1.99) | 1.4 (2.16) | 1.8 (2.44)

40. Secondary Outcome: Amount of Rescue Medication Used at Weeks 2, 4, 8, 12 and 16
Description: In case of inadequate pain relief, acetaminophen/paracetamol caplets, tablets, or capsules up to 3000 mg per day up to 3 days in a week could be taken as rescue medication between day 1 and week 56. The total dosage of acetaminophen in milligrams used during the specified week were summarized. Pre-specified intent of study for efficacy data up to W16 was to analyze participants who received placebo from Day1 and then received tanezumab 5/10 mg at W16,together,in placebo arm.Data has been reported per four arms.
Time Frame: Weeks 2, 4, 8, 12 and 16
Population: as for outcome 34
Measure: Least Squares Mean (Standard Error); unit: milligrams
Groups:
- Tanezumab 5 mg: Tanezumab (RN624 or PF-04383119) 5 mg injection administered SC once every 8 weeks from Day 1 and placebo tablets matched to tramadol PR, orally, once daily from Day 1 up to week 16.
- Tanezumab 10 mg: Tanezumab (RN624 or PF-04383119) 10 mg injection administered SC once every 8 weeks from Day 1, and placebo tablets matched to tramadol PR, orally, once daily from Day 1 up to week 16.
Arm/Group | Placebo | Tanezumab 5 mg | Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 406 | 407 | 407 | 605
milligrams
  Week 2 | 2420.1 (392.67) | 2663.2 (431.26) | 2465.7 (398.76) | 2340.4 (310.28)
  Week 4 | 2084.6 (374.33) | 1967.2 (352.25) | 1847.9 (330.64) | 1852.2 (271.70)
  Week 8 | 1757.9 (354.02) | 1682.3 (338.34) | 1612.5 (323.86) | 1512.4 (248.85)
  Week 12 | 1707.2 (379.30) | 1491.6 (330.87) | 1345.3 (297.82) | 1464.2 (265.85)
  Week 16 | 1385.0 (340.93) | 1537.8 (377.76) | 1359.0 (333.62) | 1296.8 (260.75)
Statistical Analysis 1: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 38, analysis 1]; Test type: Superiority; p = 0.6764, Negative binomial model; LS Mean Ratio = 1.10, 95% CI 2-sided [0.70 to 1.73], Standard Error of Mean 0.25
Statistical Analysis 2: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 38, analysis 1]; Test type: Superiority; p = 0.9351, Negative binomial model; LS Mean Ratio = 1.02, 95% CI 2-sided [0.65 to 1.60], Standard Error of Mean 0.23
Statistical Analysis 3: Comparison: Placebo vs Tramadol; [analysis description as in outcome 38, analysis 1]; Test type: Superiority; p = 0.8731, Negative binomial model; LS Mean Ratio = 0.97, 95% CI 2-sided [0.64 to 1.46], Standard Error of Mean 0.20
Statistical Analysis 4: Comparison: Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 38, analysis 1]; Test type: Superiority; p = 0.5370, Negative binomial model; LS Mean Ratio = 1.14, 95% CI 2-sided [0.75 to 1.72], Standard Error of Mean 0.24
Statistical Analysis 5: Comparison: Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 38, analysis 1]; Test type: Superiority; p = 0.8031, Negative binomial model; LS Mean Ratio = 1.05, 95% CI 2-sided [0.70 to 1.59], Standard Error of Mean 0.22
Statistical Analysis 6: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 38, analysis 3]; Test type: Superiority; p = 0.8192, Negative binomial model; LS Mean Ratio = 0.94, 95% CI 2-sided [0.57 to 1.55], Standard Error of Mean 0.24
Statistical Analysis 7: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 38, analysis 3]; Test type: Superiority; p = 0.6345, Negative binomial model; LS Mean Ratio = 0.89, 95% CI 2-sided [0.54 to 1.46], Standard Error of Mean 0.22
Statistical Analysis 8: Comparison: Placebo vs Tramadol; [analysis description as in outcome 38, analysis 3]; Test type: Superiority; p = 0.6103, Negative binomial model; LS Mean Ratio = 0.89, 95% CI 2-sided [0.56 to 1.40], Standard Error of Mean 0.21
Statistical Analysis 9: Comparison: Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 38, analysis 3]; Test type: Superiority; p = 0.7949, Negative binomial model; LS Mean Ratio = 1.06, 95% CI 2-sided [0.67 to 1.67], Standard Error of Mean 0.25
Statistical Analysis 10: Comparison: Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 38, analysis 3]; Test type: Superiority; p = 0.9920, Negative binomial model; LS Mean Ratio = 1.00, 95% CI 2-sided [0.63 to 1.57], Standard Error of Mean 0.23
Statistical Analysis 11: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 38, analysis 5]; Test type: Superiority; p = 0.8772, Negative binomial model; LS Mean Ratio = 0.96, 95% CI 2-sided [0.55 to 1.67], Standard Error of Mean 0.27
Statistical Analysis 12: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 38, analysis 5]; Test type: Superiority; p = 0.7614, Negative binomial model; LS Mean Ratio = 0.92, 95% CI 2-sided [0.53 to 1.60], Standard Error of Mean 0.26
Statistical Analysis 13: Comparison: Placebo vs Tramadol; [analysis description as in outcome 38, analysis 5]; Test type: Superiority; p = 0.5629, Negative binomial model; LS Mean Ratio = 0.86, 95% CI 2-sided [0.52 to 1.43], Standard Error of Mean 0.22
Statistical Analysis 14: Comparison: Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 38, analysis 5]; Test type: Superiority; p = 0.6821, Negative binomial model; LS Mean Ratio = 1.11, 95% CI 2-sided [0.67 to 1.85], Standard Error of Mean 0.29
Statistical Analysis 15: Comparison: Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 38, analysis 5]; Test type: Superiority; p = 0.8049, Negative binomial model; LS Mean Ratio = 1.07, 95% CI 2-sided [0.64 to 1.77], Standard Error of Mean 0.28
Statistical Analysis 16: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 38, analysis 7]; Test type: Superiority; p = 0.6673, Negative binomial model; LS Mean Ratio = 0.87, 95% CI 2-sided [0.47 to 1.62], Standard Error of Mean 0.27
Statistical Analysis 17: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 38, analysis 7]; Test type: Superiority; p = 0.4475, Negative binomial model; LS Mean Ratio = 0.79, 95% CI 2-sided [0.43 to 1.46], Standard Error of Mean 0.25
Statistical Analysis 18: Comparison: Placebo vs Tramadol; [analysis description as in outcome 38, analysis 7]; Test type: Superiority; p = 0.5925, Negative binomial model; LS Mean Ratio = 0.86, 95% CI 2-sided [0.49 to 1.50], Standard Error of Mean 0.25
Statistical Analysis 19: Comparison: Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 38, analysis 7]; Test type: Superiority; p = 0.9486, Negative binomial model; LS Mean Ratio = 1.02, 95% CI 2-sided [0.58 to 1.79], Standard Error of Mean 0.29
Statistical Analysis 20: Comparison: Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 38, analysis 7]; Test type: Superiority; p = 0.7673, Negative binomial model; LS Mean Ratio = 0.92, 95% CI 2-sided [0.52 to 1.61], Standard Error of Mean 0.26
Statistical Analysis 21: Comparison: Placebo vs Tanezumab 5 mg; [analysis description as in outcome 38, analysis 9]; Test type: Superiority; p = 0.7635, Negative binomial model; LS Mean Ratio = 1.11, 95% CI 2-sided [0.56 to 2.20], Standard Error of Mean 0.39
Statistical Analysis 22: Comparison: Placebo vs Tanezumab 10 mg; [analysis description as in outcome 38, analysis 9]; Test type: Superiority; p = 0.9564, Negative binomial model; LS Mean Ratio = 0.98, 95% CI 2-sided [0.50 to 1.94], Standard Error of Mean 0.34
Statistical Analysis 23: Comparison: Placebo vs Tramadol; [analysis description as in outcome 38, analysis 9]; Test type: Superiority; p = 0.8359, Negative binomial model; LS Mean Ratio = 0.94, 95% CI 2-sided [0.50 to 1.75], Standard Error of Mean 0.30
Statistical Analysis 24: Comparison: Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 38, analysis 9]; Test type: Superiority; p = 0.5914, Negative binomial model; LS Mean Ratio = 1.19, 95% CI 2-sided [0.64 to 2.21], Standard Error of Mean 0.38
Statistical Analysis 25: Comparison: Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 38, analysis 9]; Test type: Superiority; p = 0.8826, Negative binomial model; LS Mean Ratio = 1.05, 95% CI 2-sided [0.56 to 1.95], Standard Error of Mean 0.33

41. Secondary Outcome: Health Care Resource Utilization (HCRU): Number of Visits of Services Received Directly Related to Low Back Pain
Description: Low back pain HCRU assessed utilization of healthcare resources usage during last 3 months (for Baseline during the last 3 months for baseline, weeks 64 and 80, via IRT). Visits of services directly related to low back pain evaluated were: visits to primary care physician, neurologist, rheumatologist, physician assistant or nurse practitioner, pain specialist, orthopedist, physical therapist, chiropractor, alternative medicine or therapy, podiatrist, nutritionist/dietitian, radiologist, home healthcare services and other practitioner. Participants might have been counted more than once under various categories.
Time Frame: Baseline, Weeks 64 and 80
Population: as for outcome 30
Measure: Median (Full Range); unit: visits
Arm/Group | Placebo Followed by Tanezumab 5 mg | Placebo Followed by Tanezumab 10 mg | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 202 | 204 | 407 | 407 | 605
visits
  Baseline: Primary Care Physician: number analyzed (Participants) | 88 | 95 | 190 | 194 | 276
  Baseline: Primary Care Physician | 1.0 [1.0 to 8.0] | 2.0 [1.0 to 114.0] | 2.0 [1.0 to 111.0] | 2.0 [1.0 to 14.0] | 2.0 [1.0 to 562.0]
  Baseline: Neurologist: number analyzed (Participants) | 5 | 5 | 8 | 20 | 20
  Baseline: Neurologist | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 3.0] | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 6.0] | 1.0 [1.0 to 4.0]
  Baseline: Rheumatologist: number analyzed (Participants) | 6 | 8 | 17 | 24 | 27
  Baseline: Rheumatologist | 2.0 [1.0 to 2.0] | 1.0 [1.0 to 3.0] | 2.0 [1.0 to 5.0] | 1.0 [1.0 to 3.0] | 1.0 [1.0 to 6.0]
  Baseline:Physician assistant or nurse Practitioner: number analyzed (Participants) | 14 | 17 | 13 | 17 | 37
  Baseline:Physician assistant or nurse Practitioner | 1.0 [1.0 to 6.0] | 2.0 [1.0 to 10.0] | 1.0 [1.0 to 5.0] | 1.0 [1.0 to 6.0] | 1.0 [1.0 to 6.0]
  Baseline: Pain specialist: number analyzed (Participants) | 30 | 28 | 53 | 61 | 60
  Baseline: Pain specialist | 2.0 [1.0 to 22.0] | 2.0 [1.0 to 25.0] | 2.0 [1.0 to 30.0] | 2.0 [1.0 to 222.0] | 2.0 [1.0 to 11.0]
  Baseline: Orthopedist: number analyzed (Participants) | 18 | 31 | 40 | 36 | 63
  Baseline: Orthopedist | 3.0 [1.0 to 8.0] | 3.0 [1.0 to 36.0] | 3.0 [1.0 to 15.0] | 2.0 [1.0 to 12.0] | 3.0 [1.0 to 16.0]
  Baseline: Physical therapist: number analyzed (Participants) | 18 | 19 | 28 | 38 | 48
  Baseline: Physical therapist | 6.5 [1.0 to 24.0] | 8.0 [1.0 to 36.0] | 4.5 [1.0 to 20.0] | 5.5 [1.0 to 111.0] | 3.5 [1.0 to 90.0]
  Baseline: Chiropractor: number analyzed (Participants) | 19 | 23 | 38 | 47 | 76
  Baseline: Chiropractor | 3.0 [1.0 to 10.0] | 3.0 [1.0 to 36.0] | 3.5 [1.0 to 30.0] | 3.0 [1.0 to 24.0] | 3.0 [1.0 to 121.0]
  Baseline: Alternative medicine or therapy: number analyzed (Participants) | 15 | 20 | 23 | 29 | 50
  Baseline: Alternative medicine or therapy | 2.0 [1.0 to 10.0] | 2.0 [1.0 to 121.0] | 3.0 [1.0 to 111.0] | 2.0 [1.0 to 45.0] | 2.0 [1.0 to 211.0]
  Baseline: Podiatrist: number analyzed (Participants) | 2 | 0 | 4 | 5 | 5
  Baseline: Podiatrist | 2.0 [1.0 to 3.0] |  | 2.0 [1.0 to 3.0] | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 1.0]
  Baseline: Nutritionist/dietitian: number analyzed (Participants) | 0 | 6 | 6 | 6 | 3
  Baseline: Nutritionist/dietitian |  | 3.0 [1.0 to 100.0] | 1.5 [1.0 to 6.0] | 2.0 [1.0 to 4.0] | 1.0 [1.0 to 1.0]
  Baseline: Radiologist: number analyzed (Participants) | 12 | 14 | 18 | 30 | 35
  Baseline: Radiologist | 1.0 [1.0 to 3.0] | 1.5 [1.0 to 3.0] | 1.0 [1.0 to 6.0] | 1.0 [1.0 to 10.0] | 1.0 [1.0 to 4.0]
  Baseline: Home healthcare services: number analyzed (Participants) | 2 | 2 | 0 | 3 | 4
  Baseline: Home healthcare services | 7.5 [3.0 to 12.0] | 6.0 [1.0 to 11.0] |  | 1.0 [1.0 to 3.0] | 6.5 [1.0 to 36.0]
  Baseline: Other practitioner: number analyzed (Participants) | 22 | 27 | 37 | 48 | 68
  Baseline: Other practitioner | 1.0 [1.0 to 6.0] | 2.0 [1.0 to 90.0] | 1.0 [1.0 to 8.0] | 2.0 [1.0 to 111.0] | 1.0 [1.0 to 36.0]
  Week 64: Primary Care Physician: number analyzed (Participants) | 33 | 36 | 76 | 82 | 106
  Week 64: Primary Care Physician | 1.0 [1.0 to 5.0] | 1.0 [1.0 to 299.0] | 1.0 [1.0 to 211.0] | 1.0 [1.0 to 201.0] | 1.0 [1.0 to 200.0]
  Week 64: Neurologist: number analyzed (Participants) | 5 | 4 | 6 | 4 | 6
  Week 64: Neurologist | 1.0 [1.0 to 18.0] | 1.5 [1.0 to 3.0] | 1.0 [1.0 to 4.0] | 1.5 [1.0 to 3.0] | 1.0 [1.0 to 101.0]
  Week 64: Rheumatologist: number analyzed (Participants) | 3 | 5 | 11 | 13 | 10
  Week 64: Rheumatologist | 2.0 [1.0 to 14.0] | 1.0 [1.0 to 27.0] | 1.0 [1.0 to 100.0] | 1.0 [1.0 to 101.0] | 1.0 [1.0 to 2.0]
  Week 64: Physician assistant or nurse Practitioner: number analyzed (Participants) | 9 | 7 | 11 | 10 | 11
  Week 64: Physician assistant or nurse Practitioner | 1.0 [1.0 to 201.0] | 1.0 [1.0 to 8.0] | 2.0 [1.0 to 6.0] | 1.0 [1.0 to 3.0] | 1.0 [1.0 to 3.0]
  Week 64: Pain specialist: number analyzed (Participants) | 11 | 18 | 24 | 22 | 32
  Week 64: Pain specialist | 1.0 [1.0 to 16.0] | 2.0 [1.0 to 100.0] | 2.0 [1.0 to 10.0] | 1.0 [1.0 to 201.0] | 1.0 [1.0 to 4.0]
  Week 64: Orthopedist: number analyzed (Participants) | 7 | 22 | 31 | 24 | 39
  Week 64: Orthopedist | 2.0 [1.0 to 9.0] | 1.5 [1.0 to 27.0] | 1.0 [1.0 to 6.0] | 1.0 [1.0 to 201.0] | 2.0 [1.0 to 100.0]
  Week 64: Physical therapist: number analyzed (Participants) | 9 | 11 | 14 | 21 | 22
  Week 64: Physical therapist | 10.0 [1.0 to 18.0] | 8.0 [1.0 to 36.0] | 4.5 [1.0 to 20.0] | 4.0 [1.0 to 30.0] | 3.0 [1.0 to 999.0]
  Week 64: Chiropractor: number analyzed (Participants) | 12 | 10 | 25 | 24 | 38
  Week 64: Chiropractor | 6.0 [1.0 to 36.0] | 2.5 [1.0 to 100.0] | 2.0 [1.0 to 25.0] | 3.5 [1.0 to 92.0] | 2.0 [1.0 to 999.0]
  Week 64: Alternative medicine or therapy: number analyzed (Participants) | 6 | 12 | 14 | 15 | 27
  Week 64: Alternative medicine or therapy | 6.0 [1.0 to 300.0] | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 24.0] | 1.0 [1.0 to 5.0] | 1.0 [1.0 to 111.0]
  Week 64: Podiatrist: number analyzed (Participants) | 2 | 2 | 5 | 5 | 4
  Week 64: Podiatrist | 1.5 [1.0 to 2.0] | 2.0 [1.0 to 3.0] | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 1.0]
  Week 64: Nutritionist/dietitian: number analyzed (Participants) | 0 | 4 | 3 | 2 | 6
  Week 64: Nutritionist/dietitian |  | 1.0 [1.0 to 100.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 9.0]
  Week 64: Radiologist: number analyzed (Participants) | 5 | 6 | 9 | 9 | 16
  Week 64: Radiologist | 1.0 [1.0 to 3.0] | 1.5 [1.0 to 3.0] | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 2.0]
  Week 64: Home healthcare services: number analyzed (Participants) | 1 | 2 | 1 | 3 | 6
  Week 64: Home healthcare services | 8.0 [8.0 to 8.0] | 3.0 [1.0 to 5.0] | 1.0 [1.0 to 1.0] | 2.0 [1.0 to 3.0] | 16.5 [1.0 to 401.0]
  Week 64: Other practitioner: number analyzed (Participants) | 14 | 16 | 29 | 30 | 34
  Week 64: Other practitioner | 1.0 [1.0 to 18.0] | 2.0 [1.0 to 100.0] | 1.0 [1.0 to 111.0] | 1.0 [1.0 to 16.0] | 1.0 [1.0 to 6.0]
  Week 80: Primary Care Physician: number analyzed (Participants) | 15 | 16 | 31 | 37 | 41
  Week 80: Primary Care Physician | 2.0 [1.0 to 3.0] | 1.0 [1.0 to 36.0] | 1.0 [1.0 to 101.0] | 1.0 [1.0 to 4.0] | 1.0 [1.0 to 12.0]
  Week 80: Neurologist: number analyzed (Participants) | 1 | 1 | 2 | 1 | 3
  Week 80: Neurologist | 1.0 [1.0 to 1.0] | 2.0 [2.0 to 2.0] | 2.5 [2.0 to 3.0] | 2.0 [2.0 to 2.0] | 2.0 [1.0 to 3.0]
  Week 80: Rheumatologist: number analyzed (Participants) | 1 | 3 | 3 | 2 | 4
  Week 80: Rheumatologist | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  Week 80: Physician assistant or nurse Practitioner: number analyzed (Participants) | 2 | 2 | 5 | 5 | 1
  Week 80: Physician assistant or nurse Practitioner | 5.0 [1.0 to 9.0] | 50.5 [1.0 to 100.0] | 1.0 [1.0 to 3.0] | 1.0 [1.0 to 1.0] | 2.0 [2.0 to 2.0]
  Week 80: Pain specialist: number analyzed (Participants) | 5 | 5 | 6 | 12 | 7
  Week 80: Pain specialist | 2.0 [1.0 to 2.0] | 1.0 [1.0 to 11.0] | 2.5 [1.0 to 4.0] | 1.0 [1.0 to 3.0] | 1.0 [1.0 to 3.0]
  Week 80: Orthopedist: number analyzed (Participants) | 3 | 7 | 8 | 6 | 16
  Week 80: Orthopedist | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 6.0] | 1.0 [1.0 to 3.0] | 1.5 [1.0 to 2.0] | 1.5 [1.0 to 7.0]
  Week 80: Physical therapist: number analyzed (Participants) | 4 | 5 | 8 | 11 | 4
  Week 80: Physical therapist | 5.0 [1.0 to 8.0] | 12.0 [1.0 to 20.0] | 4.0 [1.0 to 16.0] | 5.0 [1.0 to 20.0] | 6.0 [6.0 to 14.0]
  Week 80: Chiropractor: number analyzed (Participants) | 2 | 6 | 7 | 12 | 12
  Week 80: Chiropractor | 401.0 [1.0 to 801.0] | 3.5 [1.0 to 9.0] | 4.0 [1.0 to 10.0] | 4.0 [1.0 to 20.0] | 3.0 [1.0 to 14.0]
  Week 80: Alternative medicine or therapy: number analyzed (Participants) | 2 | 4 | 5 | 2 | 9
  Week 80: Alternative medicine or therapy | 9.0 [3.0 to 15.0] | 2.5 [1.0 to 30.0] | 3.0 [1.0 to 4.0] | 2.5 [2.0 to 3.0] | 2.0 [1.0 to 5.0]
  Week 80: Podiatrist: number analyzed (Participants) | 2 | 1 | 1 | 1 | 2
  Week 80: Podiatrist | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 1.5 [1.0 to 2.0]
  Week 80: Nutritionist/dietitian: number analyzed (Participants) | 1 | 1 | 2 | 2 | 0
  Week 80: Nutritionist/dietitian | 1.0 [1.0 to 1.0] | 10.0 [10.0 to 10.0] | 1.0 [1.0 to 1.0] | 4.0 [2.0 to 6.0] |
  Week 80: Radiologist: number analyzed (Participants) | 4 | 0 | 2 | 5 | 7
  Week 80: Radiologist | 1.0 [1.0 to 1.0] |  | 1.5 [1.0 to 2.0] | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 1.0]
  Week 80: Home healthcare services: number analyzed (Participants) | 1 | 0 | 1 | 0 | 2
  Week 80: Home healthcare services | 1.0 [1.0 to 1.0] |  | 4.0 [4.0 to 4.0] |  | 24.5 [13.0 to 36.0]
  Week 80: Other practitioner: number analyzed (Participants) | 3 | 5 | 4 | 6 | 14
  Week 80: Other practitioner | 1.0 [1.0 to 11.0] | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 4.0] | 1.0 [1.0 to 3.0] | 1.0 [1.0 to 10.0]

42. Secondary Outcome: Health Care Resource Utilization (HCRU): Number of Participants Who Visited the Emergency Room Due to Low Back Pain
Description: Low back pain HCRU assessed utilization of healthcare resources during the last 3 months for baseline, weeks 64 and 80, via IRT. Domain evaluated was number of participants who visited the emergency room due to low back pain.
Time Frame: Baseline, Weeks 64 and 80
Population: ITT population included all randomized participants who received at least one dose of SC study medication (either tanezumab or matching placebo). Here, 'n' signifies the number of participants who had visited the emergency room at specified time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Followed by Tanezumab 5 mg | Placebo Followed by Tanezumab 10 mg | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 202 | 204 | 407 | 407 | 605
Participants
  Baseline | 10 | 14 | 27 | 17 | 26
  Week 64: number analyzed (Participants) | 135 | 138 | 285 | 285 | 414
  Week 64 | 4 | 2 | 7 | 5 | 3
  Week 80: number analyzed (Participants) | 61 | 59 | 134 | 143 | 191
  Week 80 | 0 | 3 | 3 | 0 | 4

43. Secondary Outcome: Health Care Resource Utilization (HCRU): Number of Visits to the Emergency Room Due to Low Back Pain
Description: Low back pain HCRU assessed utilization of healthcare resources during the last 3 months for baseline, weeks 64 and 80, via IRT. Domain evaluated was number of visits to the emergency room due to low back pain.
Time Frame: Baseline, Weeks 64 and 80
Population: ITT population included all randomized participants who received at least one dose of SC study medication (either tanezumab or matching placebo). Not all participants of the ITT population had data collected at each of the time points for this outcome measure. Hence, "N" signifies only those participants who were evaluable for this OM.
Measure: Median (Full Range); unit: visits
Arm/Group | Placebo Followed by Tanezumab 5 mg | Placebo Followed by Tanezumab 10 mg | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 10 | 14 | 27 | 17 | 26
visits
  Baseline | 1.0 [1.0 to 3.0] | 1.0 [1.0 to 6.0] | 1.0 [1.0 to 4.0] | 1.0 [1.0 to 5.0] | 1.0 [1.0 to 7.0]
  Week 64: number analyzed (Participants) | 4 | 2 | 7 | 5 | 3
  Week 64 | 1.0 [1.0 to 1.0] | 2.0 [2.0 to 2.0] | 1.0 [1.0 to 3.0] | 1.0 [1.0 to 6.0] | 1.0 [1.0 to 2.0]
  Week 80: number analyzed (Participants) | 0 | 3 | 3 | 0 | 4
  Week 80 |  | 1.0 [1.0 to 11.0] | 1.0 [1.0 to 2.0] |  | 1.5 [1.0 to 2.0]

44. Secondary Outcome: Health Care Resource Utilization (HCRU): Number of Participants Hospitalized Due to Low Back Pain
Description: Low back pain HCRU assessed utilization of healthcare resources during the last 3 months for baseline, weeks 64 and 80, via IRT. Domain evaluated was number of participants who were hospitalized due to low back pain.
Time Frame: Baseline, Weeks 64 and 80
Population: ITT population included all randomized participants who received at least one dose of SC study medication (either tanezumab or matching placebo). Here, 'n'= Participants who were evaluable for hospitalization due to low back pain at specified time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Followed by Tanezumab 5 mg | Placebo Followed by Tanezumab 10 mg | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 202 | 204 | 407 | 407 | 605
Participants
  Baseline: number analyzed (Participants) | 202 | 204 | 406 | 407 | 605
  Baseline | 0 | 0 | 1 | 0 | 4
  Week 64: number analyzed (Participants) | 135 | 138 | 285 | 285 | 413
  Week 64 | 0 | 0 | 0 | 1 | 1
  Week 80: number analyzed (Participants) | 61 | 59 | 134 | 143 | 191
  Week 80 | 0 | 1 | 1 | 0 | 1

45. Secondary Outcome: Health Care Resource Utilization (HCRU): Number of Nights Stayed in the Hospital Due to Low Back Pain
Description: Low back pain HCRU assessed utilization of healthcare resources during the last 3 months for baseline, weeks 64 and 80, via IRT. Domain evaluated was number of nights stayed in the hospital due to low back pain.
Time Frame: Baseline, Weeks 64 and 80
Population: as for outcome 43
Measure: Median (Full Range); unit: nights
Arm/Group | Placebo Followed by Tanezumab 5 mg | Placebo Followed by Tanezumab 10 mg | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 0 | 1 | 1 | 1 | 4
nights
  Baseline: number analyzed (Participants) | 0 | 0 | 1 | 0 | 4
  Baseline |  |  | 9.0 [9.0 to 9.0] |  | 1.0 [1.0 to 2.0]
  Week 64: number analyzed (Participants) | 0 | 0 | 0 | 1 | 1
  Week 64 |  |  |  | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  Week 80: number analyzed (Participants) | 0 | 1 | 1 | 0 | 1
  Week 80 |  | 3.0 [3.0 to 3.0] | 2.0 [2.0 to 2.0] |  | 2.0 [2.0 to 2.0]

46. Secondary Outcome: Health Care Resource Utilization (HCRU): Number of Participants Who Used Any Aids/Devices for Doing Things
Description: Low back pain HCRU assessed utilization of healthcare resources during the last 3 months for baseline, weeks 64 and 80, via IRT. Domain evaluated was number of participants who used any aids/devices for doing things. Aids such as walking aid, wheelchair, device or utensil for dress/bathe/eat and any other aids/devices.
Time Frame: Baseline, Weeks 64 and 80
Population: ITT population included all randomized participants who received at least one dose of SC study medication (either tanezumab or matching placebo). Here, 'n' = Participants who were evaluable for usage of any aids/devices for doing things.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Followed by Tanezumab 5 mg | Placebo Followed by Tanezumab 10 mg | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 202 | 204 | 407 | 407 | 605
Participants
  Baseline:Walking aid use: number analyzed (Participants) | 202 | 204 | 406 | 407 | 605
  Baseline:Walking aid use: Never | 186 | 190 | 376 | 371 | 569
  Baseline:Walking aid use: Rarely | 2 | 2 | 11 | 9 | 7
  Baseline:Walking aid use: Sometimes | 6 | 4 | 12 | 16 | 15
  Baseline:Walking aid use: Often | 6 | 5 | 4 | 7 | 9
  Baseline:Walking aid use: Always | 2 | 3 | 3 | 4 | 5
  Baseline: Wheelchair use: number analyzed (Participants) | 202 | 204 | 406 | 407 | 605
  Baseline: Wheelchair use: Never | 199 | 204 | 403 | 405 | 601
  Baseline: Wheelchair use: Rarely | 1 | 0 | 3 | 0 | 1
  Baseline: Wheelchair use: Sometimes | 2 | 0 | 0 | 2 | 3
  Baseline: Wheelchair use: Often | 0 | 0 | 0 | 0 | 0
  Baseline: Wheelchair use: Always | 0 | 0 | 0 | 0 | 0
  Baseline:Device/Utensil to dress bathe eat: number analyzed (Participants) | 202 | 204 | 406 | 407 | 605
  Baseline:Device/Utensil to dress bathe eat: Never | 192 | 196 | 390 | 396 | 596
  Baseline:Device/Utensil to dress bathe eat: Rarely | 0 | 1 | 1 | 1 | 0
  Baseline:Device/Utensil to dress bathe eat: Sometimes | 4 | 3 | 6 | 4 | 4
  Baseline:Device/Utensil to dress bathe eat: Often | 5 | 1 | 6 | 3 | 4
  Baseline:Device/Utensil to dress bathe eat: Always | 1 | 3 | 3 | 3 | 1
  Baseline:Other aids or devices: number analyzed (Participants) | 202 | 204 | 406 | 407 | 605
  Baseline:Other aids or devices: Never | 188 | 188 | 387 | 382 | 550
  Baseline:Other aids or devices: Rarely | 1 | 2 | 2 | 5 | 8
  Baseline:Other aids or devices: Sometimes | 2 | 5 | 10 | 11 | 27
  Baseline:Other aids or devices: Often | 10 | 5 | 4 | 6 | 17
  Baseline:Other aids or devices: Always | 1 | 4 | 3 | 3 | 3
  Week 64: Walking aid use: number analyzed (Participants) | 135 | 138 | 285 | 285 | 414
  Week 64: Walking aid use: Never | 125 | 131 | 277 | 273 | 397
  Week 64: Walking aid use: Rarely | 2 | 4 | 1 | 3 | 3
  Week 64: Walking aid use: Sometimes | 5 | 1 | 2 | 5 | 9
  Week 64: Walking aid use: Often | 1 | 0 | 3 | 3 | 2
  Week 64: Walking aid use: Always | 2 | 2 | 2 | 1 | 3
  Week 64: Wheelchair use: number analyzed (Participants) | 135 | 138 | 285 | 285 | 414
  Week 64: Wheelchair use: Never | 135 | 138 | 283 | 283 | 412
  Week 64: Wheelchair use: Rarely | 0 | 0 | 1 | 1 | 0
  Week 64: Wheelchair use: Sometimes | 0 | 0 | 1 | 0 | 1
  Week 64: Wheelchair use: Often | 0 | 0 | 0 | 0 | 1
  Week 64: Wheelchair use: Always | 0 | 0 | 0 | 1 | 0
  Week 64: Device/Utensil to dress bathe eat: number analyzed (Participants) | 135 | 138 | 285 | 285 | 414
  Week 64: Device/Utensil to dress bathe eat: Never | 134 | 137 | 283 | 280 | 410
  Week 64: Device/Utensil to dress bathe eat: Rarely | 0 | 0 | 0 | 2 | 0
  Week 64: Device/Utensil to dress bathe eat: Sometimes | 0 | 0 | 2 | 3 | 2
  Week 64: Device/Utensil to dress bathe eat: Often | 0 | 1 | 0 | 0 | 0
  Week 64: Device/Utensil to dress bathe eat: Always | 1 | 0 | 0 | 0 | 2
  Week 64: Other aids or devices: number analyzed (Participants) | 135 | 138 | 285 | 285 | 414
  Week 64: Other aids or devices: Never | 125 | 135 | 277 | 273 | 387
  Week 64: Other aids or devices: Rarely | 1 | 1 | 0 | 0 | 9
  Week 64: Other aids or devices: Sometimes | 5 | 1 | 5 | 7 | 8
  Week 64: Other aids or devices: Often | 2 | 1 | 1 | 3 | 7
  Week 64: Other aids or devices: Always | 2 | 0 | 2 | 2 | 3
  Week 80: Walking aid use: number analyzed (Participants) | 61 | 59 | 134 | 143 | 191
  Week 80: Walking aid use: Never | 55 | 56 | 130 | 141 | 182
  Week 80: Walking aid use: Rarely | 0 | 0 | 1 | 1 | 2
  Week 80: Walking aid use: Sometimes | 3 | 1 | 1 | 1 | 4
  Week 80: Walking aid use: Often | 2 | 1 | 1 | 0 | 2
  Week 80: Walking aid use: Always | 1 | 1 | 1 | 0 | 1
  Week 80: Wheelchair use: number analyzed (Participants) | 61 | 59 | 134 | 143 | 191
  Week 80: Wheelchair use: Never | 61 | 59 | 134 | 142 | 190
  Week 80: Wheelchair use: Rarely | 0 | 0 | 0 | 1 | 0
  Week 80: Wheelchair use: Sometimes | 0 | 0 | 0 | 0 | 0
  Week 80: Wheelchair use: Often | 0 | 0 | 0 | 0 | 0
  Week 80: Wheelchair use: Always | 0 | 0 | 0 | 0 | 1
  Week 80: Device/Utensil to dress bathe eat: number analyzed (Participants) | 61 | 59 | 134 | 143 | 191
  Week 80: Device/Utensil to dress bathe eat: Never | 60 | 57 | 132 | 142 | 190
  Week 80: Device/Utensil to dress bathe eat: Rarely | 0 | 1 | 0 | 1 | 1
  Week 80: Device/Utensil to dress bathe eat: Sometimes | 1 | 1 | 0 | 0 | 0
  Week 80: Device/Utensil to dress bathe eat: Often | 0 | 0 | 1 | 0 | 0
  Week 80: Device/Utensil to dress bathe eat: Always | 0 | 0 | 1 | 0 | 0
  Week 80: Other aids or devices: number analyzed (Participants) | 61 | 59 | 134 | 143 | 191
  Week 80: Other aids or devices: Never | 57 | 58 | 128 | 139 | 184
  Week 80: Other aids or devices: Rarely | 1 | 1 | 1 | 1 | 0
  Week 80: Other aids or devices: Sometimes | 1 | 0 | 1 | 3 | 3
  Week 80: Other aids or devices: Often | 2 | 0 | 1 | 0 | 2
  Week 80: Other aids or devices: Always | 0 | 0 | 3 | 0 | 2

47. Secondary Outcome: Health Care Resource Utilization (HCRU): Number of Participants Who Quit Job Due to Low Back Pain
Description: Low back pain HCRU assessed utilization of healthcare resources during the last 3 months for baseline, weeks 64 and 80, via IRT. Domain evaluated was number of participants who quit job due to low back pain.
Time Frame: Baseline, Weeks 64 and 80
Population: ITT population included all randomized participants who received at least one dose of SC study medication (either tanezumab or matching placebo). Here, 'n' = Participants who were evaluable for quiting job due to low back pain.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Followed by Tanezumab 5 mg | Placebo Followed by Tanezumab 10 mg | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 202 | 204 | 407 | 407 | 605
Participants
  Baseline: number analyzed (Participants) | 202 | 204 | 406 | 407 | 605
  Baseline | 17 | 14 | 28 | 31 | 47
  Week 64: number analyzed (Participants) | 135 | 138 | 285 | 285 | 414
  Week 64 | 6 | 2 | 11 | 8 | 14
  Week 80: number analyzed (Participants) | 61 | 59 | 134 | 143 | 188
  Week 80 | 4 | 2 | 4 | 3 | 3

48. Secondary Outcome: Health Care Resource Utilization (HCRU): Duration Since Quitting Job Due to Low Back Pain
Description: Low back pain HCRU assessed utilization of healthcare resources during the last 3 months for baseline, weeks 64 and 80, via IRT. Domain evaluated was duration since quitting job due to low back pain.
Time Frame: Baseline, Weeks 64 and 80
Population: ITT population. Not all participants of the ITT population had data collected at each of the time points for this outcome measure. Hence, "N" signifies only those participants who were evaluable for this OM. Additional participants apart from the ones who had responded for quitting job responded to duration since quitting job.
Measure: Median (Full Range); unit: years
Arm/Group | Placebo Followed by Tanezumab 5 mg | Placebo Followed by Tanezumab 10 mg | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 17 | 15 | 28 | 31 | 47
years
  Baseline | 2.0 [0.2 to 15.0] | 2.0 [0.3 to 15.6] | 1.0 [0.1 to 20.5] | 3.8 [0.1 to 16.0] | 2.3 [0.1 to 90.3]
  Week 64: number analyzed (Participants) | 6 | 3 | 14 | 10 | 21
  Week 64 | 1.1 [0.1 to 13.2] | 5.2 [2.5 to 7.1] | 2.2 [0.2 to 32.0] | 2.0 [0.1 to 17.0] | 2.5 [0.2 to 25.2]
  Week 80: number analyzed (Participants) | 4 | 2 | 4 | 3 | 3
  Week 80 | 8.6 [5.8 to 99.1] | 4.7 [1.0 to 8.3] | 0.2 [0.0 to 3.3] | 3.5 [0.8 to 17.1] | 3.5 [3.0 to 5.0]

49. Secondary Outcome: Treatment Satisfaction Score Determined With Treatment Satisfaction Questionnaire for Medication Version II (TSQM v II) at Weeks 16 and 56
Description: TSQM v.II: self-administered 11-item validated scale that quantified participant's level of satisfaction with study medication (7 questions scored on 7-point Likert scale [1= extremely dissatisfied, 2=very dissatisfied, 3=dissatisfied, 4=somewhat satisfied, 5=satisfied, 6=very satisfied, 7=extremely satisfied]), effectiveness and side effects/tolerability (3 questions scored on 5 point Likert scale [1= extremely dissatisfied, 2=very dissatisfied, 3=somewhat dissatisfied, 4=slightly dissatisfied, 5=not at all dissatisfied], 1 question on 2 point scale [0 =No, 1=Yes]). 11 questions of TSQM were used to calculate 4 endpoints of effectiveness, side effects, convenience and global satisfaction, each scored on a 0-100 scale with 100=best level of satisfaction. Pre-specified intent of study was to compare tanezumab Vs placebo for data up to & including W16 & comparisons of tanezumab Vs tramadol for data up to & including W56.
Time Frame: Weeks 16 and 56
Population: ITT population. Here, "N" signifies participants evaluable for this outcome measure. Data were not collected after W16 in placebo arm for this outcome measure, as those who met criteria to continue, switched to active treatment with tanezumab after W16.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 329 | 338 | 343 | 456
units on a scale
  Week 16: Effectiveness | 56.67 (1.50) | 63.69 (1.48) | 62.87 (1.48) | 61.39 (1.30)
  Week 16: Side Effects: number analyzed (Participants) | 39 | 49 | 49 | 120
  Week 16: Side Effects | 66.95 (3.76) | 79.26 (3.31) | 79.51 (3.31) | 70.83 (2.15)
  Week 16: Convenience | 73.11 (1.16) | 75.68 (1.16) | 76.37 (1.15) | 74.63 (1.04)
  Week 16: Global Satisfaction | 64.90 (1.41) | 70.32 (1.39) | 68.64 (1.38) | 67.12 (1.22)
  Week 56: Effectiveness: number analyzed (Participants) | 0 | 141 | 159 | 206
  Week 56: Effectiveness |  | 72.66 (2.12) | 72.51 (2.01) | 71.21 (1.79)
  Week 56: Side Effects: number analyzed (Participants) | 0 | 9 | 17 | 41
  Week 56: Side Effects |  | 78.92 (6.32) | 89.37 (4.76) | 76.20 (3.09)
  Week 56: Convenience: number analyzed (Participants) | 0 | 141 | 159 | 206
  Week 56: Convenience |  | 78.72 (1.69) | 80.52 (1.60) | 78.42 (1.45)
  Week 56: Global Satisfaction: number analyzed (Participants) | 0 | 141 | 159 | 206
  Week 56: Global Satisfaction |  | 78.11 (1.83) | 78.49 (1.73) | 74.57 (1.55)
Statistical Analysis 1: Comparison: Placebo vs Pooled Tanezumab 5 mg; TSQM Effectiveness; Week 16: p-value was computed using ANCOVA with covariates of baseline average LBPI score, treatment, and study site as a random effect; Test type: Superiority; p = 0.0005, ANCOVA; LS Mean Difference = 7.02, 95% CI 2-sided [3.07 to 10.97], Standard Error of Mean 2.01
Statistical Analysis 2: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 49, analysis 1]; Test type: Superiority; p = 0.0021, ANCOVA; LS Mean Difference = 6.21, 95% CI 2-sided [2.26 to 10.15], Standard Error of Mean 2.01
Statistical Analysis 3: Comparison: Placebo vs Tramadol; [analysis description as in outcome 49, analysis 1]; Test type: Superiority; p = 0.0125, ANCOVA; LS Mean Difference = 4.72, 95% CI 2-sided [1.02 to 8.42], Standard Error of Mean 1.89
Statistical Analysis 4: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 49, analysis 1]; Test type: Superiority; p = 0.2176, ANCOVA; LS Mean Difference = 2.31, 95% CI 2-sided [-1.36 to 5.97], Standard Error of Mean 1.87
Statistical Analysis 5: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 49, analysis 1]; Test type: Superiority; p = 0.4235, ANCOVA; LS Mean Difference = 1.49, 95% CI 2-sided [-2.16 to 5.14], Standard Error of Mean 1.86
Statistical Analysis 6: Comparison: Placebo vs Pooled Tanezumab 5 mg; TSQM Side Effects; Week 16: p-value was computed using ANCOVA with covariates of baseline average LBPI score, treatment, and study site as a random effect; Test type: Superiority; p = 0.0143, ANCOVA; LS Mean Difference = 12.30, 95% CI 2-sided [2.50 to 22.11], Standard Error of Mean 4.96
Statistical Analysis 7: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 49, analysis 6]; Test type: Superiority; p = 0.0124, ANCOVA; LS Mean Difference = 12.55, 95% CI 2-sided [2.76 to 22.35], Standard Error of Mean 4.96
Statistical Analysis 8: Comparison: Placebo vs Tramadol; [analysis description as in outcome 49, analysis 6]; Test type: Superiority; p = 0.3675, ANCOVA; LS Mean Difference = 3.88, 95% CI 2-sided [-4.60 to 12.36], Standard Error of Mean 4.29
Statistical Analysis 9: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 49, analysis 6]; Test type: Superiority; p = 0.0319, ANCOVA; LS Mean Difference = 8.42, 95% CI 2-sided [0.74 to 16.11], Standard Error of Mean 3.89
Statistical Analysis 10: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 49, analysis 6]; Test type: Superiority; p = 0.0276, ANCOVA; LS Mean Difference = 8.67, 95% CI 2-sided [0.97 to 16.38], Standard Error of Mean 3.90
Statistical Analysis 11: Comparison: Placebo vs Pooled Tanezumab 5 mg; TSQM Convenience; Week 16: p-value was computed using ANCOVA with covariates of baseline average LBPI score, treatment, and study site as a random effect; Test type: Superiority; p = 0.0627, ANCOVA; LS Mean Difference = 2.57, 95% CI 2-sided [-0.14 to 5.27], Standard Error of Mean 1.38
Statistical Analysis 12: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 49, analysis 11]; Test type: Superiority; p = 0.0187, ANCOVA; LS Mean Difference = 3.26, 95% CI 2-sided [0.54 to 5.97], Standard Error of Mean 1.38
Statistical Analysis 13: Comparison: Placebo vs Tramadol; [analysis description as in outcome 49, analysis 11]; Test type: Superiority; p = 0.2419, ANCOVA; LS Mean Difference = 1.52, 95% CI 2-sided [-1.03 to 4.06], Standard Error of Mean 1.30
Statistical Analysis 14: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 49, analysis 11]; Test type: Superiority; p = 0.4124, ANCOVA; LS Mean Difference = 1.05, 95% CI 2-sided [-1.46 to 3.56], Standard Error of Mean 1.28
Statistical Analysis 15: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 49, analysis 11]; Test type: Superiority; p = 0.1730, ANCOVA; LS Mean Difference = 1.74, 95% CI 2-sided [-0.76 to 4.24], Standard Error of Mean 1.27
Statistical Analysis 16: Comparison: Placebo vs Pooled Tanezumab 5 mg; TSQM Global Satisfaction; Week 16: p-value was computed using ANCOVA with covariates of baseline average LBPI score, treatment, and study site as a random effect; Test type: Superiority; p = 0.0037, ANCOVA; LS Mean Difference = 5.42, 95% CI 2-sided [1.77 to 9.08], Standard Error of Mean 1.86
Statistical Analysis 17: Comparison: Placebo vs Pooled Tanezumab 10 mg; [analysis description as in outcome 49, analysis 16]; Test type: Superiority; p = 0.0449, ANCOVA; LS Mean Difference = 3.74, 95% CI 2-sided [0.09 to 7.39], Standard Error of Mean 1.86
Statistical Analysis 18: Comparison: Placebo vs Tramadol; [analysis description as in outcome 49, analysis 16]; Test type: Superiority; p = 0.2038, ANCOVA; LS Mean Difference = 2.22, 95% CI 2-sided [-1.21 to 5.65], Standard Error of Mean 1.75
Statistical Analysis 19: Comparison: Pooled Tanezumab 5 mg vs Tramadol; [analysis description as in outcome 49, analysis 16]; Test type: Superiority; p = 0.0644, ANCOVA; LS Mean Difference = 3.20, 95% CI 2-sided [-0.19 to 6.59], Standard Error of Mean 1.73
Statistical Analysis 20: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 49, analysis 16]; Test type: Superiority; p = 0.3775, ANCOVA; LS Mean Difference = 1.52, 95% CI 2-sided [-1.86 to 4.90], Standard Error of Mean 1.72
Statistical Analysis 21: Comparison: Pooled Tanezumab 5 mg vs Tramadol; TSQM Effectiveness; Week 56: p-value was computed using ANCOVA with covariates of baseline average LBPI score, treatment, and study site as a random effect; Test type: Superiority; p = 0.5806, ANCOVA; LS Mean Difference = 1.45, 95% CI 2-sided [-3.70 to 6.60], Standard Error of Mean 2.62
Statistical Analysis 22: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 49, analysis 21]; Test type: Superiority; p = 0.6084, ANCOVA; LS Mean Difference = 1.30, 95% CI 2-sided [-3.68 to 6.27], Standard Error of Mean 2.53
Statistical Analysis 23: Comparison: Pooled Tanezumab 5 mg vs Tramadol; TSQM Side Effects; Week 56: p-value was computed using ANCOVA with covariates of baseline average LBPI score, treatment, and study site as a random effect; Test type: Superiority; p = 0.6991, ANCOVA; LS Mean Difference = 2.71, 95% CI 2-sided [-11.56 to 16.99], Standard Error of Mean 6.95
Statistical Analysis 24: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 49, analysis 23]; Test type: Superiority; p = 0.0265, ANCOVA; LS Mean Difference = 13.17, 95% CI 2-sided [1.66 to 24.68], Standard Error of Mean 5.60
Statistical Analysis 25: Comparison: Pooled Tanezumab 5 mg vs Tramadol; TSQM Convenience; Week 56: p-value was computed using ANCOVA with covariates of baseline average LBPI score, treatment, and study site as a random effect; Test type: Superiority; p = 0.8795, ANCOVA; LS Mean Difference = 0.30, 95% CI 2-sided [-3.61 to 4.21], Standard Error of Mean 1.99
Statistical Analysis 26: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 49, analysis 25]; Test type: Superiority; p = 0.2758, ANCOVA; LS Mean Difference = 2.10, 95% CI 2-sided [-1.68 to 5.87], Standard Error of Mean 1.92
Statistical Analysis 27: Comparison: Pooled Tanezumab 5 mg vs Tramadol; TSQM Global Satisfaction; Week 56: p-value was computed using ANCOVA with covariates of baseline average LBPI score, treatment, and study site as a random effect; Test type: Superiority; p = 0.1197, ANCOVA; LS Mean Difference = 3.54, 95% CI 2-sided [-0.92 to 8.00], Standard Error of Mean 2.27
Statistical Analysis 28: Comparison: Pooled Tanezumab 10 mg vs Tramadol; [analysis description as in outcome 49, analysis 27]; Test type: Superiority; p = 0.0743, ANCOVA; LS Mean Difference = 3.93, 95% CI 2-sided [-0.39 to 8.24], Standard Error of Mean 2.19

50. Secondary Outcome: Patient Reported Treatment Impact Assessment-Modified (mPRTI) Score at Weeks 16 and 56: Participant Global Preference Assessment- What is The Current or Most Recent Treatment You Were Receiving For Low Back Pain Before Enrolling?
Description: The mPRTI is a self-administered questionnaire containing participant reported treatment impact assessment (to assess participant satisfaction), participant global preference assessment (to assess previous treatment and preference to continue using the investigational product) and participant willingness to use drug again assessment. To assess previous treatment, participants responded for, 1=injectable prescription medicines, 2=prescription medicines taken by mouth, 3=surgery, 4=prescription medicines and surgery and 5=no treatment. Pre-specified intent of study was to compare tanezumab Vs placebo for data up to & including W16 & comparisons of tanezumab Vs tramadol for data up to & including W56.
Time Frame: Weeks 16 and 56
Population: as for outcome 49
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 322 | 333 | 340 | 450
Participants
  Week 16: Injectable prescription medicines | 20 | 21 | 22 | 39
  Week 16: Prescription medicines taken by mouth | 213 | 211 | 229 | 287
  Week 16: Surgery | 2 | 2 | 1 | 1
  Week 16: Prescription medicines and surgery | 7 | 9 | 10 | 14
  Week 16: No treatment | 80 | 90 | 78 | 109
  Week 56: number analyzed (Participants) | 0 | 141 | 159 | 206
  Week 56: Injectable prescription medicines |  | 6 | 13 | 9
  Week 56: Prescription medicines taken by mouth |  | 91 | 102 | 147
  Week 56: Surgery |  | 2 | 0 | 3
  Week 56: Prescription medicines and surgery |  | 7 | 4 | 3
  Week 56: No treatment |  | 35 | 40 | 44

51. Secondary Outcome: Patient Reported Treatment Impact Assessment-Modified (mPRTI) Score at Weeks 16 and 56: Participant Global Preference Assessment- Overall, do You Prefer The Drug That You Received in This Study to Previous Treatment?
Description: mPRTI : self-administered questionnaire containing participant reported treatment impact assessment (to assess participant satisfaction),participant global preference assessment (to assess previous treatment & preference to continue using investigational product) & participant willingness to use drug again assessment. To assess preference to continue using investigational product, participants responded using IRT on 5 point likert scale from 1-5, where, 1= yes, I definitely prefer drug that I am receiving now, 2= I have a slight preference for drug that I am receiving now, 3= I have no preference either way, 4= I have a slight preference for my previous treatment, 5= No, I definitely prefer my previous treatment. Higher scores indicate lesser preference to use investigational product. Pre-specified intent of study was to compare tanezumab Vs placebo for data up to & including W16 & comparisons of tanezumab Vs tramadol for data up to & including W56.
Time Frame: Weeks 16 and 56
Population: as for outcome 49
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 322 | 333 | 340 | 450
Participants
  Week 16: Yes, definitely prefer the study drug | 150 | 172 | 191 | 232
  Week 16: Slight preference for the study drug | 57 | 62 | 50 | 89
  Week 16: No preference either way | 62 | 66 | 55 | 82
  Week 16: Slight preference for my previous treatment | 24 | 14 | 23 | 17
  Week 16: No, definitely prefer my previous treatment | 29 | 19 | 21 | 30
  Week 56: number analyzed (Participants) | 0 | 141 | 159 | 206
  Week 56: Yes, definitely prefer the study drug |  | 90 | 104 | 129
  Week 56: Slight preference for the study drug |  | 30 | 36 | 42
  Week 56: No preference either way |  | 15 | 12 | 22
  Week 56: Slight preference for my previous treatment |  | 2 | 4 | 7
  Week 56: No, definitely prefer my previous treatment |  | 4 | 3 | 6

52. Secondary Outcome: Patient Reported Treatment Impact Assessment-Modified (mPRTI) Score at Weeks 16 and 56: Participant Willingness to Use Drug Again Assessment- Willing to Use The Same Drug That You Have Received in This Study For Your Low Back Pain Pain?
Description: mPRTI: self-administered questionnaire containing participant reported treatment impact assessment (to assess participant satisfaction),participant global preference assessment (to assess previous treatment and preference to continue using the investigational product) & participant willingness to use drug again assessment. To assess participants willingness to use drug again, participants responded using IRT on 5 point likert scale from 1-5, where, 1= yes, I would definitely want to use the same drug again, 2= I might want to use the same drug again, 3= I am not sure, 4= I might not want to use the same drug again, 5= no, I definitely would not want to use the same drug again. Higher scores indicate lesser willingness to use the investigational product. Pre-specified intent of study was to compare tanezumab Vs placebo for data up to & including W16 & comparisons of tanezumab Vs tramadol for data up to & including W56.
Time Frame: Weeks 16 and 56
Population: as for outcome 49
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Pooled Tanezumab 5 mg | Pooled Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 322 | 333 | 340 | 450
Participants
  Week 16: Yes, definitely want to use the same drug again | 167 | 191 | 210 | 251
  Week 16: Might want to use the same drug again | 61 | 80 | 58 | 98
  Week 16: I am not sure | 51 | 36 | 38 | 64
  Week 16: Might not want to use the same drug again | 11 | 10 | 13 | 13
  Week 16: No:definitely wouldn't want to use same drug again | 32 | 16 | 21 | 24
  Week 56: number analyzed (Participants) | 0 | 141 | 159 | 206
  Week 56: Yes, definitely want to use the same drug again |  | 99 | 114 | 133
  Week 56: Might want to use the same drug again |  | 23 | 31 | 41
  Week 56: I am not sure |  | 15 | 10 | 26
  Week 56: Might not want to use the same drug again |  | 0 | 2 | 4
  Week 56: No:definitely wouldn't want to use same drug again |  | 4 | 2 | 2

53. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and up to week 80 that were absent before treatment or that worsened relative to pretreatment state. AEs included both serious and non-serious AEs.
Time Frame: Baseline up to Week 80
Population: Safety population analyzed.Pre-specified intent of study for safety summaries until W80 was to summarize data by 4 arms.'N' in placebo arm=number of participants who received only placebo for entire study.Those who were there up to W16,but switched to tanezumab after W16 are included in tanezumab 5/10 mg arm. 'N'=participants evaluable for this OM.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo (Week 16): Placebo matched to tanezumab (RN624 or PF-04383119) injection administered SC, once every 8 weeks and placebo tablets matched to tramadol PR, orally, once daily from Day 1 up to week 16, inclusive of those participants who were randomized to placebo but received tramadol.
- Safety Evaluation: Tanezumab 5 mg: Placebo matched to tanezumab (RN624 or PF-04383119) injection administered SC, once every 8 weeks and placebo tablets matched to tramadol PR, orally, once daily from Day 1 up to week 16. At week 16, participants who met efficacy responder criteria (>=30 % reduction in average LBPI score and >=15% reduction in average LBPI score relative to baseline at any week from week 1 to week 15), then received tanezumab 5 mg SC, once every 8 weeks plus placebo tablets matched to tramadol PR, orally, once daily, from week 16 to week 56.Those participants were also included who received tanezumab 5 mg injection administered SC once every 8 weeks and placebo tablets matched to tramadol PR, orally, once daily from Day 1 up to week 56.
- Safety Evaluation: Tanezumab 10 mg: Placebo matched to tanezumab (RN624 or PF-04383119) injection administered SC, once every 8 weeks and placebo tablets matched to tramadol PR, orally, once daily from Day 1 up to week 16. At week 16, participants who met efficacy responder criteria, then received tanezumab 10 mg, SC, once every 8 weeks plus placebo tablets matched to tramadol PR, orally, once daily, from week 16 to week 56.Those participants were also included who received tanezumab 10 mg injection administered SC once every 8 weeks from Day 1 and placebo tablets matched to tramadol PR, orally, once daily from Day 1 up to week 56.
Arm/Group | Placebo (Week 16) | Safety Evaluation: Tanezumab 5 mg | Safety Evaluation: Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 215 | 506 | 502 | 602
Participants
  AEs | 125 | 319 | 347 | 421
  SAEs | 7 | 21 | 37 | 25

54. Secondary Outcome: Number of Participants With Treatment-Emergent Treatment-Related Adverse Events (AEs) and Serious Adverse Events (SAEs) up to Week 56
Description: Treatment-related AE was any untoward medical occurrence attributed to study drug in participant who received study drug. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and up to W56 that were absent before treatment or that worsened relative to pre-treatment state. Relatedness to study drug was assessed by the investigator. Pre-specified intent of study for summaries for the entire treatment period (up to week 56), data was summarized by 3 arms.
Time Frame: Baseline up to Week 56
Population: The safety population was defined as all participants treated with tanezumab or placebo SC. Here, "Overall number of participants analyzed"=participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Safety Evaluation: Tanezumab 5 mg: Placebo matched to tanezumab (RN624 or PF-04383119) injection administered SC, once every 8 weeks from Day 1 (baseline), and placebo tablets matched to tramadol PR, orally, once daily from Day 1 up to week 16. At week 16, participants who met efficacy responder criteria (>=30 % reduction in average LBPI score and >=15% reduction in average LBPI score relative to baseline at any week from week 1 to week 15), then received tanezumab 5 mg or 10 mg, SC, once every 8 weeks plus placebo tablets matched to tramadol PR, orally, once daily, from week 16 to week 56.Those participants were also included who received tanezumab 5 mg injection administered SC once every 8 weeks from Day 1 and placebo tablets matched to tramadol PR, orally, once daily from Day 1 up to week 56.
- Safety Evaluation: Tanezumab 10 mg: Placebo matched to tanezumab (RN624 or PF-04383119) injection administered SC, once every 8 weeks from Day 1 (baseline), and placebo tablets matched to tramadol PR, orally, once daily from Day 1 up to week 16. At week 16, participants who met efficacy responder criteria (>=30 % reduction in average LBPI score and >=15% reduction in average LBPI score relative to baseline at any week from week 1 to week 15), then received tanezumab 5 mg or 10 mg, SC, once every 8 weeks plus placebo tablets matched to tramadol PR, orally, once daily, from week 16 to week 56.Those participants were also included who received tanezumab 10 mg injection administered SC once every 8 weeks from Day 1 and placebo tablets matched to tramadol PR, orally, once daily from Day 1 up to week 56.
Arm/Group | Safety Evaluation: Tanezumab 5 mg | Safety Evaluation: Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 506 | 502 | 602
Participants
  AEs | 105 | 119 | 200
  SAEs | 1 | 4 | 1

55. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities With Regard to Normal Baseline
Description: Primary Abnormality criteria: HGB, hematocrit, RBC count <0.8* lower limit of normal(LLN); Ery. mean corpuscular volume/hemoglobin/ HGB concentration, RBCs distribution width <0.9*LLN, >1.1*upper limit of normal(ULN); platelets <0.5*LLN,>1.75*ULN; WBC count<0.6*LLN, >1.5*ULN; Lymphocytes,Leukocytes,Neutrophils <0.8*LLN, >1.2*ULN; Basophils,Eosinophils,Monocytes>1.2*ULN; Prothrombin time/Intl. normalized ratio>1.1*ULN; total bilirubin>1.5*ULN; aspartate aminotransferase,alanine aminotransferase,gamma GT,LDH,alkaline phosphatase >3.0*ULN; total protein; albumin<0.8*LLN, >1.2*ULN; blood urea nitrogen,creatinine,Cholesterol,triglycerides >1.3*ULN; Urate>1.2*ULN; sodium<0.95*LLN,>1.05*ULN; potassium,chloride,calcium,magnesium,bicarbonate <0.9*LLN, >1.1*ULN; phosphate<0.8*LLN, >1.2*ULN; glucose<0.6*LLN, >1.5*ULN; HGB A1C >1.3*ULN; creatine kinase>2.0*ULN, specific gravity<1.003, >1.030; pH<4.5, >8; Urine Glucose, protein,HGB,bilirubin >=1; Ketones>=1;Urine erythrocytes,Leukocytes>=20.
Time Frame: Baseline up to Week 80
Population: Safety population was analyzed."N"=participants evaluable for this OM. Pre-specified intent of study for safety summaries until W80 was to summarize data by 4 arms.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Week 16) | Safety Evaluation: Tanezumab 5 mg | Safety Evaluation: Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 129 | 434 | 433 | 488
Participants | 16 | 56 | 61 | 59

56. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities With Regard to Abnormal Baseline
Description: Primary Abnormality criteria: hemoglobin; hematocrit; RBC count < 0.8*LLN; Ery. mean corpuscular volume/ hemoglobin/ HGB concentration, erythrocytes distribution width <0.9*LLN, >1.1*ULN; platelets <0.5*LLN,>1.75*upper limit of normal (ULN); white blood cell count<0.6*LLN, >1.5*ULN; Lymphocytes, Leukocytes, Neutrophils <0.8*LLN, >1.2*ULN; Basophils, Eosinophils, Monocytes >1.2*ULN; total bilirubin>1.5*ULN; aspartate aminotransferase, alanine aminotransferase, gamma GT,LDH, alkaline phosphatase >3.0*ULN; total protein; albumin<0.8*LLN, >1.2*ULN; blood urea nitrogen, creatinine, Cholesterol, triglycerides >1.3*ULN; Urate >1.2*ULN; sodium <0.95*LLN,>1.05*ULN; potassium, chloride, calcium, magnesium, bicarbonate <0.9*LLN, >1.1*ULN; phosphate <0.8*LLN, >1.2*ULN; glucose <0.6*LLN, >1.5*ULN; Hemoglobin A1C >1.3*ULN; creatine kinase >2.0*ULN; Nitrite >=1.
Time Frame: Baseline up to Week 80
Population: as for outcome 55
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Week 16) | Safety Evaluation: Tanezumab 5 mg | Safety Evaluation: Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 92 | 332 | 308 | 373
Participants | 11 | 40 | 39 | 45

57. Secondary Outcome: Change From Baseline in Blood Pressure (BP) at Weeks 2, 4, 8, 16, 24, 32, 40, 48, 56, 64 and 80
Description: Measurement of BP included sitting systolic blood pressure (SBP) and diastolic blood pressure (DBP). Pre-specified intent of study for safety summaries until W80 was to summarize data by 4 arms.
Time Frame: Baseline, Weeks 2, 4, 8, 16, 24, 32, 40, 48, 56, 64 and 80
Population: Safety population. Data not collected after W16 in placebo arm for this OM, as those who met criteria to continue, switched to active treatment with tanezumab after W16. 'N' in placebo arm=participants who received only placebo for entire study. Those who were there up to W16,but switched to tanezumab after W16 are included in tanezumab 5/10mg arm.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Placebo (Week 16) | Safety Evaluation: Tanezumab 5 mg | Safety Evaluation: Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 215 | 506 | 502 | 602
millimeters of mercury (mmHg)
  SBP: Baseline | 122.3 (12.20) | 123.8 (13.25) | 122.6 (12.36) | 123.7 (13.77)
  SBP:Change at Week 2: number analyzed (Participants) | 191 | 488 | 478 | 560
  SBP:Change at Week 2 | -1.3 (10.50) | -2.0 (11.05) | -1.4 (10.62) | -1.4 (11.37)
  SBP:Change at Week 4: number analyzed (Participants) | 173 | 473 | 468 | 535
  SBP:Change at Week 4 | -2.1 (11.36) | -2.2 (11.46) | -1.7 (10.65) | -1.8 (11.81)
  SBP:Change at Week 8: number analyzed (Participants) | 152 | 454 | 450 | 490
  SBP:Change at Week 8 | -1.1 (11.37) | -1.0 (11.38) | -2.2 (11.02) | -1.7 (11.99)
  SBP:Change at Week 16: number analyzed (Participants) | 8 | 340 | 344 | 314
  SBP:Change at Week 16 | -0.5 (10.56) | -2.2 (10.75) | -1.4 (11.10) | -1.6 (11.96)
  SBP:Change at Week 24: number analyzed (Participants) | 0 | 288 | 295 | 269
  SBP:Change at Week 24 |  | -2.2 (10.51) | -1.8 (11.53) | -1.9 (12.67)
  SBP:Change at Week 32: number analyzed (Participants) | 0 | 240 | 255 | 229
  SBP:Change at Week 32 |  | -0.6 (11.36) | -1.4 (11.53) | -2.2 (12.54)
  SBP:Change at Week 40: number analyzed (Participants) | 0 | 218 | 239 | 218
  SBP:Change at Week 40 |  | -2.0 (11.27) | -1.6 (11.91) | -1.0 (11.99)
  SBP:Change at Week 48: number analyzed (Participants) | 0 | 211 | 229 | 208
  SBP:Change at Week 48 |  | -2.0 (12.12) | -2.2 (11.51) | -0.8 (12.46)
  SBP:Change at Week 56: number analyzed (Participants) | 0 | 202 | 222 | 204
  SBP:Change at Week 56 |  | -1.5 (11.18) | -3.0 (12.03) | -1.1 (12.03)
  SBP:Change at Week 64: number analyzed (Participants) | 0 | 199 | 209 | 195
  SBP:Change at Week 64 |  | -0.9 (11.51) | -1.9 (12.28) | -1.2 (11.59)
  SBP:Change at Week 80: number analyzed (Participants) | 0 | 193 | 201 | 191
  SBP:Change at Week 80 |  | -1.4 (10.82) | 0.1 (12.62) | -1.0 (11.77)
  DBP: Baseline | 77.9 (9.10) | 78.6 (8.98) | 77.4 (8.48) | 78.2 (9.01)
  DBP:Change at Week 2: number analyzed (Participants) | 191 | 488 | 478 | 560
  DBP:Change at Week 2 | -1.2 (7.63) | -1.1 (7.49) | -1.5 (7.91) | -0.7 (8.21)
  DBP:Change at Week 4: number analyzed (Participants) | 173 | 473 | 468 | 535
  DBP:Change at Week 4 | -1.7 (7.59) | -1.5 (7.75) | -1.1 (7.59) | -0.9 (7.94)
  DBP:Change at Week 8: number analyzed (Participants) | 152 | 454 | 450 | 490
  DBP:Change at Week 8 | 0.0 (7.24) | -1.2 (8.04) | -1.5 (8.26) | -0.8 (8.13)
  DBP:Change at Week 16: number analyzed (Participants) | 8 | 340 | 344 | 314
  DBP:Change at Week 16 | -0.6 (5.63) | -1.2 (8.21) | -1.0 (8.39) | -0.8 (8.15)
  DBP:Change at Week 24: number analyzed (Participants) | 0 | 288 | 295 | 269
  DBP:Change at Week 24 |  | -1.2 (8.04) | -0.8 (8.13) | -1.0 (7.76)
  DBP:Change at Week 32: number analyzed (Participants) | 0 | 240 | 255 | 229
  DBP:Change at Week 32 |  | -0.6 (7.80) | -0.5 (8.10) | -0.4 (8.39)
  DBP:Change at Week 40: number analyzed (Participants) | 0 | 218 | 239 | 218
  DBP:Change at Week 40 |  | -1.4 (8.56) | -1.1 (8.13) | -0.7 (8.36)
  DBP:Change at Week 48: number analyzed (Participants) | 0 | 211 | 229 | 208
  DBP:Change at Week 48 |  | -2.1 (9.05) | -1.3 (8.23) | -0.7 (7.93)
  DBP:Change at Week 56: number analyzed (Participants) | 0 | 202 | 222 | 204
  DBP:Change at Week 56 |  | -1.3 (8.92) | -1.3 (8.05) | -0.4 (7.75)
  DBP:Change at Week 64: number analyzed (Participants) | 0 | 199 | 209 | 195
  DBP:Change at Week 64 |  | -0.7 (8.03) | -0.0 (9.13) | -0.6 (8.95)
  DBP:Change at Week 80: number analyzed (Participants) | 0 | 193 | 201 | 191
  DBP:Change at Week 80 |  | -1.0 (8.13) | 0.5 (9.07) | -0.1 (8.55)

58. Secondary Outcome: Change From Baseline in Heart Rate at Weeks 2, 4, 8, 16, 24, 32, 40, 48, 56, 64 and 80
Description: Heart rate was measured at sitting position. Pre-specified intent of study for safety summaries until W80 was to summarize data by 4 arms.
Time Frame: Baseline, Weeks 2, 4, 8, 16, 24, 32, 40, 48, 56, 64 and 80
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo (Week 16) | Safety Evaluation: Tanezumab 5 mg | Safety Evaluation: Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 215 | 506 | 502 | 602
beats per minute
  Baseline | 73.3 (10.86) | 73.1 (10.23) | 72.5 (10.10) | 73.2 (10.61)
  Change at Week 2: number analyzed (Participants) | 191 | 488 | 478 | 560
  Change at Week 2 | 0.8 (9.14) | 0.5 (9.09) | 0.3 (9.23) | -0.2 (9.24)
  Change at Week 4: number analyzed (Participants) | 173 | 473 | 468 | 535
  Change at Week 4 | 1.6 (9.32) | 0.6 (8.82) | 0.4 (9.47) | 0.2 (9.57)
  Change at Week 8: number analyzed (Participants) | 152 | 454 | 450 | 490
  Change at Week 8 | 1.2 (8.88) | 0.1 (9.41) | -0.1 (9.87) | 0.0 (9.89)
  Change at Week 16: number analyzed (Participants) | 8 | 340 | 344 | 314
  Change at Week 16 | 5.1 (10.66) | -0.6 (9.99) | -1.0 (9.65) | -0.8 (10.13)
  Change at Week 24: number analyzed (Participants) | 0 | 288 | 295 | 269
  Change at Week 24 |  | 0.0 (9.32) | -0.3 (9.77) | 0.2 (10.09)
  Change at Week 32: number analyzed (Participants) | 0 | 240 | 255 | 229
  Change at Week 32 |  | 0.5 (9.82) | -0.3 (9.94) | 0.6 (9.72)
  Change at Week 40: number analyzed (Participants) | 0 | 218 | 239 | 218
  Change at Week 40 |  | 1.2 (10.14) | -0.5 (9.77) | 1.3 (9.55)
  Change at Week 48: number analyzed (Participants) | 0 | 211 | 229 | 208
  Change at Week 48 |  | 0.5 (9.72) | -0.5 (10.79) | 0.9 (10.33)
  Change at Week 56: number analyzed (Participants) | 0 | 202 | 222 | 204
  Change at Week 56 |  | 0.4 (10.31) | 0.2 (10.50) | 0.7 (11.10)
  Change at Week 64: number analyzed (Participants) | 0 | 199 | 209 | 195
  Change at Week 64 |  | 1.1 (10.66) | 0.8 (10.08) | 0.7 (10.22)
  Change at Week 80: number analyzed (Participants) | 0 | 193 | 201 | 191
  Change at Week 80 |  | 1.1 (10.93) | 1.2 (9.83) | 0.9 (11.48)

59. Secondary Outcome: Change From Baseline in Electrocardiogram (ECG) Parameters at Weeks 16, 56 and 80
Description: A 12-lead ECG was recorded after participants had rested for at least 5 minutes in the supine position in a quiet environment. All standard intervals {RR interval, PR interval, QRS interval, QT interval, QT interval corrected using Bazett's formula (QTcB) and QT interval corrected using Fridericia's formula (QTcF)} were collected. Pre-specified intent of study for safety summaries until W80 was to summarize data by 4 arms.
Time Frame: Baseline, Weeks 16, 56 and 80
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: millisecond
Arm/Group | Placebo (Week 16) | Safety Evaluation: Tanezumab 5 mg | Safety Evaluation: Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 215 | 506 | 502 | 602
millisecond
  RR Interval: Baseline: number analyzed (Participants) | 215 | 506 | 502 | 599
  RR Interval: Baseline | 928.5 (150.40) | 911.4 (140.72) | 915.4 (138.41) | 918.9 (138.55)
  RR Interval:Change at Week 16: number analyzed (Participants) | 6 | 338 | 335 | 308
  RR Interval:Change at Week 16 | 868.2 (235.72) | 897.1 (129.55) | 912.1 (142.81) | 894.9 (139.62)
  RR Interval:Change at Week 56: number analyzed (Participants) | 0 | 200 | 221 | 202
  RR Interval:Change at Week 56 |  | 894.5 (138.03) | 893.0 (144.30) | 881.5 (136.11)
  RR Interval:Change at Week 80: number analyzed (Participants) | 0 | 190 | 199 | 190
  RR Interval:Change at Week 80 |  | 870.5 (130.84) | 889.6 (143.10) | 876.5 (134.79)
  PR Interval: Baseline: number analyzed (Participants) | 213 | 506 | 501 | 596
  PR Interval: Baseline | 156.2 (20.51) | 157.3 (23.32) | 158.1 (22.93) | 157.8 (23.44)
  PR Interval:Change at Week 16: number analyzed (Participants) | 6 | 337 | 334 | 308
  PR Interval:Change at Week 16 | 158.8 (12.37) | 158.3 (21.99) | 159.6 (21.84) | 158.6 (23.37)
  PR Interval:Change at Week 56: number analyzed (Participants) | 0 | 199 | 221 | 202
  PR Interval:Change at Week 56 |  | 158.5 (21.78) | 158.1 (20.85) | 159.2 (22.13)
  PR Interval:Change at Week 80: number analyzed (Participants) | 0 | 190 | 198 | 189
  PR Interval:Change at Week 80 |  | 158.7 (22.15) | 157.7 (21.60) | 158.3 (21.46)
  QRS Interval: Baseline: number analyzed (Participants) | 215 | 506 | 502 | 599
  QRS Interval: Baseline | 90.9 (8.72) | 92.5 (11.06) | 93.5 (12.30) | 93.1 (12.02)
  QRS Interval:Change at Week 16: number analyzed (Participants) | 6 | 338 | 335 | 308
  QRS Interval:Change at Week 16 | 97.0 (8.29) | 93.4 (11.95) | 94.5 (13.27) | 93.9 (12.53)
  QRS Interval:Change at Week 56: number analyzed (Participants) | 0 | 200 | 221 | 202
  QRS Interval:Change at Week 56 |  | 92.8 (12.71) | 95.4 (12.62) | 94.2 (13.73)
  QRS Interval:Change at Week 80: number analyzed (Participants) | 0 | 190 | 199 | 190
  QRS Interval:Change at Week 80 |  | 93.0 (11.55) | 95.0 (12.53) | 94.4 (13.16)
  QT Interval: Baseline: number analyzed (Participants) | 215 | 504 | 502 | 599
  QT Interval: Baseline | 394.7 (29.67) | 393.1 (29.52) | 394.6 (27.54) | 393.7 (29.06)
  QT Interval:Change at Week 16: number analyzed (Participants) | 6 | 337 | 334 | 308
  QT Interval:Change at Week 16 | 379.8 (34.29) | 391.1 (28.13) | 393.5 (29.09) | 391.2 (30.30)
  QT Interval:Change at Week 56: number analyzed (Participants) | 0 | 200 | 221 | 201
  QT Interval:Change at Week 56 |  | 389.3 (27.11) | 392.8 (29.47) | 389.7 (29.44)
  QT Interval:Change at Week 80: number analyzed (Participants) | 0 | 190 | 198 | 190
  QT Interval:Change at Week 80 |  | 386.6 (27.67) | 393.0 (29.90) | 388.7 (29.33)
  QTCB Interval: Baseline: number analyzed (Participants) | 215 | 504 | 502 | 599
  QTCB Interval: Baseline | 411.7 (20.49) | 413.5 (20.19) | 414.4 (21.60) | 412.6 (22.39)
  QTCB Interval:Change at Week 16: number analyzed (Participants) | 6 | 337 | 334 | 308
  QTCB Interval:Change at Week 16 | 411.8 (17.50) | 414.5 (19.76) | 413.9 (22.67) | 415.3 (20.13)
  QTCB Interval:Change at Week 56: number analyzed (Participants) | 0 | 200 | 221 | 201
  QTCB Interval:Change at Week 56 |  | 413.5 (21.27) | 417.7 (22.02) | 416.8 (21.71)
  QTCB Interval:Change at Week 80: number analyzed (Participants) | 0 | 190 | 198 | 190
  QTCB Interval:Change at Week 80 |  | 416.1 (19.27) | 418.8 (22.13) | 417.0 (21.71)
  QTCF Interval: Baseline: number analyzed (Participants) | 215 | 504 | 502 | 599
  QTCF Interval: Baseline | 405.6 (18.22) | 406.3 (18.85) | 407.4 (18.93) | 405.9 (20.28)
  QTCF Interval:Change at Week 16: number analyzed (Participants) | 6 | 337 | 334 | 308
  QTCF Interval:Change at Week 16 | 400.3 (10.69) | 406.3 (18.45) | 406.7 (20.35) | 406.8 (19.04)
  QTCF Interval:Change at Week 56: number analyzed (Participants) | 0 | 200 | 221 | 201
  QTCF Interval:Change at Week 56 |  | 405.0 (18.46) | 408.9 (19.75) | 407.3 (19.74)
  QTCF Interval:Change at Week 80: number analyzed (Participants) | 0 | 190 | 198 | 190
  QTCF Interval:Change at Week 80 |  | 405.7 (17.70) | 409.7 (19.74) | 407.1 (19.81)

60. Secondary Outcome: Change From Baseline in Heart Rate (as Assessed by ECG) at Weeks 16, 56 and 80
Description: as for outcome 58
Time Frame: Baseline, Weeks 16, 56 and 80
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo (Week 16) | Safety Evaluation: Tanezumab 5 mg | Safety Evaluation: Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 215 | 506 | 502 | 602
beats per minute
  Baseline: number analyzed (Participants) | 215 | 506 | 502 | 599
  Baseline | 66.4 (11.34) | 67.4 (10.34) | 67.1 (10.31) | 66.9 (10.64)
  Change at Week 16: number analyzed (Participants) | 6 | 338 | 335 | 308
  Change at Week 16 | 72.3 (14.42) | 68.3 (10.00) | 67.4 (10.35) | 68.8 (10.99)
  Change at Week 56: number analyzed (Participants) | 0 | 200 | 221 | 202
  Change at Week 56 |  | 68.6 (10.29) | 68.9 (11.02) | 69.7 (11.26)
  Change at Week 80: number analyzed (Participants) | 0 | 190 | 199 | 190
  Change at Week 80 |  | 70.5 (10.57) | 69.3 (11.61) | 70.1 (10.98)

61. Secondary Outcome: Number of Participants With Confirmed Orthostatic Hypotension
Description: Orthostatic hypotension was defined as postural change (supine to standing) that met the following criteria: For systolic BP <=150 mmHg (mean supine): Reduction in systolic BP>=20 mmHg or reduction in diastolic BP>=10 mmHg at the 1 and/or 3 minute standing BP measurements. For systolic BP >150 mmHg (mean supine): Reduction in systolic BP>=30 mmHg or reduction in diastolic BP>=15 mmHg at the 1 and/or 3 minute standing BP measurements. If the 1 minute or 3 minute standing BP in a sequence met the orthostatic hypotension criteria, then that sequence was considered positive. If 2 of 2 or 2 of 3 sequences were positive, then orthostatic hypotension was considered confirmed. Pre-specified intent of study for safety summaries until W80 was to summarize data by 4 arms. Data not collected after W16 in placebo arm for this OM, as those who met criteria to continue, switched to active treatment with tanezumab after W16.
Time Frame: Baseline, Weeks 2, 4, 8, 16, 24, 32, 40, 48, 56, 64 and 80
Population: Safety population analyzed. 'N' in placebo arm=participants who received only placebo for entire study, those who were there up to W16,but switched to tanezumab after W16 are included in tanezumab 5/10mg arm. Hence, N=participants evaluable for this OM.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Week 16) | Safety Evaluation: Tanezumab 5 mg | Safety Evaluation: Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 215 | 503 | 501 | 601
Participants
  Baseline | 0 | 1 | 0 | 2
  Week 2: number analyzed (Participants) | 186 | 482 | 477 | 552
  Week 2 | 1 | 0 | 0 | 0
  Week 4: number analyzed (Participants) | 171 | 473 | 465 | 527
  Week 4 | 0 | 2 | 0 | 2
  Week 8: number analyzed (Participants) | 151 | 452 | 445 | 485
  Week 8 | 0 | 0 | 0 | 1
  Week 16: number analyzed (Participants) | 21 | 339 | 352 | 321
  Week 16 | 0 | 1 | 1 | 0
  Week 24: number analyzed (Participants) | 0 | 286 | 297 | 266
  Week 24 | 0 | 0 | 0 | 0
  Week 32: number analyzed (Participants) | 0 | 241 | 255 | 228
  Week 32 | 0 | 0 | 0 | 0
  Week 40: number analyzed (Participants) | 0 | 218 | 236 | 218
  Week 40 | 0 | 0 | 0 | 1
  Week 48: number analyzed (Participants) | 0 | 211 | 227 | 208
  Week 48 | 0 | 1 | 0 | 0
  Week 56: number analyzed (Participants) | 0 | 202 | 223 | 204
  Week 56 | 0 | 0 | 1 | 0
  Week 64: number analyzed (Participants) | 0 | 198 | 209 | 194
  Week 64 | 0 | 1 | 0 | 0
  Week 80: number analyzed (Participants) | 0 | 192 | 200 | 191
  Week 80 | 0 | 1 | 1 | 0

62. Secondary Outcome: Change From Screening in Survey of Autonomic Symptom (SAS) Scores at Weeks 24, 56 and 80
Description: The SAS is a 12 item (11 for females) questionnaire, from which the total number of symptoms (0-12 for males and 0-11 for females) is calculated. Each positive symptom is rated from 1 (not at all) to 5 (a lot). The total impact score was the sum of all symptom rating scores, with 0 assigned where the participant did not have the particular symptom. The range for the total impact score is 0-60 for males and 0-55 for females, higher scores indicating higher impact. Pre-specified intent of study for safety summaries until W80 was to summarize data by 4 arms.
Time Frame: Screening (up to maximum of 37 days prior to Baseline), Weeks 24, 56 and 80
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (Week 16) | Safety Evaluation: Tanezumab 5 mg | Safety Evaluation: Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 215 | 506 | 502 | 602
units on a scale
  Number of symptoms reported: Screening | 0.45 (0.79) | 0.43 (0.75) | 0.50 (0.82) | 0.48 (0.74)
  Number of symptoms reported: Change at Week 24: number analyzed (Participants) | 0 | 287 | 295 | 268
  Number of symptoms reported: Change at Week 24 |  | 0.32 (1.45) | 0.28 (1.37) | 0.51 (1.34)
  Number of symptoms reported: Change at Week 56: number analyzed (Participants) | 0 | 202 | 223 | 204
  Number of symptoms reported: Change at Week 56 |  | 0.50 (1.57) | 0.30 (1.37) | 0.60 (1.49)
  Number of symptoms reported: Change at Week 80: number analyzed (Participants) | 0 | 193 | 201 | 191
  Number of symptoms reported: Change at Week 80 |  | 0.41 (1.38) | 0.42 (1.45) | 0.45 (1.47)
  Total Symptom Impact Score: Screening | 0.93 (1.62) | 0.95 (1.69) | 1.10 (1.88) | 1.06 (1.71)
  Total Symptom Impact Score: Change at Week 24: number analyzed (Participants) | 0 | 287 | 295 | 268
  Total Symptom Impact Score: Change at Week 24 |  | 1.03 (4.05) | 0.76 (3.55) | 1.37 (3.68)
  Total Symptom Impact Score: Change at Week 56: number analyzed (Participants) | 0 | 202 | 223 | 204
  Total Symptom Impact Score: Change at Week 56 |  | 1.49 (4.53) | 0.96 (3.87) | 1.74 (3.96)
  Total Symptom Impact Score: Change at Week 80: number analyzed (Participants) | 0 | 193 | 201 | 191
  Total Symptom Impact Score: Change at Week 80 |  | 1.47 (4.26) | 1.28 (4.10) | 1.43 (3.94)

63. Secondary Outcome: Percentage of Participants With Adjudicated Joint Safety Outcomes
Description: Incidence of participants with any of the joint safety adjudication outcomes of primary osteonecrosis, rapidly progressive OA (type 1 and type 2), subchondral insufficiency fracture (or SPONK), or pathological fracture.
Time Frame: Baseline up to Week 80
Population: Safety population was analyzed. Pre-specified intent of study for safety summaries until W80 was to summarize data by 4 arms. 'N' in placebo arm=participants who received only placebo for entire study, those who were there up to W16,but switched to tanezumab after W16 are included in tanezumab 5/10mg arm.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Week 16) | Safety Evaluation: Tanezumab 5 mg | Safety Evaluation: Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 215 | 506 | 502 | 602
percentage of participants
  Composite Joint Safety Endpoint | 0 [0.0 to 1.7] | 1.0 [0.3 to 2.3] | 2.6 [1.4 to 4.4] | 0.2 [0.0 to 0.9]
  Rapidly Progressive OA | 0 [0.0 to 1.7] | 1.0 [0.3 to 2.3] | 1.8 [0.8 to 3.4] | 0.2 [0.0 to 0.9]
  Rapidly Progressive OA type 1 | 0 [0.0 to 1.7] | 1.0 [0.3 to 2.3] | 1.4 [0.6 to 2.9] | 0.2 [0.0 to 0.9]
  Rapidly Progressive OA type 2 | 0 [0.0 to 1.7] | 0 [0.0 to 0.7] | 0.4 [0.0 to 1.4] | 0 [0.0 to 0.6]
  Primary Osteonecrosis | 0 [0.0 to 1.7] | 0 [0.0 to 0.7] | 0 [0.0 to 0.7] | 0 [0.0 to 0.6]
  Pathological Fracture | 0 [0.0 to 1.7] | 0 [0.0 to 0.7] | 0 [0.0 to 0.7] | 0 [0.0 to 0.6]
  Subchondral Insufficiency Fracture | 0 [0.0 to 1.7] | 0 [0.0 to 0.7] | 0.8 [0.2 to 2.0] | 0 [0.0 to 0.6]

64. Secondary Outcome: Percentage of Participants With Total Joint Replacements
Description: Percentage of participants who underwent at least one total knee, hip or shoulder joint replacement surgery.
Time Frame: Baseline up to Week 80
Population: Safety population. Pre-specified intent of study for safety summaries until W80 was to summarize data by 4 arms. N in placebo arm=number of participants who received only placebo for entire study, those who were there up to W16,but switched to tanezumab treatment after W16 are included in tanezumab 5/10 mg arm.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo (Week 16) | Safety Evaluation: Tanezumab 5 mg | Safety Evaluation: Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 215 | 506 | 502 | 602
percentage of participants | 0 [0.0 to 1.7] | 0 [0.0 to 0.7] | 1.4 [0.6 to 2.9] | 0 [0.0 to 0.6]

65. Secondary Outcome: Change From Baseline in Neuropathy Impairment Score (NIS) at Weeks 2, 4, 8, 16, 24, 32, 40, 48, 56, 64 and 80
Description: NIS is a standardized instrument used to evaluate participant for signs of peripheral neuropathy. NIS is the sum of scores of 37 items, from both the left and right side, where 24 items scored from 0 (normal) to 4 (paralysis), higher score indicated higher abnormality/impairment and 13 items scored from 0 (normal), 1 (decreased) and 2 (absent), higher score indicated higher impairment. NIS possible overall score ranged from 0 (no impairment) to 244 (maximum impairment), higher scores indicated increased impairment. Pre-specified intent of study for safety summaries until W80 was to summarize data by 4 arms.
Time Frame: Baseline, Weeks 2, 4, 8, 16, 24, 32, 40, 48, 56, 64 and 80
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo (Week 16) | Safety Evaluation: Tanezumab 5 mg | Safety Evaluation: Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 215 | 506 | 502 | 602
units on a scale
  Baseline: number analyzed (Participants) | 215 | 506 | 502 | 601
  Baseline | 1.00 (3.55) | 0.58 (2.28) | 0.86 (2.54) | 0.78 (2.62)
  Change at Week 2: number analyzed (Participants) | 190 | 488 | 475 | 565
  Change at Week 2 | 0.02 (1.29) | 0.05 (1.12) | -0.08 (1.34) | -0.15 (1.31)
  Change at Week 4: number analyzed (Participants) | 198 | 492 | 487 | 579
  Change at Week 4 | -0.14 (1.35) | -0.02 (0.96) | -0.17 (1.57) | -0.16 (1.36)
  Change at Week 8: number analyzed (Participants) | 200 | 495 | 490 | 590
  Change at Week 8 | 0.01 (1.97) | -0.09 (1.41) | -0.17 (1.99) | 0.08 (3.53)
  Change at Week 16: number analyzed (Participants) | 200 | 495 | 490 | 590
  Change at Week 16 | -0.02 (1.91) | -0.06 (1.37) | -0.06 (1.94) | 0.02 (1.84)
  Change at Week 24: number analyzed (Participants) | 0 | 495 | 491 | 590
  Change at Week 24 |  | -0.10 (1.58) | -0.09 (1.77) | 0.03 (2.32)
  Change at Week 32: number analyzed (Participants) | 0 | 495 | 491 | 590
  Change at Week 32 |  | -0.14 (1.60) | -0.12 (1.73) | 0.03 (1.90)
  Change at Week 40: number analyzed (Participants) | 0 | 495 | 491 | 590
  Change at Week 40 |  | -0.13 (1.44) | -0.13 (1.81) | -0.02 (1.97)
  Change at Week 48: number analyzed (Participants) | 0 | 495 | 491 | 590
  Change at Week 48 |  | -0.14 (1.33) | -0.10 (1.85) | 0.00 (1.92)
  Change at Week 56: number analyzed (Participants) | 0 | 495 | 491 | 590
  Change at Week 56 |  | -0.16 (1.38) | -0.09 (2.07) | -0.03 (1.97)
  Change at Week 64: number analyzed (Participants) | 0 | 495 | 491 | 590
  Change at Week 64 |  | -0.07 (2.39) | -0.09 (2.06) | -0.06 (2.03)
  Change at Week 80: number analyzed (Participants) | 0 | 495 | 491 | 590
  Change at Week 80 |  | -0.09 (1.94) | -0.12 (2.15) | -0.07 (2.06)

66. Secondary Outcome: Number of Participants With Anti Tanezumab Antibodies
Description: Human serum ADA samples were analyzed for the presence or absence of anti-tanezumab antibodies by using a semi quantitative enzyme linked immunosorbent assay (ELISA). Participants listed as having anti-tanezumab antibodies had ADA titer level >=3.32. Less than 3.32 was considered below the limit of quantitation. Pre-specified intent of study for safety summaries until W80 was to summarize data by 4 arms.
Time Frame: Baseline, Weeks 8, 16, 32, 40, 48, 56, 64 and 80
Population: The safety population was defined as all participants treated with tanezumab or placebo SC. Here, 'n' = participants who had at least one ADA sample for ADA assessment at specified timepoints. Data not collected after W16 in placebo arm for this OM, as those who met criteria to continue, switched to active treatment with tanezumab after W16.
Measure: Count of Participants; unit: Participants
Groups:
- Safety Evaluation: Tanezumab 5 mg: Tanezumab (RN624 or PF-04383119) 5 mg injection administered SC once every 8 weeks from Day 1 and placebo tablets matched to tramadol PR, orally, once daily from Day 1 up to week 56.
- Safety Evaluation: Tanezumab 10 mg: Tanezumab (RN624 or PF-04383119) 10 mg injection administered SC once every 8 weeks from Day 1, and placebo tablets matched to tramadol PR, orally, once daily from Day 1 up to week 56.
Arm/Group | Placebo (Week 16) | Safety Evaluation: Tanezumab 5 mg | Safety Evaluation: Tanezumab 10 mg | Tramadol
Number analyzed (Participants) | 409 | 407 | 407 | 602
Participants
  Baseline: number analyzed (Participants) | 402 | 404 | 402 | 600
  Baseline | 45 | 38 | 39 | 68
  Week 8: number analyzed (Participants) | 341 | 347 | 345 | 484
  Week 8 | 37 | 32 | 54 | 49
  Week 16: number analyzed (Participants) | 200 | 235 | 241 | 313
  Week 16 | 27 | 36 | 46 | 32
  Week 32: number analyzed (Participants) | 0 | 166 | 181 | 228
  Week 32 |  | 32 | 48 | 23
  Week 40: number analyzed (Participants) | 0 | 0 | 0 | 0
  Week 48: number analyzed (Participants) | 0 | 145 | 160 | 207
  Week 48 |  | 31 | 49 | 23
  Week 56: number analyzed (Participants) | 0 | 138 | 157 | 204
  Week 56 |  | 22 | 41 | 21
  Week 64: number analyzed (Participants) | 0 | 135 | 146 | 193
  Week 64 |  | 15 | 32 | 19
  Week 80: number analyzed (Participants) | 0 | 131 | 143 | 189
  Week 80 |  | 14 | 14 | 19

ADVERSE EVENTS:
Time Frame: Baseline up to Week 80
Description: Same event may appear as both an adverse event (AE) and serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. N in placebo arm=participants who received only placebo for entire study, those who were there upto W16,but switched to tanezumab after W16 included in tanezumab 5/10mg arm.
Arm/Group | Placebo (Week 16) | Safety Evaluation: Tanezumab 5 mg | Safety Evaluation: Tanezumab 10 mg | Tramadol
All-Cause Mortality (participants affected / at risk) | 1/215 | 2/506 | 2/502 | 1/602
Serious Adverse Events (participants affected / at risk) | 7/215 | 21/506 | 37/502 | 25/602
Other Adverse Events (participants affected / at risk) | 65/215 | 201/506 | 203/502 | 275/602
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Week 16) (N=215) | Safety Evaluation: Tanezumab 5 mg (N=506) | Safety Evaluation: Tanezumab 10 mg (N=502) | Tramadol (N=602)
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 2
Pupils unequal (Eye disorders) | 0 | 1 | 0 | 0
Uveitis (Eye disorders) | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oesophageal rupture (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 1 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0
Biliary dyskinesia (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Amoebic colitis (Infections and infestations) | 0 | 0 | 1 | 0
Arthritis infective (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 1
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Procedural nausea (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0
Rapidly progressive osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 5 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0
Subchondral insufficiency fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 0 | 0
Guillain-Barre syndrome (Nervous system disorders) | 0 | 0 | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 0 | 0 | 2 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0
Foetal death (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
Unintended pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Aneurysm (Vascular disorders) | 0 | 1 | 0 | 0
Aneurysm ruptured (Vascular disorders) | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 1
Deafness neurosensory (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Depression suicidal (Psychiatric disorders) | 1 | 0 | 0 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0 | 0 | 0
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Week 16) (N=215) | Safety Evaluation: Tanezumab 5 mg (N=506) | Safety Evaluation: Tanezumab 10 mg (N=502) | Tramadol (N=602)
Constipation (Gastrointestinal disorders) | 3 | 9 | 12 | 52
Nausea (Gastrointestinal disorders) | 5 | 16 | 16 | 78
Nasopharyngitis (Infections and infestations) | 11 | 31 | 32 | 37
Upper respiratory tract infection (Infections and infestations) | 4 | 25 | 34 | 30
Fall (Injury, poisoning and procedural complications) | 4 | 26 | 20 | 18
Arthralgia (Musculoskeletal and connective tissue disorders) | 22 | 68 | 71 | 65
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 39 | 33 | 33
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 12 | 36 | 27 | 31
Dizziness (Nervous system disorders) | 4 | 12 | 11 | 44
Headache (Nervous system disorders) | 13 | 39 | 36 | 50
Somnolence (Nervous system disorders) | 6 | 5 | 7 | 33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2016-07-18): https://cdn.clinicaltrials.gov/large-docs/53/NCT02528253/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-18): https://cdn.clinicaltrials.gov/large-docs/53/NCT02528253/SAP_001.pdf